
A Phase 3, Double-blind, Randomized, Multicenter, Parallel Group, Placebo-controlled Sequential Dose Titration Study to Evaluate Efficacy, Safety and Pharmacokinetics of Mirabegron in Pediatric Subjects from 5 to < 18 Years of Age with Overactive Bladder

ISN/Protocol: 178-CL-204

Double-blind Phase 3 Study with Mirabegron and Placebo in Pediatric Subjects from 5 to < 18 Years of Age with Overactive Bladder (Dolphin Study)

# ISN/Protocol 178-CL-204

# **Version 2.0 Incorporating Substantial Amendment 1** [see Section 13]

# 11 Feb 2021

EudraCT 2016-001767-37
Pediatric Investigational Plan EMEA-000597-PIP02-10-M07

Sponsor:

Astellas Pharma Global Development Inc.

1 Astellas Way Northbrook, IL 60062, US

Protocol History:

Version 1.0 [29 Oct 2019]

Version 1.1 Incorporating Nonsubstantial Amendment 1 [13Nov2019]

The information contained in this document is supplied as a background for clinical investigations. This document contains confidential information, which is the intellectual property of Astellas. By accepting or reviewing this document, you agree to hold this information in confidence and not copy or disclose it to others or use it for unauthorized purposes except (1) as otherwise agreed to in writing; (2) where required by applicable law; (3) where disclosure is directly related to the care and safety of the research subject; and (4) where disclosure of such information is made to a member of the investigator's team who agrees to hold this information in confidence.

# **Table of Contents**

| SI | GNATUI | RES | 8 |
|---|---|---|---|
| C | ONTACT | T DETAILS OF SPONSOR'S KEY PERSONNEL | 11 |
| 1 | PRO | OTOCOL SUMMARY | 12 |
| | 1.1 | Synopsis | 12 |
| | 1.2 | Study Schema | 21 |
| | 1.3 | Schedule of Assessments | 22 |
| | 1.3.1 | Sample Collection Schedule ······ | 25 |
| 2 | INT | | 25 |
| | 2.1 | Background ····· | 25 |
| | 2.1.1 | Treatment of Overactive Bladder in Pediatric Population | 25 |
| | 2.1.2 | Nonclinical and Clinical Data | 26 |
| | 2.3 | | 26 |
| | 2.1 | 1.2.2 Clinical Data ·································· | |
| | 2.1.3 | | 29 |
| | 2.2 | | 30 |
| | 2.3 | Risk-Benefit Assessment | |
| 3 | | | 32 |
| 4 | STU | | 34 |
| | 4.1 | | 34 |
| | 4.2 | Dose Rationale | 35 |
| | 4.3 | End of Study Definition | 36 |
| 5 | STU | UDY POPULATION | <b>37</b> |
| | 5.1 | Inclusion Criteria | 37 |
| | 5.2 | Exclusion Criteria ······ | 38 |
| | 5.3 | Restrictions During the Study ······ | 40 |
| | 5.4 | Screen Failures | 40 |
| | 5.4.1 | Rescreen | 40 |
| | 5.4 | 4.1.1 Rescreen for Urinary Tract Infection or Constipation | 40 |
| | 5.4 | 4.1.2 Rescreen for Other Eligibility Criteria | 40 |
| 6 | INV | VESTIGATIONAL PRODUCT(S) AND OTHER STUDY TREATMENT(S) ···· | 41 |
| | 6.1 | Investigational Product(s) Administered and Other Study Treatment(s) | 41 |
| 11 | Feb 2021 | Astellas Page 2 | of 1 |

7

| 6.1.1 | Investigational Product(s) | 41 |
|---|---|---|
| 6.1.2 | Other Study Treatment(s) | 43 |
| 6.2 | Preparation/Handling/Storage/Accountability | 44 |
| 6.2.1 | Packaging and Labeling | 44 |
| 6.2.2 | Handling, Storage and Accountability | 44 |
| 6.3 | Randomization and Blinding | 44 |
| 6.3.1 | Blinding Method | 44 |
| 6.3.2 | Confirmation of the Indistinguishability of the Investigational Product ······· | 44 |
| 6.3.3 | Retention of the Assignment Schedule and Procedures for Treatment Code Breaking | 45 |
| 6.3.4 | Breaking the Treatment Code for Emergency | 45 |
| 6.3.5 | Breaking the Treatment Code by the Sponsor | 45 |
| 6.3.6 | Assignment and Allocation | 45 |
| 6 | , and the second se | 45 |
| 6 | 3.6.2 Randomization Number | 46 |
| 6 | 3.6.3 Subject Replacement ······ | 46 |
| 6.4 | Investigational Product(s) and Other Study Treatment(s) Compliance | 46 |
| 6.4.1 | Investigational Product(s) | 46 |
| 6.4.2 | Other Study Treatment(s) | 46 |
| 6.5 | Previous and Concomitant Treatment (Medication and Nonmedication Therapy)···· | 46 |
| 6.6 | Dose Modification ····· | 47 |
| 6.7 | Criteria for Continuation of Treatment(s) | 47 |
| STU | UDY PROCEDURES AND ASSESSMENTS | 47 |
| 7.1 | Efficacy Assessments | 48 |
| 7.1.1 | Bladder Electronic Diary | 48 |
| 7.2 | Safety Assessments | 48 |
| 7.2.1 | Adverse Events | 48 |
| 7.2.2 | Laboratory Assessments | 48 |
| 7.2.3 | Vital Signs and Electrocardiograms | 49 |
| 7.3 | 2.3.1 Clinic-measurement of Vital Signs and Electrocardiograms | 49 |
| 7.3 | 2.3.2 Self-measurement of Vital Signs | 50 |
| 7.2.4 | | 50 |
| 7.2.5 | Post Void Residual Volume Assessments ······ | 50 |
| 7.2.6 | Acceptability and Palatability Questionnaire | 51 |


| | 7.2.7 | Order of Assessments ······ | 51 |
|---|---|---|---|
| | 7.3 | Adverse Events and Other Safety Aspects ····· | 51 |
| | 7.3.1 | Time Period for Collecting Adverse Event and Serious Adverse Event Information | 51 |
| | 7.3.2 | Method of Detecting Adverse Events and Serious Adverse Events | 51 |
| | 7.3.3 | Follow-up of Adverse Events ······ | 51 |
| | 7.3.4 | Reporting of Serious Adverse Events | 52 |
| | 7.3.5 | Disease-related Events and/or Disease-related Outcomes Not Qualifying as | |
| | | Adverse Events or Serious Adverse Events | 52 |
| | 7.3.6 | Adverse Events of Special Interest | 52 |
| | 7.3.7 | 1 | 53 |
| | 7.3.8 | Supply of New Information Affecting the Conduct of the Study | 53 |
| | 7.3.9 | Urgent Safety Measures | 53 |
| | 7.3.10 | | 53 |
| | 7.4 | Pharmacokinetics | 54 |
| | 7.5 | Pharmacodynamics Immunogenicity ······ | 54 |
| | 7.6 | Electronic Clinical Outcome Assessment ······ | 54 |
| | 7.7 | Other Assessments ····· | 56 |
| | 7.8 | Total Amount of Blood | 56 |
| 8 | DIS | CONTINUATION | 56 |
| | 8.1 | Discontinuation of Individual Subject(s) From Study Treatment(s) | 56 |
| | 8.2 | Discontinuation of Individual Subject(s) From Study ···································· | 57 |
| | 8.2.1 | Lost to Follow-up | 57 |
| | 8.3 | Discontinuation of the Study Site | 57 |
| | 8.4 | | .57 |
| 9 | STA | ATISTICAL METHODOLOGY | 58 |
| | 9.1 | Sample Size ····· | 58 |
| | 9.2 | Analysis Sets····· | 59 |
| | 9.2.1 | Full Analysis Set ······ | 59 |
| | 9.2.2 | Per Protocol Set | 59 |
| | 9.2.3 | Safety Analysis Set | 59 |
| | 9.2.4 | Pharmacokinetics Analysis Set ······ | 59 |
| | 9.2.5 | Pharmacodynamic Analysis Set ······ | 59 |
| | 9.3 | Demographics and Baseline Characteristics ······ | 59 |
| 11 | Feb 2021 | Astellas Page | 4 of 15 |

| | 9.3.1 | Demographics | 60 |
|---|---|---|---|
| | 9.3.2 | Subject Disposition | 60 |
| | 9.3.3 | Previous and Concomitant Treatment (Medication and Nonmedication | |
| | | Therapy) | 60 |
| | 9.3.4 | Medical History | 60 |
| | 9.3.5 | Investigational Product Exposure | 60 |
| | 9.4 | Analysis of Efficacy | 61 |
| | 9.4.1 | Analysis of Primary Endpoint ······ | 61 |
| | 9.4 | | 61 |
| | 9.4 | 4.1.2 Secondary Analysis | 61 |
| | 9.4 | | ·62 |
| | 9.4.2 | Analysis of Secondary Endpoints ····· | 62 |
| | 9.4.3 | Analysis of Exploratory Endpoints | 62 |
| | 9.5 | Analysis of Safety | 63 |
| | 9.5.1 | Adverse Events ····· | 63 |
| | 9.5.2 | Laboratory Assessments · | 63 |
| | 9.5.3 | Vital Signs····· | 63 |
| | 9.5.4 | Physical Examination · | 64 |
| | 9.5.5 | Electrocardiogram······ | 64 |
| | 9.5.6 | Post Void Residual Volume | 64 |
| | 9.5.7 | Acceptability and Palatability Questionnaire | 64 |
| | 9.6 | Analysis of Pharmacokinetics | 64 |
| | 9.6.1 | Estimation of Pharmacokinetic Parameters | 64 |
| | 9.7 | Analysis of Pharmacodynamics Immunogenicity | 64 |
| | 9.8 | Other Analyses ····· | 65 |
| | 9.9 | Major Protocol Deviations ···································· | 65 |
| | 9.10 | Interim Analysis (and Early Discontinuation of the Study) | 65 |
| | 9.11 | Additional Conventions | 65 |
| 10 | OP1 | ERATIONAL CONSIDERATIONS | 65 |
| | 10.1 | Data Collection ······ | 65 |
| | 10.2 | Demographics and Baseline Characteristics | 66 |
| | 10.2.1 | | 66 |
| | 10.2.2 | | 66 |
| | 10.2.3 | | 66 |
| | | <i>b</i> = 1 = 1 = 1 = 0.0000 | |

| 66 |
|-----------|
| 67 |
| 67 |
| 67 |
| 67 |
| <b>68</b> |
| 69 |
| 69 |
| 69 |
| 69 |
| 69 |
| <b>70</b> |
| <b>70</b> |
| <b>70</b> |
| 71 |
| 72 |
| 72 |
| 73 |
| 73 |
| 74 |
| 74 |
| 74 |
| 74 |
| 74 |
| 74 |
| 75 |
| 76 |
| 78 |
| 78 |
| 78 |
| 78 |
| 78 |

| | 12.4. | Criteria for Causal Relationship to Investigational Product | 79 |
|---|---|---|---|
| | 12.4. | 4 Criteria for Defining the Severity of an Adverse Event | 30 |
| | 12.4. | .5 Reporting Procedures for Serious Adverse Events ···································· | 30 |
| | 12.4. | | 32 |
| | 12 | $\varepsilon$ | 32 |
| | 12 | 2.4.6.2 Lack of Efficacy ··································· | 32 |
| | 12 | 2.4.6.3 Medication Error, Overdose and "Off-label Use" | 33 |
| | 12 | 2.4.6.4 Misuse/Abuse 8 | 33 |
| | 12 | 1 | 33 |
| | 12 | | 33 |
| | 12 | | 33 |
| | 12.5 | Liver Safety Monitoring and Assessment ······ 8 | 34 |
| | 12.6 | List of Excluded Concomitant Medications 8 | 37 |
| | 12.7 | Laboratory Assessments ····· 8 | 39 |
| | 12.8 | Acceptability and Palatability Questionnaire for Tablets | )() |
| | 12.9 | Acceptability and Palatability Questionnaire for Oral Suspension | 91 |
| | 12.10 | Centiles of Heart Rate for Normal Children from Birth to 18 Years of Age | 93 |
| | 12.11 | Centers for Disease Control and Prevention Data Table of Stature for Age Chart for Males | 94 |
| | 12.12 | Centers for Disease Control and Prevention Data Table of Stature for Age Chart for Females 10 | )1 |
| | 12.13 | Clinical Study Continuity · | )8 |
| | 12.14 | List of Abbreviations and Definition of Key Study Terms | 4 |
| 13 | AT | TACHMENT 1: SUBSTANTIAL AMENDMENT 1 ··································· | 1 <b>7</b> |
| 14 | CO | OORDINATING INVESTIGATOR'S SIGNATURE ···································· | 56 |
| 15 | SP | ONSOR'S SIGNATURES ···································· | 57 |

Sponsor: APGD ISN/Protocol: 178-CL-204 EudraCT number 2016-001767-37


# **SIGNATURES**

# 1. SPONSOR'S SIGNATURES

Required signatures (e.g., protocol authors and contributors, etc.) are located in [Section 15 Sponsor's Signatures].


# 2. COORDINATING INVESTIGATOR'S SIGNATURE

The coordinating investigator's signature is located in [Section 13 Coordinating Investigator's Signature].

ISN/Protocol: 178-CL-204


# 3. INVESTIGATOR'S SIGNATURE

A Phase 3, Double-blind, Randomized, Multicenter, Parallel Group, Placebo-controlled Sequential Dose Titration Study to Evaluate Efficacy, Safety and Pharmacokinetics of Mirabegron in Pediatric Subjects from 5 to < 18 Years of Age with Overactive Bladder

ISN/Protocol: 178-CL-204

ISN/Protocol 178-CL-204

**Version 2.0 Incorporating Substantial Amendment 1** 

#### 11 Feb 2021

I have read all pages of this protocol for which Astellas is the sponsor. I agree to conduct the study as outlined in the protocol and to comply with all the terms and conditions set out therein. I confirm that I will conduct the study in accordance with International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Good Clinical Practice (GCP) guidelines and applicable local regulations. I will also ensure that subinvestigator(s) and other relevant members of my personnel have access to copies of this protocol and the ICH GCP guidelines to enable them to work in accordance with the provisions of these documents.

| Principal Inves | ture: | |
|-----------------|-------|--------------------|
| Signature: | | |
| | | Date (DD Mmm YYYY) |
| Printed Name: | | |
| Address: | | |

Sponsor: APGD ISN/Protocol: 178-CL-204 EudraCT number 2016-001767-37


# CONTACT DETAILS OF SPONSOR'S KEY PERSONNEL

| 24-hour Contact for Serious<br>Adverse Events | Please fax or email the serious adverse events/special situations worksheet to: |
|---|---|
| G 54 11 40 45 | Astellas Pharma Global Development Inc. |
| See [Appendix 12.4.5] | US Pharmacovigilance |
| Reporting Procedures for Serious Adverse Events | North America fax number: +1-888-396-3750 |
| Schous Adverse Events | North America alternate fax number: +1-847-317-1241 |
| | International fax number: +44-800-471-5263 |
| | Email: safety-us@astellas.com |
| Medical Monitor/Study<br>Physician | PPD |
| Thysician | |
| | Medical Specialties Therapeutic Area, Tokyo |
| | Astellas Pharma Inc. |
| | 2-5-1, Nihonbashi-Honcho, Chuo-ku |
| | Tokyo 103-8411, Japan |
| | PPD |
| Clinical Research Contact(s) | PPD |
| | Astellas Pharma Global Development Inc. |
| | 1 Astellas Way |
| | Northbrook, IL, 60062 |
| | PPD |
| | Astellas Pharma Global Development Inc. |
| | 1 Astellas Way |
| | Northbrook, IL, 60062 |
| | PPD |


# 1 PROTOCOL SUMMARY

# 1.1 Synopsis

| Date and Version of Protocol Synopsis: | 11 Feb 2021, Version 2.0 |
|---|---|
| Sponsor: Astellas Pharma Global Development Inc. (APGD) | Protocol Number:<br>178-CL-204 |
| Compound Name:<br>YM178 (mirabegron) | Phase of Development:<br>Phase 3 |

ISN/Protocol: 178-CL-204

# Title of Study:

A Phase 3, Double-blind, Randomized, Multicenter, Parallel Group, Placebo-controlled Sequential Dose Titration Study to Evaluate Efficacy, Safety and Pharmacokinetics of Mirabegron in Pediatric Subjects from 5 to < 18 Years of Age with Overactive Bladder

## **Planned Study Period:**

From approximately 1Q2020 to 2Q2023

### **Study Objective(s) and Endpoint(s):**

The primary, secondary and exploratory objectives and endpoints for this study are listed in the table below.

## **Study Objectives and Endpoints**

Primary and secondary objectives and endpoints apply to children only; exploratory objectives and endpoints also apply to adolescents.

| Objectives | Endpoints |
|---|---|
| Primary | |
| • To evaluate the efficacy of mirabegron in children (5 to < 12 years of age) with OAB | <ul> <li>Change from baseline at the end of the 12-week treatment period:</li> <li>Mean number of micturitions per 24 hours</li> </ul> |
| Secondary | |
| • To evaluate the efficacy of mirabegron in children (5 to < 12 years of age) with OAB | <ul> <li>Change from baseline at the end of the 12-week treatment period: <ul> <li>Mean volume voided per 24 hours</li> <li>Maximum volume voided</li> <li>Mean number of daytime incontinence episodes per 24 hours</li> <li>Mean number of nighttime incontinence episodes per 24 hours</li> <li>Mean number of daytime micturitions per 24 hours</li> </ul> </li> <li>Number of dry (incontinence-free) days per 7 days at the end of the 12-week treatment period</li> </ul> |
| To evaluate the safety and tolerability of<br>mirabegron in pediatric subjects with OAB | <ul> <li>Nature, frequency and severity of AEs</li> <li>Clinical laboratory tests (hematology, biochemistry and urinalysis)</li> <li>Vital signs (blood pressure and pulse)</li> <li>Routine 12-lead ECG</li> <li>PVR volume</li> <li>Acceptability and palatability questionnaire</li> </ul> |

Sponsor: APGD ISN/Protocol: 178-CL-204

EudraCT number 2016-001767-37


| Objectives | Endpoints |
|---|---|
| Secondary continued | |
| To evaluate the pharmacokinetics after multiple<br>dose administration of mirabegron in pediatric<br>subjects with OAB | Steady-state C <sub>max</sub> , AUC <sub>tau</sub> , C <sub>trough</sub> , T <sub>max</sub> , CL/F, and Vz/F. Additional parameters may be calculated based on the population pharmacokinetic model used |
| Exploratory | |
| To evaluate the efficacy of mirabegron in pediatric subjects (5 to < 18 years) with OAB OAB | <ul> <li>Percentage of subjects with a reduction in daytime incontinence episodes (&lt; 50% reduction [nonresponder], 50% [partial responder] and 100% [responder])</li> <li>Improvement from baseline in worst incontinence grading</li> <li>Change from baseline at the end of the 12-week treatment period adjusted for fluid intake: <ul> <li>Mean number of micturitions per 24 hours</li> </ul> </li> <li>Change from baseline at the end of the 12-week treatment period (adolescents only): <ul> <li>Mean number of micturitions per 24 hours</li> <li>Mean number of daytime micturitions per 24 hours</li> <li>Mean volume voided per 24 hours</li> <li>Mean number of incontinence episodes per 24 hours</li> </ul> </li> <li>Number of dry (incontinence-free) days per 7 days at the end of the 12-week treatment period (adolescents only)</li> <li>Mean number of daytime grade 3 or 4 (PPIUS) urgency episodes per 24 hours (adolescents only)</li> </ul> |

AE: adverse event; ECG: electrocardiogram; OAB: overactive bladder; PPIUS: patient perception of intensity of urgency scale; PVR: post void residual.

#### **Estimand**

The estimand of most clinical importance for this study is defined by the following 4 attributes:

- Target population: all children who took at least 1 dose of the study drug, and in whom a nonmissing measurement for micturition frequency at baseline and after administration of the study drug is available
- Outcome measurement: micturition frequency/day (24 hours)
- Intercurrent events:
  - 1. Discontinuation from treatment (if week 12/EoT not obtained)
  - 2. AE urinary tract infection (UTI) (if occurred in week 12/EoT)
  - 3. Other muscarinic antagonists or botulinum toxin (if taken during the last 2 weeks prior to week 12/EoT assessment); in all cases, a hypothetical strategy will be applied
- Population-based summary: Change from baseline to week 12/EoT in micturition frequency/day (= primary endpoint, primary estimator), compared to placebo

For this placebo-controlled study, this "de jure" estimand chosen is considered the appropriate choice. As some effect is expected early in the study and with continued treatment could be expected to be maintained, it's considered appropriate to impute for subjects with missing values at visit 7/week 12/EoT by their last recorded post baseline visit value prior to it. This strategy also assumes that the responses after the intercurrent event would be same as for patients continuing on their respective treatment.


# Planned Total Number of Study Sites and Location(s):

Approximately 65 study sites

Europe, Latin America, Africa, Middle East, Asia-Pacific and North America

## **Study Population:**

Male and female pediatric subjects 5 to < 18 years of age with overactive bladder (OAB; as defined according to the International Children's Continence Society [ICCS]) who have had received 4 weeks of urotherapy prior to randomization

ISN/Protocol: 178-CL-204

#### Number of Subjects to be Enrolled/Randomized:

Approximately 368 children enrolled to achieve 184 children (5 to < 12 years of age) randomized and approximately 64 adolescents enrolled to achieve at least 32 adolescents (12 to < 18 years of age) randomized (at least 92 children and 16 adolescents must be randomized to mirabegron)

#### **Study Design Overview:**

This is a double-blind, randomized, multicenter, parallel group, placebo-controlled sequential dose titration study to evaluate efficacy, safety and pharmacokinetics of mirabegron in pediatric subjects with OAB. Subjects will have to receive 4 weeks of urotherapy prior to randomization.

The study consists of 3 periods with a total duration of 18 weeks.

• Screening period/urotherapy (4 weeks):

This period starts with visit 1/week -4 (screening) and ends with visit 3/week 0 (baseline). After informed consent/assent has been obtained and immediately after eligibility has been confirmed at visit 1/week -4 (screening), subjects using prohibited medication will complete 1 week of washout (if applicable), while beginning 4 weeks of urotherapy.

After a successful screening visit (visit 1/week -4 [screening]), all subjects will complete a 2-day bladder e-diary (weekend) to get acquainted with the bladder e-diary and the assessments. Completion of this bladder e-diary should start in the weekend prior to visit 2. All subjects will also complete a 7-day bladder e-diary the week prior to the baseline visit. The 7-day diary will consist of a 5-day weekday bladder e-diary and 2-day weekend e-diary.

• Double-blind, placebo-controlled period (12 weeks):

This period starts with the day after visit 3/week 0 (baseline) and ends with visit 7/week 12 (end of treatment [EoT]).

At visit 3/week 0 (baseline) inclusion and exclusion criteria will be evaluated. Subjects continuing urotherapy who still meet the OAB entry criteria at baseline will be randomized. Subjects whose symptoms are not satisfactorily controlled with urotherapy and still fulfill the inclusion/exclusion criteria will enter the study. These subjects will be randomized to receive mirabegron in pediatric equivalent dose 25 mg (PED25) or placebo using a 1:1 ratio. Subjects with a body weight of  $\geq$  35 kg are to receive the tablet unless unable to swallow tablets and would be provided the oral suspension as an alternative. Subjects with a body weight < 35 kg or those who cannot be dosed with the tablet will receive an oral suspension. Daily investigational product (IP) administration will start on day 1 (i.e., the day after this visit) and continue at this dose until visit 5/week 4 (i.e., for 4 weeks). Urotherapy will continue throughout the study treatment period until visit 7/week 12 (EoT).

At visit 5/week 4, dose up-titration to mirabegron in pediatric equivalent dose 50 mg (PED50) will be performed unless the investigator determines that the subject is adequately treated for OAB at the PED25 dose or if there are safety concerns identified and considered associated with the use of PED25. Dose down-titration from PED50 to PED25 can be done at any time thereafter for safety reasons.

Subjects will start with the subsequent 7-day bladder e-diaries approximately 7 days prior to the indicated visit (or TC).

Pharmacokinetic blood samples will be collected at visit 5/week 4 and visit 7/week 12 (EoT) as indicated in the Schedule of Assessments.


## • Follow-up period (2 weeks):

This period starts the day after visit 7/week 12 (EoT) and ends with visit 8/week 14 (end of study [EoS]). The follow-up period is applicable to all subjects who have been randomized and received IP.

ISN/Protocol: 178-CL-204

At visit 7/week 12 (EoT), IP administration will be stopped and a safety observation period of 2 weeks will start.

An independent Data and Safety Monitoring Board (DSMB) will be established. A separate charter will describe the responsibilities of the DSMB.

The IP will not be provided after study completion without written approval from the sponsor.

#### **Inclusion/Exclusion Criteria:**

#### **Inclusion Criteria**

Subject is eligible for the study if all of the following apply:

# Inclusion at Visit 1/Week -4 (Screening)

- 1. Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved written informed consent/assent and privacy language as per national regulations (e.g., General Data Protection Regulations for European Union study sites) must be obtained from the subject and/or from the subject's parent(s)/legal guardian(s) prior to any study-related procedures (including withdrawal of prohibited medication, if applicable); assent by the subject is obtained as required by local law.
- 2. Subject has OAB defined according to the ICCS criteria.
- 3. Subject is a male or female between 5 to < 18 years of age, at screening.
- 4. Subject weighs at least 13 kg at screening.
- 5. Subject is able to take the IP in accordance with the protocol.
- 6. Subject agrees to drink an adequate fluid volume during urine collection weekends, as instructed by the investigator.
- 7. Subject and subject's parent(s)/legal guardian(s) agree that the subject will not participate in another interventional study while participating in the present study.
- 8. Subject and subject's parent(s)/legal guardian(s) are willing and able to comply with the study requirements and with the concomitant medication restrictions.
- 9. Female subject is not pregnant (see [Appendix 12.3 Contraception Requirements]) and at least 1 of the following conditions apply:
  - a. Not a female of childbearing potential (see [Appendix 12.3 Contraception Requirements]).
  - b. Female of childbearing potential who agrees to follow the contraceptive guidance (see [Appendix 12.3 Contraception Requirements]) from the time of informed consent/assent through at least 30 days after final IP administration.
- 10. Female subject must agree not to breastfeed starting at screening and throughout the study period and for 30 days after final IP administration.
- 11. Female subject must not donate ova starting at first dose of IP and throughout the study period and for 30 days after final IP administration.
- 12. Male subject with female partner(s) of childbearing potential (including breastfeeding partner[s]) must agree to use contraception (see [Appendix 12.3 Contraception Requirements]) throughout the treatment period and for 30 days after final IP administration.
- 13. Male subject must agree not to donate sperm during the treatment period and for 30 days after final IP administration.
- 14. Male subject with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 30 days after final IP administration.

# Additional Inclusion at Visit 3/Week 0 (Baseline)

15. Subject must have a micturition frequency of at least 8 times (on average) per day, in the 7 days prior to visit 3/week 0 (baseline), as recorded in the bladder e-diary.


16. Subject must have at least 1 daytime incontinence episode (on average) per day, during the 7-day period before visit 3/baseline, as recorded in the bladder e-diary.

ISN/Protocol: 178-CL-204

17. Subject whose symptoms are not satisfactorily controlled with urotherapy and still fulfills the inclusion/exclusion criteria will enter the study.

#### **Exclusion Criteria**

Subject will be excluded from participation in this study if any of the following apply:

### Exclusion at Visit 1/Week -4 (Screening)

- 1. Subject has extraordinary daytime only urinary frequency according to the ICCS definition.
  - This applies to a toilet-trained child who has the frequent need to void that is associated with small micturition volumes solely during the day.
  - The daytime voiding frequency is at least once per hour with an average voided volume of < 50% of expected bladder capacity (EBC) (typically 10% to 15%).
  - Incontinence is rare and nocturia is absent.
- 2. Subject has an uroflow indicative of pathology other than OAB.
- 3. Subject has monosymptomatic enuresis.
- 4. Subject has dysfunctional voiding.
- 5. Subject has bladder outlet obstruction, except if successfully treated.
- 6. Subject has anatomical anomalies (surgically treated or untreated) that affect lower urinary tract function.
- 7. Subject with hematuria on dipstick test. In the case of hematuria on dipstick test in a female during menstruation, the test can be repeated before randomization (after the end of menstruation).
- 8. Subject with diabetes insipidus.
- 9. Subject has kidney or bladder stones.
- 10. Subject has suffered from chronic UTI or has had more than 3 UTIs in the 2 months prior to visit 1/week -4 (screening).
- 11. Criterion has been removed.
- 12. Subject has stage 2 hypertension or subject has stage 1 hypertension that is not well controlled, as defined by the 2017 American Academy of Pediatrics Clinical Practice Guidelines.
- 13. Subject has QTcF > 440 msec on screening ECG, a risk of QT prolongation (e.g., hypokalemia, long QT syndrome [LQTS] or family history of LQTS or exercise-induced syncope) or is currently taking medication known to prolong the QT interval.
- 14. Subject's aspartate aminotransferase (AST) or alanine aminotransferase (ALT) is  $\geq 2 \times$  upper limit of normal (ULN) or total bilirubin (TBL) is  $\geq 1.5 \times$  ULN according to age and sex (subjects with Gilbert's syndrome are excepted from the bilirubin threshold).
- 15. Subject has mild or moderate renal impairment (estimated glomerular filtration rate according to the modified Schwartz of < 60 mL/min per 1.73 m<sup>2</sup>).
- 16. Subject has a symptomatic (symptoms can include pain, fever, hematuria, new onset foul-smelling urine) UTI. Note: if the UTI is treated successfully (clinical recovery: confirmed by dipstick test and repeated dipstick test after 14 days [both should be negative]), the subject can be rescreened.
- 17. Subject has a history or presence of any malignancy.
- 18. Subject uses any drugs that are sensitive cytochrome P450 2D6 (CYP2D6) substrates with a narrow therapeutic index, sensitive P-glycoprotein (P-gp) substrates, or moderate or strong cytochrome CYP3A4/5 or P-gp inhibitors or inducers after the start of washout.
- 19. Subject is using or has used prohibited prior and/or concomitant medication(s) [Appendix 12.6 List of Excluded Concomitant Medications] that cannot be discontinued.
- 20. Subject has known or suspected hypersensitivity to mirabegron or any components of the formulations used.
- 21. Subject has participated in another clinical study (and/or subject has received any investigational


therapy within 30 days (or 5 half-lives of the drug, or the limit set by national law, whichever is longer) prior to visit 1/week -4 (screening).

ISN/Protocol: 178-CL-204

- 22. Subject received urinary catheterization within 2 weeks prior to screening.
- 23. Subject has constipation as defined by the Rome IV criteria that cannot be successfully treated prior to study entry.
- 24. Female subject who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
- 25. Subject has any condition, which in the opinion of the investigator, makes the subject unsuitable for study participation.

#### Additional Exclusion at Visit 3/Week 0 (Baseline)

- 26. Subject has extraordinary daytime only urinary frequency according to the ICCS definition based on the bladder e-diary.
- 27. Subject has monosymptomatic enuresis confirmed by the bladder e-diary.
- 28. Subject has a maximum voided volume (morning volume excluded) > EBC for age ([age +1]  $\times$  30) in mL, based on the bladder e-diary.
- 29. Subject has polyuria defined as voided urine volumes of > 40 mL/kg baseline body weight during 24 hours or > 2.8 L urine for a child weighing ≥ 70 kg (ICCS definition) [Austin et al, 2014], based on bladder e-diary.
- 30. Subject has PVR volume > 20 mL (lowest PVR volume result) as measured by ultrasonography.
- 31. Subject suffers from a symptomatic (symptoms can include pain, fever, hematuria, new onset foul-smelling urine) UTI. Note: if a symptomatic UTI is present, all visit 3/week 0 (baseline) assessments must be postponed until the UTI is successfully treated (clinical recovery: confirmed by dipstick test and repeated dipstick test after 14 days [both should be negative]), and the urotherapy should continue. The postponed visit 3/week (baseline) should be within 14 days of the intended visit 3/week 0 (baseline).
- 32. Subject with hematuria on dipstick test. In the case of hematuria on dipstick test in a female during menstruation, the test can be repeated before randomization (after the end of menstruation).
- 33. Subject has a pulse > 99<sup>th</sup> percentile for age.
- 34. Subject has stage 2 hypertension or subject has stage 1 hypertension that is not well controlled, as defined by the 2017 American Academy of Pediatrics Clinical Practice Guidelines.
- 35. Any reason, in the opinion of the investigator, that makes the subject unsuitable for study participation.

# **Investigational Product(s):**

#### Name/Use:

Mirabegron tablets in 25 mg and 50 mg (test product) and matching placebo Mirabegron oral suspension containing 8 mg/mL (test product) and matching placebo

#### Dose(s):

Once daily dosing according to the table below.


**Body Weight-based Doses for Tablets or Suspension** 

| | Body Weight Range†<br>(kg) | Oral Suspension Volume‡ (mL) | Tablet Dose (mg) |
|---|---|---|---|
| | 13 to < 22 | 3 | - |
| PED25 | 22 to < 35 | 4 | - |
| | ≥ 35 | 6 | 25 |
| | 13 to < 22 | 6 | - |
| PED50 | 22 to < 35 | 8 | - |
| | ≥ 35 | 11 | 50 |

ISN/Protocol: 178-CL-204

PED25: pediatric equivalent dose 25 mg; PED50: pediatric equivalent dose 50 mg

- † Subjects with a body weight  $\geq$  35 kg will receive the tablet. Subjects with a body weight  $\leq$  35 kg or those who cannot be dosed with the tablet will receive an oral suspension.
- ‡ Oral suspension containing 8 mg/mL.

The starting dose will be PED25 starting administration the day after visit 3/week 0 (baseline). At visit 5/week 4, dose up-titration to PED50 will be performed unless the investigator determines that the subject is adequately treated for OAB at the PED25 dose or if there are safety concerns identified and considered associated with the use of PED25. Dose down-titration from PED50 to PED25 can be done at any time thereafter for safety reasons.

#### **Mode(s) of Administration:**

IP will be administered orally, once daily in the morning around the same time of day and around time of food intake (i.e., within 1 hour before or after breakfast).

Tablets will be administered with a sip of water (tablet should be taken as a whole and should not be chewed, divided or crushed). Oral suspension will be administered via an oral syringe with a sip of water afterwards.

#### **Dose Modifications:**

Dose down-titration from PED50 to PED25 can be done at any time for safety reasons.

#### **Other Study Treatment(s):**

During the screening period, all subjects will receive 4 weeks of urotherapy. At visit 3/week 0 (baseline), inclusion and exclusion criteria will be evaluated. Subjects continuing urotherapy who still meet the OAB entry criteria at baseline will be randomized. Urotherapy will continue throughout the study treatment period until visit 7/week 12 (EoT).

# **Concomitant Treatment (Medication and Nonmedication Therapy) Restrictions or Requirements:**

Subjects are not allowed to use ongoing treatment with any of the following prohibited medications after the start of the washout:

- Any medication, other than the IP, used for the treatment of OAB (including tricyclic antidepressants, 1st generation H1 antagonists and alpha blockers)
- Any drugs that are sensitive CYP2D6 substrates with a narrow therapeutic index or sensitive P-glycoprotein substrates
- Any medications known to prolong the QT interval
- Any medication that is a moderate or strong cytochrome CYP3A4/5 or P-gp inhibitor or inducers including natural and herbal remedies
- Intradetrusor botulinum toxin injections; except if given > 9 months prior screening and symptoms reappeared comparable to those before botulinum toxin injections


• Nonmedication therapies like urotherapy, chiropractic, physical therapy will also be collected on the nonmedication therapy case report form.

The site will need to make special notes for those subjects who do not follow urotherapy for 7 or more consecutive days in electronic case report forms.

ISN/Protocol: 178-CL-204

These treatments are prohibited from being started after the start of the washout period. All other concomitant treatment use will be reported.

The use of previous and concomitant treatment within 30 days prior to signing the informed consent and throughout the study will be documented on the appropriate electronic case report form.

## **Duration of Treatment:**

Once daily dosing for 12 weeks

#### **Treatment Discontinuation Criteria:**

## **Discontinuation of Individual Subject(s) From Study Treatment(s):**

A subject must discontinue study treatment for any of the following reasons:

- Subject requests to stop treatment.
- Any clinical adverse events, laboratory abnormality or intercurrent illness, in the opinion of the investigator, indicates continued treatment is not in the best interest of the subject
- If signs or symptoms of hypersensitivity to mirabegron are observed (e.g., anaphylactic reaction, erythema multiforme or exfoliative dermatitis).
- ALT or AST  $> 8 \times ULN$ .
- ALT or AST  $> 5 \times$  ULN for more than 2 weeks.
- ALT or AST >  $3 \times \text{ULN}$  and TBL >  $2 \times \text{ULN}$  or international normalized ratio (INR) > 1.5 (if INR testing is applicable/evaluated).
- ALT or AST  $> 3 \times$  ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash and/or eosinophilia (> 5%).
- Female subject becomes pregnant.
- Prolongation of QT > QTcF > 440 msec and/or QT interval prolongation > 30 msec versus baseline.
- Subject with (systolic blood pressure  $\geq 160$  mm Hg or diastolic blood pressure  $\geq 100$  mmHg.

If a subject discontinues treatment prematurely, the subject will be encouraged to complete all scheduled visits to record all available information.

## **Discontinuation of the Study:**

The independent data monitoring committee will review safety data periodically and provide a recommendation to the sponsor if the study should continue or be stopped due to safety concerns. The sponsor may terminate this study prematurely, either in its entirety or at any study site, for reasonable cause provided that written notice is submitted in advance of the intended termination. Advance notice is not required if the study is stopped due to safety concerns. If the sponsor terminates the study for safety reasons, the sponsor will immediately notify the investigator and subsequently provide written instructions for study termination. The study may also be stopped as a result of the outcome of the interim analysis.

#### **Statistical Methods:**

#### **Sample Size Justification:**

Efficacy of mirabegron in children will be based on both primary and secondary endpoints. Given the clinical hurdle to demonstrate efficacy in a population challenging to recruit, an alpha-level of 10% would appear reasonable and justified. In a study with propiverine in children, a difference in mean number of micturition episodes/24 hours of 0.8 between propiverine and placebo was observed, with a SD between 2.2 and 2.3. Assuming at least similar efficacy of mirabegron, with a treatment effect of 0.9 micturitions per day between mirabegron and placebo and a common SD of 2.3, a sample size of 82 evaluable subjects (children) per treatment group is assumed per treatment group would provide a


power of 80%. Under the assumption that after randomization about 10% of the subjects will not be evaluable for the analysis of the primary endpoint (i.e., not fulfilling the criteria for inclusion in full analysis set), at least 184 children (5 to < 12 years of age) must be randomized in order to have at least 164 evaluable children for the analysis of the primary efficacy endpoint. For adolescents, no formal sample size will be calculated, at least 32 adolescents (12 to < 18 years of age) must be randomized, yielding at least 16 adolescents on mirabegron. Further assuming a 50% screen failure rate, approximately 368 children have to be enrolled to achieve 184 children (5 to < 12 years of age) randomized and approximately 64 adolescents will be enrolled to achieve at least 32 adolescents (12 to < 18 years of age) randomized (at least 92 children and 16 adolescents must be randomized to mirabegron). Recruitment will continue until the minimum number to be randomized in both children and adolescents have been achieved.

ISN/Protocol: 178-CL-204

## **Efficacy:**

The primary analysis of the primary efficacy end-point in children (5 to < 12 years of age), change from baseline to visit 7/week 12 (EoT) in mean number of micturitions per 24 hours, will be analyzed using an analysis of covariance (ANCOVA). The ANCOVA model will include treatment group, sex and geographical region as fixed effects and the mean number of micturitions per 24 hours at visit 3/week 0 (baseline) as covariate.

The secondary analysis will be a repeated measures ANCOVA. This model will include treatment group, visit (week 4, 8, 12), sex, geographical region and the interaction between treatment group and visit as fixed effects and mean number of micturitions per 24 hours at baseline as covariate. Mirabegron will be compared to placebo using a linear contrast within the repeated measures ANCOVA model, with 2-sided significance level of alpha = 0.1 and 90% CI.

In addition to the parametric ANCOVA, a nonparametric ANCOVA will also be performed: (stratified) rank ANCOVA.

#### Safety:

Safety endpoints will be summarized using descriptive statistics. Safety parameters such as vital signs will be summarized with respect to age- and sex-specific percentiles. Clinical laboratory tests (hematology, biochemistry and urinalysis [urinalysis dipstick]) and electrocardiogram results will also be summarized.

#### Pharmacokinetics:

Pharmacokinetic parameters will be summarized using descriptive statistics.

## Pharmacodynamics | Immunogenicity:

Not applicable.

#### **Interim Analyses:**

A blinded interim analysis will be performed after 50% of children planned to be randomized have had their week 12/EoT assessment. The interim analysis will determine if the chance of a positive study with respect to the primary endpoint at the EoS is high enough to justify continuation of the study; otherwise, the study will be stopped for futility.

Sponsor: APGD
EudraCT number 2016-001767-37

ISN/Protocol: 178-CL-204


# 1.2 Study Schema

# Figure 1 Study Schema



EoS: end of study; EoT: end of treatment; ICF: informed consent form; PED25: pediatric equivalent dose 25 mg; PED50: pediatric equivalent dose 50 mg

EudraC1 number 2010-001/6/-


# 1.3 Schedule of Assessments

# Table 1 Schedule of Assessments

| | Screening Period/Urotherapy<br>(4 weeks) | | Double-blind Placebo-controlled Period (12 weeks) | | | | Follow-up Period<br>(2 weeks) | |
|---|---|---|---|---|---|---|---|---|
| | Visit 1 | Visit 2/TC <sup>a</sup> | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 |
| Schedule of Assessments | Week -4<br>Screening | Week -2 | Week 0<br>Baseline | Week 2<br>TC <sup>a</sup> | Week 4 | Week 8<br>TC <sup>a</sup> | Week 12<br>(EoT) <sup>b</sup> | Week 14<br>(EoS) <sup>b,c</sup> |
| | Day -28 | Day -14 | Day -1 | Day 14 | Day 28 | Day 56 | Day 84 | Day 98 |
| | (-3 days) | (± 5 days) | | (± 3 days) | (± 3 days) | $(\pm 3 \text{ days})$ | (± 3 days) | (+ 3 days) |
| Obtaining Informed Consent/Assent | X | | | | | | | |
| Inclusion and Exclusion Criteria | X | | X | | | | | |
| Washout | X <sup>d</sup> | | | | | | | |
| Urotherapy | X | X | X | X | X | X | X | |
| Demographics and Medical History | X | | | | | | | |
| Previous and Concomitant Medication | X | | X | X | X | X | X | X |
| Physical Examination | X | | | | X | | X | |
| Height and Body Weight | X | | X | | | | X | |
| Uroflow | X | | | | | | | |
| Dose Titration <sup>e</sup> | | | | | X | | | |
| Dispense IPf | | | X | | X | | | |
| Drug Accountability | | | X | | X | | X | |
| Vital Signs <sup>g</sup> | X | | X | | X | | X | X |
| $SBPM^h$ | | X | X | X | X | X | X | |
| Routine 12-lead ECG <sup>g</sup> | X | | X | | X | | X | |
| Clinical Laboratory Tests (Hematology and Biochemistry) | X | | Xi | | X | | X | Xi |
| Clinical Laboratory Tests (Urinalysis) | X | | Xi | | X | | X | Xi |
| Pregnancy Test <sup>j</sup> | X | | X | | X | | X | X |
| PVR Volume <sup>k</sup> | | | X | | X | | X | X |
| AEs | X | X | X | X | X | X | X | X |
| Bladder e-diary <sup>a,l</sup> | | X | X | X | X | X | X | |

Table continued on next page

Sponsor: APGD ISN/Protocol: 178-CL-204

EudraCT number 2016-001767-37


| | Screening Period/Urotherapy<br>(4 weeks) | | Double-blind Placebo-controlled Period (12 weeks) | | | | Follow-up Period (2 weeks) | |
|---|---|---|---|---|---|---|---|---|
| | Visit 1 | Visit 2/TC <sup>a</sup> | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 |
| Schedule of Assessments | Week -4 | Week -2 | Week 0 | Week 2 | Week 4 | Week 8 | Week 12 | Week 14 |
| | Screening | | Baseline | TCa | | TCa | (EoT) <sup>b</sup> | (EoS) <sup>b,c</sup> |
| | Day -28 | Day -14 | Day -1 | Day 14 | Day 28 | Day 56 | Day 84 | Day 98 |
| | (-3 days) | (± 5 days) | | (± 3 days) | (± 3 days) | (± 3 days) | (± 3 days) | (+ 3 days) |
| Acceptability and Palatability Questionnaire <sup>m</sup> | | | | | | | X | |
| Pharmacokinetics <sup>n</sup> | | | | | X | | X | |

AE: adverse event; ECG: electrocardiogram; e-diary: electronic diary; EoS: end of study; EoT: end of treatment; IP: investigational product; PED25: pediatric equivalent dose 25 mg; PED50: pediatric equivalent dose 50 mg; PVR: post void residual; SBPM: self blood pressure monitoring; TC: telephone call

- a. For the visits where a TC is indicated, there is no need for the subject to visit the clinic provided that the bladder e-diary data are reviewed by the investigator prior to the TC and discussed and confirmed with the subject or parent(s)/legal guardian(s) during the TC. Urotherapy is also to be discussed and confirmed with the subject or parent(s)/legal guardian(s) during each TC.
- b. Subjects who withdraw early from the study after having received IP should complete both the EoT and EoS visits.
- c. The EoS visit (visit 8/week 14 [EoS]) should take place at least 14 days after the EoT visit (visit 7/week 12 [EoT]).
- d. Subjects using prohibited medication will complete 1 week of washout (if applicable), while beginning 4 weeks of urotherapy.
- e. Dose up-titration to PED50 to occur at visit 5/week 4 unless investigator determines OAB is adequately controlled. Dose down-titration from PED50 to PED25 can be done at any time for safety reasons.
- f. Daily IP administration will start on day 1 (i.e., the day after visit 3/week 0 [baseline]).
- g. Blood pressure, pulse, body temperature and ECGs will all be measured in single measurements. Subject to be in the sitting position (when possible, otherwise supine, but always in the same position for each procedure). Subject should have been calm and without distress for at least 5 minutes. Preferably, the right arm should be used to measure vital signs. Body temperature will be measured with an ear thermometer. Clinic measurements will be used to assess eligibility.
- h. SBPM will be measured once in the morning and evening during the 2-day weekend bladder e-diary collection period. SBPM measurements should start in the weekend prior to week -2 and be taken in the weekend prior to the indicated visit (or TC). SBPM will be measured on 2 consecutive days at 1 and 2 weeks after start of dosing with PED25 (day 1) and after up-titration to PED50, if not already covered by the scheduled SBPM. Measurements will be taken in the sitting position (when possible, otherwise supine, but always in the same position). Preferably, the right arm should be used. Subject should have been calm and without distress for at least 5 minutes. Morning measurement should be taken before IP intake and evening measurement should be taken prior to bedtime.
- i. Additional hematology, biochemistry and urinalysis (urinalysis dipstick) tests will be performed at visit 3/week 0 (baseline) and visit 8/week 14 (EoS) only if an AE related to hematology, biochemistry or urinalysis parameters occurred since the previous visit or at the discretion of the investigator.
- j. Urine pregnancy test will be performed for females of childbearing potential at all on-site visits.

Footnotes continued on next page

Sponsor: APGD

EudraCT number 2016-001767-37


k. PVR volume will be assessed by ultrasonography at visit 3/week 0 (baseline), visit 5/week 4, visit 7/week 12 (EoT) and visit 8/week 14 (EoS). For each subject, the same method should be used throughout the study. The bladder should only be emptied when it was initially filled with preferably > 50% of the bladder capacity for age. Every attempt should be made to measure PVR volume within a minute of voiding. A PVR volume of ≤ 20 mL is sufficient and the assessment does not have to be repeated. If the PVR volume is > 20 mL, the PVR volume assessment should be repeated (filled with preferably > 50% of the bladder capacity for age). If the subject is unable to complete a second measurement, it is up to the investigator to judge whether it can be skipped (and write the reason in the case report form). At visit 3/week 0 (baseline), the lowest PVR volume result measured should be used to evaluate the exclusion criterion. In case the lowest PVR volume measured is > 20 mL at visit 3/week 0 (baseline), the subject should be excluded from the study.

- 1. At the end of a successful screening visit (visit 1/week -4 [screening]), all subjects will be provided with a device to collect diary information. At the weekend prior to the week -2 visit, the subject will complete the 2-day bladder e-diary to get acquainted with the data collection. The 2-day diary will be reviewed at the week -2 visit. If completion is successful, all subjects will start with the 7-day bladder e-diary completion approximately 7 days prior to the indicated visit (or TC). The bladder e-diary is used for a 7-day period to record micturition frequency and incontinence episodes; it also contains a 2-day weekend period to record additional volume measurements and vital signs.
- m. The acceptability and palatability questionnaire will be completed on one weekend day proceeding at visit 7/week 12 (EoT).
- n. There will be 2 pharmacokinetic sampling days at visit 5/week 4 and visit 7/week 12 (EoT). Both pharmacokinetic sampling days will consist of collecting 1 predose (trough) sample. On pharmacokinetic sampling days, dosing should occur in the clinic and breakfast should be eaten at the clinic within 1 hour before dosing.


# 1.3.1 Sample Collection Schedule

There will be 2 pharmacokinetic sampling days at visit 5/week 4 and visit 7/week 12 (EoT). Both pharmacokinetic sampling days will consist of collecting 1 predose (trough) sample. On pharmacokinetic sampling days, dosing should occur in the clinic and breakfast should be eaten at the clinic within 1 hour before dosing.

ISN/Protocol: 178-CL-204

 Table 2
 Sample Collection Schedule

| Visit | Time Point | Collection Window | Whole Blood<br>Pharmacokinetics |
|---|---|---|---|
| Visit 5/week 4 | Predose (trough) | Approximately 24 hours after previous dose | X |
| Visit 7/week 12<br>(EoT) | Predose (trough) | Approximately 24 hours after previous dose | X |

EoT: end of treatment

#### 2 INTRODUCTION

# 2.1 Background

The present study is designed to evaluate efficacy, safety and pharmacokinetics of mirabegron in pediatric subjects with overactive bladder (OAB).

The study is part of the sponsor's clinical program for development of mirabegron for the treatment OAB in pediatric patients. Current drug therapy for OAB consists of oral antimuscarinics such as oxybutynin. Although the vast majority (approximately 90%) of patients can be treated successfully with this, development of alternative therapy is desirable because of insufficient efficacy and/or the side effects of available therapies.

Mirabegron is a first-in-class, selective human beta 3-adrenergic receptor (AR) agonist, represents a class of drugs for treatment of OAB with a direct mechanism of action. Mirabegron activation of beta 3-AR in the human bladder results in a relaxation of the detrusor smooth muscle during the fill-void cycle without interfering with the voiding contraction. Mirabegron is currently available as 25 mg and 50 mg tablets. An oral suspension is also being investigated for the treatment of OAB and neurogenic detrusor overactivity (NDO) in the pediatric population.

The population for this pediatric clinical efficacy study (Study 178-CL-204) with mirabegron is pediatric patients with OAB.

# 2.1.1 Treatment of Overactive Bladder in Pediatric Population

Classical treatment of OAB in pediatric patients consists of urotherapy followed by antimuscarinic therapy if the urotherapy is not sufficient. Other therapies for OAB are also described.


EudraCT number 2016-001767-37

# **Urotherapy**

Standard urotherapy includes information on and demystification of the voiding function and dysfunction, instruction on voiding habits (such as regular voiding, voiding posture), life style advice regarding fluid intake, prevention of constipation, recording of symptoms and voiding habits in bladder diaries and support via regular follow-up by a caregiver.

ISN/Protocol: 178-CL-204

Specific interventions include various forms of pelvic floor training (relaxation, contraction), behavioral modification, electrical stimulation, catherization and biofeedback (use of objective measures, e.g., uroflow or surface electromyography (EMG) to show children how far they relax their pelvic floor during voiding). Urotherapy can also include elements of cognitive behavioral therapy [Nevéus et al, 2006].

# Other Therapies for OAB

Alternative drug therapy for OAB includes antimuscarinic therapy such as oxybutynin.

Neuromodulation is also used in patients who do not respond adequately to drug therapy.

## 2.1.2 Nonclinical and Clinical Data

Detailed information from nonclinical and clinical studies conducted with mirabegron can be found in the Investigator's Brochure. Nonclinical and clinical data are also summarized in the current locally-available product information for mirabegron.

#### 2.1.2.1 Nonclinical Data

The standard nonclinical pharmacology studies as conducted for the use of mirabegron in adult patients with OAB are also relevant for its use in adolescent pediatric patients with OAB or NDO. Primary nonclinical pharmacology data for mirabegron qualitatively but not quantitatively translates to human clinical use in OAB. Other pharmacological effects such as the glucogenolytic effects of mirabegron in rodents did not translate to an effect in humans. These differences relate to species differences in molecular biology of the beta 3-AR, differences in receptor distribution, and differences in coupling to downstream effector mechanisms. From these factors only receptor expression or receptor-effector coupling efficiency are likely to vary by age. No detailed information is available on potential differences in expression for beta 3-AR in humans or animals during maturation. The sparse data available [Derweesh et al, 2000] suggest that any changes in beta-adrenergic responsiveness in rat urinary bladder could be expected at older age rather than at infancy or adolescence.

#### 2.1.2.2 Clinical Data

The main clinical aspects of mirabegron prolonged-release tablets in adults are described in the current locally-available product information for mirabegron.

To support the doses and formulations (tablets and oral suspension) selected for this study, the pediatric development program for mirabegron includes 4 phase 1 studies [Table 3].


Table 3 Overview of Current Supporting Mirabegron Studies in the Pediatric Clinical Development Program for Neurogenic Detrusor Overactivity and Overactive Bladder

| Study Number | Study Title | Study Progress |
|---|---|---|
| 178-CL-201 | A phase 1, single dose, 4-period crossover study to assess the bioavailability of mirabegron oral suspension relative to the mirabegron prolonged-release tablet and to assess the effect of food on the pharmacokinetics of mirabegron oral suspension in healthy young male and female subjects | Completed |
| 178-CL-202 | A multicentre, open-label, single ascending dose phase 1 study to evaluate the pharmacokinetics, safety and tolerability of mirabegron OCAS tablets in pediatric subjects from 5 to less than 18 years of age with NDO or OAB | Completed |
| 178-CL-203 | A multicentre, open-label, single dose, phase 1 study to evaluate the pharmacokinetics, safety and tolerability of mirabegron oral suspension in pediatric subjects from 3 to less than 12 years of age with NDO or OAB | Completed |
| 178-CL-208 | A phase 1, single dose, 3-period crossover study to assess the bioavailability of an oral suspension of 8 mg/mL mirabegron relative to the oral suspension of 2 mg/mL mirabegron and to assess the effect of food on the pharmacokinetics of the oral suspension of 8 mg/mL mirabegron in healthy male and female adult subjects | Completed |
| 178-CL-206A | An open-label, baseline-controlled, multicenter, phase 3 dose-<br>titration study followed by a fixed dose observation period to<br>evaluate efficacy, safety and pharmacokinetics of mirabegron in<br>children and adolescents from 3 to less than 18 years of age with<br>NDO on CIC | Completed |

CIC: Clean Intermittent Catheterization; NDO: neurogenic detrusor overactivity; OAB: overactive bladder; OCAS: oral-controlled absorption system.

The data from Studies 178-CL-201 and 178-CL-202 were used to support the use of tablets in pediatric subjects with a body weight of ≥ 35 kg in this study. For those pediatric subjects that cannot be dosed with tablets because their body weight is < 35 kg or because they cannot swallow the tablets, an oral suspension with a strength of 2 mg/mL was developed. The results of Studies 178-CL-201 and 178-CL-202 were used to support the use of the 2 mg/mL in Study 178-CL-203. With the results of the Study 178-CL-203, it became apparent that with a strength of 2 mg/mL the volume of the doses the patients have to take every day would be too high (up to 44 mL). To overcome this issue, an oral suspension of 8 mg/mL was developed. To support the use of this 8 mg/mL mirabegron oral suspension in pediatric subjects, Study 178-CL-208 was conducted. The study follows a single dose, 3 period, crossover design in healthy adult subjects. Subjects received the following three treatments in random order: 1) 11 mL of 8 mg/mL oral suspension of mirabegron under fasted conditions, 2) 11 mL of 8 mg/mL oral suspension of mirabegron under fed conditions and 3) 44 mL of 2 mg/mL oral suspension of mirabegron under fasted conditions.

The primary objective of Study 178-CL-208 was to assess the relative bioavailability of the 8 mg/mL oral suspension compared to the 2 mg/mL oral suspension under fasted conditions.

Sponsor: APGD ISN/Protocol: 178-CL-204 EudraCT number 2016-001767-37


The results of Study 178-CL-208 show that the bioavailability of both strengths is comparable [Table 4].

Table 4 Study 178-CL-208 Results: Relative Bioavailability of the Mirabegron 8 mg/mL Oral Suspension Formulation versus 2 mg/mL Oral Suspension Formulation (Pharmacokinetics Analysis Set)

| Parameter (units) | Geometric LS Mean for<br>8 mg/mL Suspension<br>Fasted<br>(n = 24) | Geometric LS Mean for<br>2 mg/mL Oral Suspension<br>Fasted<br>(n = 23) | Geometric LS<br>Mean Ratio<br>(%)† | 90% CI of<br>Ratio (%)† |
|---|---|---|---|---|
| AUC <sub>inf</sub> (ng•h/mL) | 253 | 251 | 100.6 | (90.9,<br>111.3) |
| AUC <sub>last</sub> (ng•h/mL) | 234 | 232 | 100.9 | (90.6,<br>112.4) |
| C <sub>max</sub> (ng/mL) | 12.1 | 11.3 | 106.7 | (84.2,<br>135.2) |

LS: least squares

The analysis was performed on logarithm-transformed pharmacokinetic parameters using a linear mixed model with treatment and investigational period as fixed effects and accounting for the longitudinal nature of the data by subject using a repeated statement. The covariance matrix is structured by period.

† The geometric LS mean ratios (and associated 90% CIs) were obtained by back-transforming (antilogging) the LS means of the treatment differences.

This study demonstrated that 88 mg mirabegron administered as the 8 mg/mL oral suspension formulation was bioequivalent to 88 mg mirabegron administered as the 2 mg/mL oral suspension formulation. An effect of food in line with the literature data for 50 mg mirabegron prolonged-release tablets was observed for the 8 mg/mL mirabegron oral suspension formulation.

Study 178-CL-206A was a phase 3, 52-week, open-label, baseline-controlled, dose-titration multicenter study evaluating the efficacy and safety of mirabegron tablets and oral suspension (8 mg/mL) in 86 pediatric patients with NDO using clean intermittent catheterization (CIC), including 55 children aged 3 to < 12 years and 31 adolescents aged 12 to < 18 years. Patients received mirabegron tablets or oral suspension once daily for up to 52 weeks, starting at pediatric equivalent dose 25 mg (PED25) and up-titrated to pediatric equivalent dose 50 mg (PED50).

This study showed a statistically significant improvement that was present at week 4 and sustained throughout the efficacy treatment period. Secondary and sensitivity analyses of the primary endpoint confirmed the primary analysis. Mirabegron appeared to be safe and well tolerated by pediatric patients with NDO under the condition of Study 178-CL-206A.

The detailed results of Studies 178-CL-201, 178-CL-202, 178-CL-203, 178-CL-208 and 178-CL-206A are reported in the Investigator's Brochure.

The doses described in [Section 2.1.2.2 Clinical Data] suggest tablets for subjects with a body weight of  $\geq$  35 kg unless unable to swallow tablets and would be provided the oral suspension as an alternative, and the 8 mg/mL oral suspension for subjects with a body weight  $\leq$  35 kg.

11 Feb 2021 Astellas 

Sponsor: APGD EudraCT number 2016-001767-37 - CONFIDENTIAL - ISN/Protocol: 178-CL-204

## Safety and Tolerability

In Study 178-CL-203 the safety and tolerability of the oral suspension when dosed in children was evaluated and it was concluded that it was safe and well tolerated.

From the 9 subjects who completed the study (6 with NDO and 3 with OAB) 1 treatment emergent adverse event (TEAE) was reported: pyrexia on day 1 in an NDO subject. The intensity was mild and was judged by the investigator not to be related to study drug. No clinically significant electrocardiogram (ECG) abnormalities have been seen throughout the study, there were no QT interval using Fridericia's correction formula (QTcF) values > 450 msec and no QT interval prolongation > 30 msec versus baseline was observed (mean of triplicates).

A 24-hour continuous 12-lead ECG recording was recorded in all subjects on a reference day and on the dosing day. The main objective of the continuous 12-lead ECG recording was to evaluate the effect of mirabegron on heart rate in a time-matched manner, taking into account the circadian rhythm. A median increase in 24-hour heart rate of 5.1 bpm was observed. This was not considered as clinically relevant due to the multiple blood draws, the low number of subjects and the absence of a placebo treatment group.

Some changes in laboratory values were observed, but they were not considered as clinically relevant.

For Study 178-CL-208 single doses of 88 mg mirabegron oral suspension to adults were safe and well tolerated. Eleven of 24 subjects reported 22 adverse events (AEs). All except for 2 events (1 headache moderate and 1 dysmenorrhea moderate) were mild. Twenty AEs were considered not related; 2 were considered possibly related (dizziness, mild and orthostatic dizziness mild).

For study 178-CL-206A mirabegron tablets and oral suspension (8 mg/mL) once daily for up to 52 weeks, starting at PED25 and up-titrated to PED50 was generally well tolerated by pediatric patients in the completed clinical study. One of 86 (1.2%) patients (an adolescent) reported bradycardia. Using Fleming et al [2011], 3 of 50 (6.0%) children and 2 of 28 (7.1%) adolescents had potentially clinically relevant pulse rate readings during the study. Only 1 of 78 (1.3%) patients (a child) met the criteria for a TEAE of hypertension which was considered not related to the study drug by the investigator.

There were no clinically significant vital signs, clinical laboratory value or 12-lead ECG findings. Based on the mean visual analogue scale score for palatability, the suspension was acceptable in pediatric population and did not require further taste adjustment. The oral suspension when dosed in children was considered to be safe and well tolerated.

# 2.1.3 Summary of Key Safety Information for Investigational Product(s)

Mirabegron has not been approved or marketed for use in pediatric subjects.

Detailed reference safety information (RSI) can be found in the Investigator's Brochure for mirabegron.


Mirabegron has been approved in more than 81 countries worldwide. In adults, the safety of mirabegron treatment has been well characterized in 5863 subjects (95% with OAB) in the phase 2/3 registration studies treated with mirabegron at doses ranging from 25 to 200 mg once daily. Identified risks include increased heart rate and tachycardia, hypersensitivity reactions, increased blood pressure and urinary retention. Potential risks include QT prolongation, urinary tract infection (UTI), fetal disorders after exposure during pregnancy and events induced by concomitant treatment with cytochrome P450 2D6 (CYP2D6) substrates with a narrow therapeutic index. The risks of QT prolongation, increased heart rate or increased blood pressure are greater with increasing exposure at supratherapeutic doses and can be mitigated with optimal dose selection. The maximum therapeutic dose of mirabegron based on the overall benefit-risk is 50 mg once daily in adults.

ISN/Protocol: 178-CL-204

# 2.2 Study Rationale

OAB is recognized by the International Children's Continence Society (ICCS) [Austin et al, 2014], this study is intended to assess the effects of mirabegron in pediatric patients with OAB to understand its potential role in therapy. This study (Study 178-CL-204) is part of the sponsor's clinical program to develop mirabegron for OAB in pediatric subjects. In the EU, the development of mirabegron for the indication of OAB is outlined in the pediatric investigational plan (PIP) for mirabegron and has been approved by the Pediatric Committee. This study is part of PIP commitment.

# 2.3 Risk-Benefit Assessment

This study will be conducted as a double-blind, randomized, multicenter, parallel group, placebo-controlled sequential dose titration study in pediatric subjects from 5 to < 18 years of age with OAB.

The study design and dose rationale are presented in [Section 4 Study Design and Dose Rationale].

Mirabegron tablets have been approved for the indication of OAB in adult subjects. Mirabegron oral suspension has been shown to be safe and well tolerated in 2 phase 1 studies in healthy adult subjects (Studies 178-CL-201 and 178-CL-208). In the pediatric phase 1 studies executed thus far, mirabegron tablets and mirabegron oral suspension had an acceptable safety profile and were well tolerated. Given the available data on mirabegron in the adult population and in the pediatric population to date, the risk-benefit attributes are well defined and can be managed through ongoing safety assessments throughout study conduct as defined in the Schedule of Assessments [Table 1].

The important identified and potential risks in adults are recognized as potential drug safety risks for this study (Study 178-CL-204). These risks will be monitored on a regular basis and can be mitigated as follows:

 The initial dose of mirabegron will be based on the subject's body weight and is predicted to achieve plasma concentrations equivalent to the steady-state exposures Sponsor: APGD ISN/Protocol: 178-CL-204 EudraCT number 2016-001767-37


expected with 25 mg mirabegron administered once daily in adults (PED25). This low dose is chosen considering possible beta-adrenergic side effects of mirabegron.

- At visit 5/week 4 (i.e., after 4 weeks on PED25), dose up-titration to PED50 will be performed unless the investigator determines that the subject is adequately treated for OAB at the PED25 dose or if there are safety concerns identified and considered associated with the use of PED25. Dose down-titration from PED50 to PED25 can be done at any time thereafter for safety reasons. By striving to get an efficacious dose of mirabegron early after start of dosing, the risk for bladder and kidney damage is mitigated.
- Potential fetal disorders after exposure during pregnancy is mitigated by the inclusion criteria
- Hypersensitivity reactions (immediate or nonimmediate and cutaneous or noncutaneous) will be monitored by AE monitoring and will require discontinuation of study treatment
- Potential UTI will be monitored by urinalysis at each visit in the clinic
- Increased blood pressure will be monitored by at-home and clinic measurements and can be mitigated by dose titration
- Increased heart rate and tachycardia will be monitored by at-home and clinic measurements and can be mitigated by dose titration
- Potential QT prolongation will be monitored by ECG at each visit at the clinic and can be mitigated by dose titration
- Potential events by concomitant treatment with CYP2D6 substrates with narrow therapeutic index is mitigated by excluding these medications

For activation of thermogenesis in brown fat, weight loss will be monitored by regular body weight measurements and the potential activation of thermogenesis will be monitored by body temperature measurements.

For both the tablet and the oral suspension formulation, all excipients are pharmaceutical grade materials and are considered safe for the intended pediatric population. Their concentrations remain below the acceptable daily intake as set by the joint Food and Agriculture Organization (FAO) of the UN and the WHO (joint FAO/WHO Expert Committee on Food Additives, 2015).

The protocol is designed to monitor safety and mitigate risk to the pediatric subject by optimizing the number of vital signs, ECG and post void residual (PVR) volume assessments, minimizing the number of blood draws (safety and pharmacokinetic sampling) and focusing the number of study visits.

The use of population pharmacokinetics for the analysis of the pharmacokinetic profile of mirabegron allows reduction of the number of blood draws for pharmacokinetic analysis to 2. Butterfly needles can be used and are allowed to stay in place to reduce the number of punctures.

The blood draws for clinical laboratory tests have been minimized to lessen subject burden while ensuring subject safety. Additional hematology and biochemistry tests will be performed at visit 3/week 0 (baseline) and visit 8/week 14 (end of study [EoS]) only if an AE

11 Feb 2021 Astellas 

Sponsor: APGD ISN/Protocol: 178-CL-204 EudraCT number 2016-001767-37


related to hematology, biochemistry or urinalysis parameters occurred since the previous visit or at the discretion of the investigator.

The assessments to be performed are routine assessments and generally do not pose any particular risk to the subjects. Every effort will be made to reduce the anxiety felt by subjects, e.g., during a blood test, topical anesthetic will be offered at venipuncture to minimize distress of the subject.

Subjects may experience AEs associated with the assessments performed during the study, such as local irritations due to ECG recording, and bleeding, hematoma as a result of blood collection, or the experience of transient stinging or burning during emptying or of the passing of a little blood as a result of the urodynamic investigation. There is also a small risk of developing a bladder infection in relation to the urodynamic procedure.

An independent Data and Safety Monitoring Board (DSMB) will be established [Section 10.4 Study Organization]. A separate charter will describe the responsibilities of the DSMB.

# 3 STUDY OBJECTIVE(S) AND ENDPOINT(S)

The primary, secondary and exploratory objectives and endpoints for this study are listed in [Table 5]. Primary and secondary objectives and endpoints apply to children only; exploratory objectives and endpoints also apply to adolescents.

Table 5 Study Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| • To evaluate the efficacy of mirabegron in children (5 to < 12 years of age) with OAB | <ul> <li>Change from baseline at the end of the 12-week treatment period:</li> <li>Mean number of micturitions per 24 hours</li> </ul> |
| Secondary | 1 |
| To evaluate the efficacy of mirabegron in<br>children (5 to < 12 years of age) with OAB | Change from baseline at the end of the 12-week treatment period: |
| | <ul> <li>Mean volume voided per 24 hours</li> </ul> |
| | <ul> <li>Maximum volume voided</li> </ul> |
| | <ul> <li>Mean number of daytime incontinence<br/>episodes per 24 hours</li> </ul> |
| | <ul> <li>Mean number of nighttime incontinence<br/>episodes per 24 hours</li> </ul> |
| | <ul> <li>Mean number of daytime micturitions per</li> <li>24 hours</li> </ul> |
| | • Number of dry (incontinence-free) days per 7 days at the end of the 12-week treatment period |
| Table continued on next page | |

Sponsor: APGD ISN/Protocol: 178-CL-204

EudraCT number 2016-001767-37


| Objectives | Endpoints |
|---|---|
| To evaluate the safety and tolerability of mirabegron in pediatric subjects with OAB | <ul> <li>Nature, frequency and severity of AEs</li> <li>Clinical laboratory tests (hematology, biochemistry and urinalysis)</li> <li>Vital signs (blood pressure and pulse)</li> <li>Routine 12-lead ECG</li> <li>PVR volume</li> <li>Acceptability and palatability questionnaire</li> </ul> |
| To evaluate the pharmacokinetics after multiple<br>dose administration of mirabegron in pediatric<br>subjects with OAB | Steady-state C <sub>max</sub> , AUC <sub>tau</sub> , C <sub>trough</sub> , T <sub>max</sub> , CL/F and Vz/F. Additional parameters may be calculated based on the population pharmacokinetic model used |
| Exploratory | |
| To evaluate the efficacy of mirabegron in pediatric subjects (5 to < 18 years) with OAB | <ul> <li>Percentage of subjects with a reduction in daytime incontinence episodes (&lt; 50% reduction [nonresponder], 50% [partial responder] and 100% [responder])</li> <li>Improvement from baseline in worst incontinence grading</li> <li>Change from baseline at the end of the 12-week treatment period adjusted for fluid intake: <ul> <li>Mean number of micturitions per 24 hours</li> </ul> </li> <li>Change from baseline at the end of the 12-week treatment period (adolescents only): <ul> <li>Mean number of micturitions per 24 hours</li> <li>Mean number of daytime micturitions per 24 hours</li> <li>Mean volume voided per 24 hours</li> <li>Mean number of incontinence episodes per 24 hours</li> </ul> </li> <li>Number of dry (incontinence-free) days per 7 days at the end of the 12-week treatment period (adolescents only)</li> <li>Mean number of daytime grade 3 or 4 (PPIUS) urgency episodes per 24 hours (adolescents only)</li> </ul> |

AE: adverse event; ECG: electrocardiogram; OAB: overactive bladder; PPIUS: patient perception of intensity of urgency scale; PVR: post void residual.

## 3.1 Estimand

The estimand of most clinical importance for this study is defined by the following 4 attributes:

- Target population: all children who took at least 1 dose of the study drug, and in whom a nonmissing measurement for micturition frequency at baseline and after administration of the study drug is available
- Outcome measurement: micturition frequency/day (24 hours)
- Intercurrent events:
  - 1. Discontinuation from treatment (if week 12/EoT not obtained)
  - 2. AE UTI (if occurred in week 12/EoT)

Sponsor: APGD ISN/Protocol: 178-CL-204

EudraCT number 2016-001767-37


3. Other muscarinic antagonists or botulinum toxin see [Appendix 12.6 List of Excluded Concomitant Medications]) (if taken during the last 2 weeks prior to week 12/EoT assessment); in all cases, a hypothetical strategy will be applied

• Population-based summary: Change from baseline to week 12/EoT in micturition frequency/day (= primary endpoint, primary estimator), compared to placebo

For this placebo-controlled study, this "de jure" estimand chosen is considered the appropriate choice. As some effect is expected early in the study and with continued treatment could be expected to be maintained, it's considered appropriate to impute for subjects with missing values at visit 7/week 12/EoT by their last recorded post baseline visit value prior to it. This strategy also assumes that the responses after the intercurrent event would be same as for patients continuing on their respective treatment.

# 4 STUDY DESIGN AND DOSE RATIONALE

# 4.1 Study Design

This is a double-blind, randomized, multicenter, parallel group, placebo-controlled sequential dose titration study to evaluate efficacy, safety and pharmacokinetics of mirabegron in pediatric subjects with OAB. Male and female pediatric subjects 5 to < 18 years of age with OAB; as defined according to the ICCS [Austin et al, 2014] who have had received 4 weeks of urotherapy prior to randomization.

Planned total number of study sites includes approximately 65 study sites across Europe, Latin America, Africa, Middle East, Asia-Pacific and North America.

The study consists of 3 periods with a total duration of 18 weeks.

• Screening period/urotherapy (4 weeks):

This period starts with visit 1/week -4 (screening) and ends with visit 3/week 0 (baseline). After informed consent/assent has been obtained and immediately after eligibility has been confirmed at visit 1/week -4 (screening), subjects using prohibited medication will complete 1 week of washout (if applicable), while beginning 4 weeks of urotherapy.

After a successful screening visit (visit 1/week -4 [screening]), all subjects will need to complete a 2-day bladder e-diary (weekend) to get acquainted with the bladder e-diary and the assessments. Completion of this bladder e-diary should start in the weekend prior to visit 2. All subjects will also complete a 7-day bladder e-diary the week prior to the baseline visit. The 7-day diary will consist of a 5-day weekday bladder e-diary and 2-day weekend e-diary.

• Double-blind, placebo-controlled period (12 weeks):

This period starts with the day after visit 3/week 0 (baseline) and ends with visit 7/week 12 (EoT).

At visit 3/week 0 (baseline), inclusion and exclusion criteria will be evaluated. Subjects continuing urotherapy who still meet the OAB entry criteria at baseline will be

Sponsor: APGD ISN/Protocol: 178-CL-204 EudraCT number 2016-001767-37


randomized. Subjects whose symptoms are not satisfactorily controlled with urotherapy and still fulfill the inclusion/exclusion criteria will enter the study. These subjects will be randomized to receive mirabegron in PED25 or placebo using a 1:1 ratio. Subjects with a body weight of  $\geq$  35 kg are to receive the tablet unless unable to swallow tablets and would be provided the oral suspension as an alternative. Subjects with a body weight < 35 kg or those who cannot be dosed with the tablet will receive an oral suspension. Daily investigational product (IP) administration will start on day 1 (i.e., the day after this visit) and continue at this dose until visit 5/week 4 (i.e., for 4 weeks). Urotherapy will continue throughout the study treatment period until visit 7/week 12 (EoT).

At visit 5/week 4, dose up-titration to mirabegron in PED50 will be performed unless the investigator determines that the subject is adequately treated for OAB at the PED25 dose or if there are safety concerns identified and considered associated with the use of PED25. Dose down-titration from PED50 to PED25 can be done at any time thereafter for safety reasons.

Subjects will start with the subsequent 7-day bladder e-diaries approximately 7 days prior to the indicated visit (or TC).

Pharmacokinetic blood samples will be collected at visit 5/week 4 and visit 7/week 12 (EoT) as indicated in the Schedule of Assessments [Table 1].

# • Follow-up period (2 weeks):

This period starts the day after visit 7/week 12 (EoT) and ends with visit 8/week 14 (EoS). The follow-up period is applicable to all subjects who have been randomized and received IP.

At visit 7/week 12 (EoT), IP administration will be stopped and a safety observation period of 2 weeks will start.

An independent DSMB will be established. A separate charter will describe the responsibilities of the DSMB.

A blinded interim analysis will be performed after 50% of children planned to be randomized have had their week 12/EoT assessment. The interim analysis will determine if the chance of a positive study with respect to the primary endpoint at the EoS is high enough to justify continuation of the study; otherwise, the study will be stopped for futility.

The IP will not be provided after study completion without written approval from the sponsor.

## 4.2 Dose Rationale

The target exposures of 69 and 188 ng•h/mL for PED25 and PED50 were derived from the adult phase 3 program and are the mean steady-state area under plasma concentration-time curve over dosing interval (AUC<sub>tau</sub>) values following 25 and 50 mg prolonged-release tablets once daily in adults.


A population pharmacokinetic model was used to predict the pediatric equivalent dose for subjects in Study 178-CL-204. In brief, this population pharmacokinetic model was developed on adult phase 3 data, and allometric (weight-based) scaling was added to all clearance and volume terms to allow for scaling of the pharmacokinetics to pediatric subjects. The model was validated on pediatric data in Study 178-CL-202 (single ascending-dose study) and was shown to appropriately predict the pharmacokinetics of mirabegron in pediatric subjects.

ISN/Protocol: 178-CL-204

Simulations were then performed to determine a body weight at which subjects would have steady-state exposures comparable to those in adults when dosed with 25 or 50 mg daily; this weight was determined to be  $\geq$  35 kg. Based on prior experience obtained in an ongoing Astellas study in another program in patients with NDO (Study 905-CL-047) the average age at which children reach a body weight of 35 kg is approximately 11 years. The dosing recommendation based on this modeling is in line with the literature [Momper et al, 2013] in which a meta-analysis of compounds submitted to the US FDA with a similar indication in adults and adolescents showed that in almost all cases, the adolescents required the same dose as the adults.

Therefore, subjects with a body weight of  $\geq 35$  kg can be dosed with mirabegron tablets unless unable to swallow tablets and would be provided the oral suspension as an alternative. Subjects with a body weight < 35 kg cannot be dosed with the 25 and 50 mg tablets because that would exceed the target exposures. Subjects with a body weight < 35 kg will therefore be dosed with mirabegron oral suspension.

Mirabegron oral suspension (8 mg/mL) has been developed for use in the pediatric population. The population pharmacokinetic model referred to above includes a formulation factor to account for the different (lower) relative bioavailability of the oral suspension compared to the tablet. This factor has been used in simulations to predict the suspension doses and weight categories that would have a reasonable variance around the target exposures.

For dosing with oral suspension, the weight range to be covered is from 13 kg (the approximate body weight of a 5-year-old child, according to the National Health and Nutrition Examination Survey database [McDowell et al, 2008]) to 35 kg (above which pediatric subjects could be dosed with the tablet formulation). Subjects with a body weight < 13 kg will not be included in the study. Suspension dosing for body weights  $\ge 35$  kg was also determined for cases in which a pediatric subject in that weight category who cannot be dosed with the tablets. The simulation resulted in the 3 body weight categories that can be found in the dosing schedule (see [Table 7]).

# 4.3 End of Study Definition

The study start is defined as the date the first subject and/or the subject's parent(s)/legal guardian(s) sign(s) informed consent/assent. End of the study is defined as the last visit or scheduled procedure shown in the Schedule of Assessments [Table 1] for the last subject in the study.
#### ISN/Protocol: 178-CL-204

## 5 STUDY POPULATION

All screening assessments must be completed and reviewed to confirm the potential subject meets all eligibility criteria. Prospective approval of protocol deviations to eligibility criteria (also known as protocol waivers or exemptions) is not permitted.

### 5.1 Inclusion Criteria

Subject is eligible for the study if all of the following apply:

### Inclusion at Visit 1/Week -4 (Screening)

- 1. Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved written informed consent/assent and privacy language as per national regulations (e.g., General Data Protection Regulations for European Union study sites) must be obtained from the subject and/or from the subject's parent(s)/legal guardian(s) prior to any study-related procedures (including withdrawal of prohibited medication, if applicable); assent by the subject is obtained as required by local law.
- 2. Subject has OAB defined according to the ICCS criteria.
- 3. Subject is a male or female between 5 to < 18 years of age, at screening.
- 4. Subject weighs at least 13 kg at screening.
- 5. Subject is able to take the IP in accordance with the protocol.
- 6. Subject agrees to drink an adequate fluid volume during urine collection weekends, as instructed by the investigator.
- 7. Subject and subject's parent(s)/legal guardian(s) agree that the subject will not participate in another interventional study while participating in the present study.
- 8. Subject and subject's parent(s)/legal guardian(s) are willing and able to comply with the study requirements and with the concomitant medication restrictions.
- 9. Female subject is not pregnant (see [Appendix 12.3 Contraception Requirements]) and at least 1 of the following conditions apply:
  - a. Not a female of childbearing potential (see [Appendix 12.3 Contraception Requirements]).
  - b. Female of childbearing potential who agrees to follow the contraceptive guidance (see [Appendix 12.3 Contraception Requirements]) from the time of informed consent/assent through at least 30 days after final IP administration.
- 10. Female subject must agree not to breastfeed starting at screening and throughout the study period and for 30 days after final IP administration.
- 11. Female subject must not donate ova starting at first dose of IP and throughout the study period and for 30 days after final IP administration.
- 12. Male subject with female partner(s) of childbearing potential (including breastfeeding partner[s]) must agree to use contraception (see [Appendix 12.3 Contraception Requirements]) throughout the treatment period and for 30 days after final IP administration.
- 13. Male subject must agree not to donate sperm during the treatment period and for 30 days after final IP administration.

Sponsor: APGD - CONFIDENTIAL -

EudraCT number 2016-001767-37

14. Male subject with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 30 days after final IP administration.

ISN/Protocol: 178-CL-204

### Additional Inclusion at Visit 3/Week 0 (Baseline)

- 15. Subject must have a micturition frequency of at least 8 times (on average) per day, in the 7 days prior to visit 3/week 0 (baseline), as recorded in the bladder e-diary.
- 16. Subject must have at least 1 daytime incontinence episode (on average) per day, during the 7-day period before visit 3/baseline, as recorded in the bladder e-diary.
- 17. Subject whose symptoms are not satisfactorily controlled with urotherapy and still fulfills the inclusion/exclusion criteria will enter the study.

#### 5.2 **Exclusion Criteria**

Subject will be excluded from participation in this study if any of the following apply:

### Exclusion at Visit 1/Week -4 (Screening)

- 1. Subject has extraordinary daytime only urinary frequency according to the ICCS definition.
  - This applies to a toilet-trained child who has the frequent need to void that is associated with small micturition volumes solely during the day.
  - The daytime voiding frequency is at least once per hour with an average voided volume of < 50% of expected bladder capacity (EBC) (typically 10% to 15%).
  - Incontinence is rare and nocturia is absent.
- Subject has an uroflow indicative of pathology other than OAB.
- Subject has monosymptomatic enuresis.
- Subject has dysfunctional voiding.
- Subject has bladder outlet obstruction, except if successfully treated.
- Subject has anatomical anomalies (surgically treated or untreated) that affect lower urinary tract function.
- Subject with hematuria on dipstick test. In the case of hematuria on dipstick test in a female during menstruation, the test can be repeated before randomization (after the end of menstruation).
- Subject with diabetes insipidus.
- Subject has kidney or bladder stones.
- 10. Subject has suffered from chronic UTI or has had more than 3 UTIs in the 2 months prior to visit 1/week -4 (screening).
- 11. Criterion has been removed.
- 12. Subject has stage 2 hypertension or subject has stage 1 hypertension that is not well controlled, as defined by the 2017 American Academy of Pediatrics Clinical Practice Guidelines.
- 13. Subject has QTcF > 440 msec on screening ECG, a risk of QT prolongation (e.g., hypokalemia, long QT syndrome [LQTS] or family history of LQTS or exercise-induced syncope) or is currently taking medication known to prolong the QT interval.


14. Subject's aspartate aminotransferase (AST) or alanine aminotransferase (ALT) is  $\geq$  2 × upper limit of normal (ULN) or total bilirubin (TBL) is  $\geq$  1.5 × ULN according to age and sex (subjects with Gilbert's syndrome are excepted from the bilirubin threshold).

ISN/Protocol: 178-CL-204

- 15. Subject has mild or moderate renal impairment (estimated glomerular filtration rate according to the modified Schwartz of < 60 mL/min per 1.73 m<sup>2</sup>).
- 16. Subject has a symptomatic (symptoms can include pain, fever, hematuria, new onset foul-smelling urine) UTI. Note: if the UTI is treated successfully (clinical recovery: confirmed by dipstick test and repeated dipstick test after 14 days [both should be negative]), the subject can be rescreened.
- 17. Subject has a history or presence of any malignancy.
- 18. Subject uses any drugs that are sensitive cytochrome P450 2D6 (CYP2D6) substrates with a narrow therapeutic index, sensitive P-glycoprotein (P-gp) substrates, or moderate or strong cytochrome CYP3A4/5 or P-gp inhibitors or inducers after the start of washout.
- 19. Subject is using or has used prohibited prior and/or concomitant medication(s) [Appendix 12.6 List of Excluded Concomitant Medications] that cannot be discontinued.
- 20. Subject has known or suspected hypersensitivity to mirabegron or any components of the formulations used.
- 21. Subject has participated in another clinical study (and/or subject has received any investigational therapy within 30 days (or 5 half-lives of the drug, or the limit set by national law, whichever is longer) prior to visit 1/week -4 (screening).
- 22. Subject received urinary catheterization within 2 weeks prior to screening.
- 23. Subject has constipation as defined by the Rome IV criteria that cannot be successfully treated prior to study entry.
- 24. Female subject who has been pregnant within 6 months prior to screening or breastfeeding within 3 months prior to screening.
- 25. Subject has any condition, which in the opinion of the investigator, makes the subject unsuitable for study participation.

### Additional Exclusion at Visit 3/Week 0 (Baseline)

- 26. Subject has extraordinary daytime only urinary frequency according to the ICCS definition based on the bladder e-diary.
- 27. Subject has monosymptomatic enuresis confirmed by the bladder e-diary.
- 28. Subject has a maximum voided volume (morning volume excluded) > EBC for age ([age +1]  $\times$  30) in mL, based on the bladder e-diary.
- 29. Subject has polyuria defined as voided urine volumes of > 40 mL/kg baseline body weight during 24 hours or > 2.8 L urine for a child weighing  $\ge 70$  kg (ICCS definition) [Austin et al, 2014], based on bladder e-diary.
- 30. Subject has PVR volume > 20 mL (lowest PVR volume result) as measured by ultrasonography.
- 31. Subject suffers from a symptomatic (symptoms can include pain, fever, hematuria, new onset foul-smelling urine) UTI. Note: if a symptomatic UTI is present, all visit 3/week 0 (baseline) assessments must be postponed until the UTI is successfully treated (clinical recovery: confirmed by dipstick test and repeated dipstick test after

Sponsor: APGD ISN/Protocol: 178-CL-204 EudraCT number 2016-001767-37


14 days [both should be negative]), and the urotherapy should continue. The postponed visit 3/week 0 (baseline) should be within 14 days of the intended visit 3/week 0 (baseline).

- 32. Subject with hematuria on dipstick test. In the case of hematuria on dipstick test in a female during menstruation, the test can be repeated before randomization (after the end of menstruation).
- 33. Subject has a pulse > 99<sup>th</sup> percentile for age.
- 34. Subject has stage 2 hypertension or subject has stage 1 hypertension that is not well controlled, as defined by the 2017 American Academy of Pediatrics Clinical Practice Guidelines.
- 35. Any reason, in the opinion of the investigator, that makes the subject unsuitable for study participation.

# 5.3 Restrictions During the Study

Restrictions for foods and drinks are not applicable. On visit days where a pharmacokinetic sample is planned in the clinic, dosing should occur in the clinic and breakfast should be eaten at the clinic within 1 hour before dosing.

### 5.4 Screen Failures

A screen failure is defined as a potential subject who signed the informed consent form (ICF)/assent and/or whose parent(s)/legal guardian(s) signed the ICF/assent, but did not meet 1 or more criteria required for participation in the study and was not enrolled.

For screen failures, the demographic data, date of signing the ICF/assent, inclusion and exclusion criteria, AEs up to the time of screen failure and reason for screen failure will be collected in the electronic data source. Rescreening is only allowed once for an individual subject.

### 5.4.1 Rescreen

### 5.4.1.1 Rescreen for Urinary Tract Infection or Constipation

In addition, if a subject has UTI/constipation at visit 3/week 0 (baseline), all visit 3/week 0 (baseline) assessments must be postponed until the UTI/constipation is successfully treated (clinical recovery), and the urotherapy should continue. Then the subject's postponed visit 3/week 0 (baseline) assessments should be completed within 14 days of the intended visit 3/week 0 (baseline) or the subject will be documented as a screen failure and can be re-screened. If the postponed visit 3/week 0 (baseline) is rescheduled within 14 days of the intended visit 3/week 0 (baseline) visit, then the subject's 7-day e-diary will be restarted with respect to the postponed visit 3/week 0 (baseline) visit.

### 5.4.1.2 Rescreen for Other Eligibility Criteria

Results of screening assessments that do not meet the parameters required by eligibility criteria (e.g., clinical laboratory tests, vital signs, physical examination, ECG, etc.) may be repeated once within the 4-week screening period without the need to register the subject as a screen failure. If any exclusion criteria are met or more than 4 weeks elapse from the date of signing the ICF/assent, the subject must be documented as a screen failure. In order to

11 Feb 2021 Astellas 


rescreen a subject previously registered as a screen failure, a new ICF/assent must be signed and the subject will be entered into screening with a new subject identification number. The old subject number will also be entered to link the subject's data.

ISN/Protocol: 178-CL-204

# 6 INVESTIGATIONAL PRODUCT(S) AND OTHER STUDY TREATMENT(S)

# 6.1 Investigational Product(s) Administered and Other Study Treatment(s)

### **6.1.1** Investigational Product(s)

Mirabegron prolonged-release (or extended-release) tablets were approved in Japan in 2011, and to date have been approved in more than 81 countries worldwide; trade names include Betanis® [BETANIS® prescribing information, Jun 2012], Betmiga® [BETMIGA® prescribing information, Apr 2018] and Myrbetric® [MYRBETRIC® prescribing information, Jun 2012]. The approved indication is the treatment of OAB with symptoms of urge urinary incontinence, urgency and urinary frequency in adults.

Mirabegron oral suspension has been developed as an appropriate formulation for weight-based dosing in smaller children.

Sponsor: APGD

ISN/Protocol 178-CL-204

EudraCT number 2016-001767-37


 Table 6
 Investigational Product(s)

| Name | Mirabegron | Matching Placebo | Mirabegron | Matching Placebo |
|---|---|---|---|---|
| Use | Test product | Placebo | Test product | Placebo |
| Dosage Formulation | Tablet | Tablet | Oral suspension | Oral suspension |
| Physical Description | Brown (25 mg) or yellow (50 mg) film-coated tablet | Brown (25 mg) or yellow (50 mg) film-coated tablet | Yellowish white granules reconstituted with water to prepare oral suspension | Yellowish white granules reconstituted with water to prepare oral suspension |
| <b>Unit Dose Strength</b> | 25 and 50 mg | To match mirabegron | 8 mg/mL | To match mirabegron |
| Packaging and Labeling | -35 tablets of Mirabegron 25 mg<br>in a wallet<br>-35 tablets of Mirabegron 50 mg<br>and 7 tablets of Mirabegron 25<br>mg in a wallet | 35 tablets of Mirabegron 25 mg<br>placebo in a wallet<br>-35 tablets of Mirabegron 50 mg<br>placebo and 7 tablets of<br>Mirabegron 25 mg placebo in a<br>wallet | 1 bottle of Mirabegron 830 mg<br>granules for oral suspension | 1 bottle of placebo Mirabegron<br>830 mg granules for oral<br>suspension |
| <b>Route of Administration</b> | Oral | Oral | Oral | Oral |
| Administration Instruction | IP will be administered orally, once daily in the morning around the same time of day and around time of food intake (i.e., within 1 hour before or after breakfast). Tablets will be administered with a sip of water (tablet should be taken as a whole and should not be chewed, divided or crushed). | | IP will be administered orally, once daily in the morning around the same time of day and around time of food intake (i.e., within 1 hour before or after breakfast). Oral suspension will be administered via an oral syringe with a sip of water afterwards. Detailed information on the preparation of the mirabegron oral suspension will be provided to the subject and subject's parent(s)/legal guardian(s) in local language. | |
| IMP or Non-IMP | IMP | IMP | IMP | IMP |
| Sourcing | Provided centrally by sponsor | Provided centrally by sponsor | Provided centrally by sponsor | Provided centrally by sponsor |

IMP: investigational medicinal product; IP: investigational product


For detailed information on mirabegron prolonged-release tablets, please refer to the current locally-available product information for mirabegron. For detailed information on mirabegron granules for oral suspension, please refer to the Investigator's Brochure and Investigational Medicinal Product Dossier.

ISN/Protocol: 178-CL-204

IP will be administered according to [Table 7].

Table 7 Body Weight-based Doses for Tablets or Suspension

| | Body Weight Range†<br>(kg) | Oral Suspension Volume‡ (mL) | Tablet Dose (mg) |
|---|---|---|---|
| | 13 to < 22 | 3 | - |
| PED25 | 22 to < 35 | 4 | - |
| | ≥ 35 | 6 | 25 |
| | 13 to < 22 | 6 | - |
| PED50 | 22 to < 35 | 8 | - |
| | ≥ 35 | 11 | 50 |

PED25: pediatric equivalent dose 25 mg; PED50: pediatric equivalent dose 50 mg

The starting dose will be PED25 starting administration the day after visit 3/week 0 (baseline). At visit 5/week 4, dose up-titration to PED50 will be performed unless the investigator determines that the subject is adequately treated for OAB at the PED25 dose or if there are safety concerns identified and considered associated with the use of PED25. Dose down-titration from PED50 to PED25 can be done at any time thereafter for safety reasons.

### 6.1.2 Other Study Treatment(s)

During the screening period, all subjects will receive 4 weeks of urotherapy. At visit 3/week 0 (baseline) inclusion and exclusion criteria will be evaluated. Subjects continuing urotherapy who still meet the OAB entry criteria at baseline will be randomized. Urotherapy will continue throughout the study treatment period until visit 7/week 12 (EoT).

Urotherapy is to be discussed and confirmed with the subject or parent(s)/legal guardian(s) during each visit (or TC) to ensure compliance.

Standard urotherapy includes information on and demystification of the voiding function and dysfunction, instruction on voiding habits (such as regular voiding, voiding posture), life style advice regarding fluid intake, prevention of constipation, recording of symptoms and voiding habits in bladder diaries and support via regular follow-up by a caregiver.

Specific interventions include various forms of pelvic floor training (relaxation, contraction), behavioral modification, electrical stimulation, catherization and biofeedback (use of objective measures, e.g., uroflow or EMG to show children how far they relax their pelvic floor during voiding). Urotherapy can also include elements of cognitive behavioral therapy [Nevéus et al, 2006].

<sup>†</sup> Subjects with a body weight ≥ 35 kg will receive the tablet. Subjects with a body weight < 35 kg or those who cannot be dosed with the tablet will receive an oral suspension.

<sup>‡</sup> Oral suspension containing 8 mg/mL.

## Sponsor: APGD ISN/Protocol: 178-CL-204

## 6.2 Preparation/Handling/Storage/Accountability

# 6.2.1 Packaging and Labeling

All IP used in this study will be prepared, packaged and labeled under the responsibility of qualified personnel at Astellas Pharma Europe B.V. (APEB) or sponsor's designee in accordance with APEB or sponsor's designee standard operating procedures (SOPs), Good Manufacturing Practice (GMP) guidelines, International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Good Clinical Practice (GCP) guidelines, and applicable local laws/regulations.

Each IP package will bear a label conforming to regulatory guidelines, GMP and local laws and regulations that identifies the contents as an investigational drug.

A qualified person of APEB or sponsor's designee will perform the final release of the medication according to the requirements of the EU Directive 2003/94/EC annex 13.

### 6.2.2 Handling, Storage and Accountability

- 1. The investigator or designee must confirm appropriate temperature conditions have been maintained during transit for all IP received and any discrepancies are reported and resolved before use of the IP.
- 2. Only subjects enrolled in the study may receive IP and only authorized study site personnel (listed under delegation log) may supply or administer IP. Only IP with appropriate expiry/retest dating may be dispensed.
- 3. All IP must be stored in a secure, environmentally controlled and monitored (manual or automated) area in accordance with the labeled storage conditions and access must be limited to the investigator and authorized study site personnel.
- 4. The investigator, institution or the head of the medical institution (where applicable) is responsible for accountability, reconciliation and record maintenance (i.e., receipt, reconciliation and final disposition records).

The site must return IP to the Sponsor or designee at the EoS or upon expiration. If due to institutional policy or local law, used IP cannot be returned to the Sponsor or designee the IP may be destroyed according to local law.

# 6.3 Randomization and Blinding

### 6.3.1 Blinding Method

This is a double-blind study. Subjects will be randomized to receive mirabegron or placebo in a blinded manner such that neither the investigator, sponsor's study management team, clinical personnel, nor the subject will know which IP is being administered. The randomization number will be assigned based on information obtained from the interactive response technology (IRT) system.

### 6.3.2 Confirmation of the Indistinguishability of the Investigational Product

The appearance of both the dosage form and packaging of mirabegron are identical to those of their matching placebo.

11 Feb 2021 Astellas 


# 6.3.3 Retention of the Assignment Schedule and Procedures for Treatment Code Breaking

The randomization list and treatment assignment blind will be maintained by the IRT system.

ISN/Protocol: 178-CL-204

### 6.3.4 Breaking the Treatment Code for Emergency

The treatment code for each randomized subject will be obtained from the IRT system in the event of a medical emergency requiring knowledge of the treatment assigned to the subject. The IRT system will be programmed with blind-breaking instructions that can only be requested by the investigator or sub investigator(s) designated to have access to perform blind-breaking. In case of a medical emergency, the investigator has the sole responsibility for determining if unblinding of the subject's treatment assignment is warranted. Subject safety must always be the first consideration in making such determination. If the investigator decides that unblinding is warranted, the investigator should make every effort to contact the sponsor prior to unblinding a subject's treatment assignment unless this could delay emergency treatment for the subject.

Prior to the initial IP shipment, the investigator must have confirmed ability to access code-break through the IRT system and must have a designated backup (e.g., redundant processes) to support emergency unblinding requirements.

Prior to randomization, subjects should be provided with information that includes the study site emergency contact number and back-up contact number in case of a medical emergency. Any unblinding by the investigational personnel must be reported immediately to the sponsor and include an explanation of why the IP was unblinded. If unblinding is associated with a serious adverse event (SAE), the investigator is to follow the instructions in [Appendix 12.4.5 Reporting Procedures for Serious Adverse Events].

Care will be taken to limit knowledge of the treatment assignment, in case this can affect the blinding of other subjects or future study assessment for the subject.

### 6.3.5 Breaking the Treatment Code by the Sponsor

The sponsor may break the treatment code for subjects who experience a suspected unexpected serious adverse reaction (SUSAR) in order to determine if the individual case or a group of cases requires expedited regulatory reporting. Individual emergency codes will be provided to the limited personnel who are responsible to break the codes for all SUSAR cases for reporting purposes.

### 6.3.6 Assignment and Allocation

### 6.3.6.1 Subject Number

Subjects will be assigned a subject number at study entry (i.e., signing the ICF/assent). The subject numbers will be sequential and rising. The subject number will comprise of 10 digits; 5 digits for the site number (provided by the sponsor) and 5 digits for the consecutive subject number.


Subjects will be randomized to receive IP according to the randomization schedule obtained via the IRT system. The study site personnel will dispense the treatment according to the IRT system's assignment. Specific procedures for randomization through the IRT system are contained in the study procedures manual.

ISN/Protocol: 178-CL-204

### 6.3.6.2 Randomization Number

Subjects will be randomized in a 1:1 ratio to receive treatment according to the randomization schedule obtained via the IRT system. The study site personnel will dispense the treatment according to the IRT system's assignment. Specific procedures for randomization through the IRT system are contained in the study procedures manual.

### 6.3.6.3 Subject Replacement

An enrolled subject who withdraws or discontinues before dosing or before randomization will be considered a screen failure. Randomized subjects who withdraw or discontinue will not be replaced.

# 6.4 Investigational Product(s) and Other Study Treatment(s) Compliance

### 6.4.1 Investigational Product(s)

Subject compliance with IP and other study treatment(s) will be assessed at each visit. Compliance will be assessed by counting or weighing returned IP at each clinic visit. Deviations from the prescribed dose regimen will be recorded in the electronic data source.

If compliance less than 80%, the investigator or designee is to counsel the subject and/or the subject's parent(s)/legal guardian(s) and ensure steps are taken to improve compliance.

### **6.4.2** Other Study Treatment(s)

Subjects will have to receive 4 weeks of urotherapy prior to randomization and will continue urotherapy throughout the study. Urotherapy is to be discussed and confirmed with the subject or parent(s)/legal guardian(s) during each TC to ensure subject compliance.

Specific interventions include various forms of pelvic floor training (relaxation, contraction), behavioral modification, electrical stimulation, catherization and biofeedback (use of objective measures, e.g., uroflow or surface EMG to show children how far they relax their pelvic floor during voiding). Urotherapy can also include elements of cognitive behavioral therapy [Nevéus et al, 2006].

# 6.5 Previous and Concomitant Treatment (Medication and Nonmedication Therapy)

Subjects are not allowed to use ongoing treatment with any of the following prohibited medications after the start of the washout:

• Any medication, other than the IP, used for the treatment of OAB (including tricyclic antidepressants, 1<sup>st</sup> generation H1 antagonists and alpha blockers)


• Any drugs that are sensitive CYP2D6 substrates with a narrow therapeutic index or sensitive P-gp substrates

- Any medications known to prolong the QT interval
- Any medication that is a moderate or strong cytochrome CYP3A4/5 or P-gp inhibitor or inducers including natural and herbal remedies

ISN/Protocol: 178-CL-204

- Intradetrusor botulinum toxin injections; except if given > 9 months prior screening and symptoms reappeared comparable to those before botulinum toxin injections
- Nonmedication therapies like urotherapy, chiropractic, physical therapy will also be collected on the nonmedication therapy case report form (CRF).
  - The site will need to make special notes for those subjects who do not follow urotherapy for 7 or more consecutive days in electronic case report forms (eCRFs).

Please refer to [Appendix 12.6 List of Excluded Concomitant Medications] for drug classes or specific medications that are prohibited during participation in the study. These treatments are prohibited from being started after the start of the washout period. All other concomitant treatment use will be reported.

The use of previous and concomitant treatment within 30 days prior to signing the informed consent and throughout the study will be documented on the appropriate eCRF.

### 6.6 Dose Modification

At visit 5/week 4 (i.e., after 4 weeks on PED25), dose up-titration to PED50 will be performed unless the investigator determines that the subject is adequately treated for OAB at the PED25 dose or if there are safety concerns identified and considered associated with the use of PED25.

At any time, down-titration from PED50 to PED25 can be performed if there is an AE possibly related to the drug that is considered bothersome by the subject or that leads to medical intervention (e.g., initiation of medication therapy to treat the AE). Of note, PED25 is the lowest dose to be used in this study.

Criteria for discontinuation of individual subject(s) from study treatment are listed in [Section 8.1 Discontinuation of Individual Subject(s) from Study Treatment(s)].

# 6.7 Criteria for Continuation of Treatment(s)

Mirabegron (PED25/PED50) will not be made available after conclusion of the study to subjects who are still receiving and benefitting from study treatment in countries where the product does not have marketing approval and is not commercially available.

### 7 STUDY PROCEDURES AND ASSESSMENTS

Refer to the Alternate Schedule of Assessments [Table 12] in [Appendix 12.13 Clinical Study Continuity] for acceptable alternate methods to assess safety and efficacy parameters in the event the study is interrupted due to a crisis (e.g., natural disaster, pandemic).

Sponsor: APGD ISN/Protocol: 178-CL-204

## 7.1 Efficacy Assessments

## 7.1.1 Bladder Electronic Diary

The bladder diary is part of the subject's e-diary. After a successful visit 1/screening, all subjects start with the completion of a 2-day weekend e-diary to get acquainted with the e-diary and the assessments. Completion of this diary should start in the weekend prior to visit 2.

The e-diary data is reviewed by the investigator or designee prior to the start of visit 2 and discussed and confirmed with the subject or the subject's parent(s)/caregiver(s) during the (telephone) visit 2. If the investigator is under the impression that the subject and/or the subject's parent(s)/caregiver(s) can perform all the required assessments and are able to complete all required forms with credible data, completion is considered successful.

If successful completion of the 2-day weekend e-diary is confirmed at visit 2, subjects will start with collection of the 7-day bladder e-diary approximately 7 days prior to visit 3/week 0 (baseline). The 7-day bladder e-diary consists of a 5-day weekday bladder e-diary, which is used to collect micturition frequency and incontinence episodes; the remaining consists of the 2-day weekend diary.

After successful randomization, subsequent bladder e-diaries will be completed by the subject or subject's parent(s)/caregiver(s) in the week prior to visit 4/week 2, visit 5/week 4, visit 6/week 8 and visit 7/week 12. Completion of 7-day bladder diaries should start approximately 7 days prior to the indicated visit (or telephone contact).

# 7.2 Safety Assessments

### 7.2.1 Adverse Events

See [Section 7.3 Adverse Events and Other Safety Aspects] for information regarding AE collection and data handling.

### 7.2.2 Laboratory Assessments

Blood samples for hematology and biochemistry and urine samples for urinalysis will be collected as indicated in the Schedule of Assessments [Table 1]. All clinical laboratory assessments will be performed at a central laboratory except for urinalysis dipsticks which will be conducted locally to support study eligibility or AEs. A urine pregnancy test in female subjects of childbearing potential will be performed at all on-site visits. A topical anesthetic cream or plaster must be offered at the point of venipuncture to minimize distress of the subject. For sampling the arm opposite to the arm used for blood pressure measurements should be used (i.e., preferably the left arm). Blood sampling should occur after vital signs and ECG measurements.

Sample collection, handling and storage will be described in a laboratory manual. All clinical laboratory test results, including ULNs used in exclusion and discontinuation criteria, will be compared to age appropriate norms.


ponsor: APGD ISN/Protocol: 178-CL-204

Scheduled blood sampling will only be performed at screening (visit 1), week 4 (visit 5) and EoT (visit 7) to keep the burden to subjects at a minimum. Additional hematology, biochemistry and urinalysis (urinalysis dipstick) tests will be performed at visit 3/week 0 (baseline) and visit 8/week 14 (EoS) only if an AE related to hematology, biochemistry or urinalysis parameters occurred since the previous visit or at the discretion of the investigator. If any of the clinical laboratory tests results are outside the normal range at any scheduled time point during the study, the investigator may decide to repeat the test(s) on new samples. The clinical relevance of the abnormal results will be documented. Clinically relevant changes will be recorded as AEs (see [Section 7.3 Adverse Events and Other Safety Aspects]).

Refer to the Alternate Schedule of Assessments [Table 12] for acceptable alternate methods to assess safety and efficacy parameters in the event the study is interrupted due to a crisis (e.g., natural disaster, pandemic).

### 7.2.3 Vital Signs and Electrocardiograms

### 7.2.3.1 Clinic-measurement of Vital Signs and Electrocardiograms

Blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]), pulse, and routine 12-lead ECG measurements will be taken as indicated in the Schedule of Assessments [Table 1].

The preferred method of measurement is via the auscultatory technique. If this method is not available at the study site, measurements will be per standard clinic practices. Single measurements of blood pressure, pulse, body temperature and ECGs will be measured in the sitting position (when possible, otherwise supine, but always in the same position). Subject should have been calm and without distress for at least 5 minutes. Preferably, the right arm should be used to measure vital signs. Body temperature will be measured with an ear thermometer as per standard of care. Clinic measurements will be used to assess eligibility.

For ECGs, dates and times may be generated by the machine's internal clock and are considered source data. The results are to be interpreted by qualified personnel in real time for the management of the subjects' clinical condition. The principal investigator/designee will initial and date and provide his/her clinical interpretation on each report. Any abnormalities must be evaluated in clinical context (based on subject's medical history and concomitant medication) and the investigator should determine if it is clinically significant. The results (normal, abnormal not clinically significant, abnormal clinically significant) are to be recorded in the eCRFs.

The original print-out and an electronic copy of all scheduled and unscheduled ECG tracings should be maintained on site as source data.

Clinic measurements will be used to assess eligibility. Clinically relevant adverse changes in vital signs and ECGs will be recorded as an AE (see [Appendix 12.4.1 Definition of Adverse Events]).


ISN/Protocol: 178-CL-204

### 7.2.3.2 Self-measurement of Vital Signs

Self-blood pressure monitoring (SBPM; SBP and DBP) will be measured as indicated in the Schedule of Assessments [Table 1] and whenever deemed necessary by the investigator.

SBPM will be measured once in the morning and evening during the 2-day weekend bladder e-diary collection period. Measurements will be taken in the sitting position (when possible, otherwise supine, but always in the same position). Preferably, the right arm should be used. Subject should have been calm and without distress for at least 5 minutes. Morning measurement should be taken before IP intake and evening measurement should be taken prior to bedtime.

Devices for measuring blood pressure will be provided to subjects for home measurements. Detailed on-site training to use the SBPM device and a booklet with operating instructions in local language will be provided to the subject and the subject's parent(s)/legal guardian(s). Results will be directly entered by the subject or subject's parent(s)/legal guardian(s) in the e-diary (see [Section 10.1 Data Collection]).

#### 7.2.4 **Physical Examination**

Physical examination will be performed as indicated in the Schedule of Assessments [Table 1] and whenever there is a medical indication.

The physical examination will be performed as described in the study site's SOPs for physical examination. In this study, the physical examination will be done to evaluate general physical condition and encompasses standard, full physical examinations to assess general appearance, skin, eyes, ears, nose, throat, neck, cardiovascular, chest and lungs, abdomen, musculoskeletal, neurologic status, mental status and lymphatic systems.

New or worsening clinically significant physical examination findings after signing of ICF will be recorded as AEs if they meet the criteria in [Section 7.3 Adverse Events and Other Safety Aspects].

#### 7.2.5 Post Void Residual Volume Assessments

PVR volume will be assessed by ultrasonography at visit 3/week 0 (baseline), visit 5/week 4, visit 7/week 12 (EoT) and visit 8/week 14 (EoS). For each subject, the same method should be used throughout the study. The bladder should only be emptied when it was initially filled with preferably > 50% of the bladder capacity for age. Every attempt should be made to measure PVR volume within a minute of voiding. A PVR volume of  $\leq 20$  mL is sufficient and the assessment does not have to be repeated. If the PVR volume is > 20 mL, the PVR volume assessment should be repeated (filled with preferably > 50% of the bladder capacity for age). If the subject is unable to complete a second measurement, it is up to the investigator to judge whether it can be skipped (and write the reason in the CRF). At visit 3/week 0 (baseline), the lowest PVR volume result measured should be used to evaluate the exclusion criterion. In case the lowest PVR volume measured is > 20 mL at visit 3/week 0 (baseline), the subject should be excluded from the study.


### 7.2.6 Acceptability and Palatability Questionnaire

The acceptability and palatability questionnaire will be completed as indicated in the Schedule of Assessments [Table 1]. For each IP formulation, a separate questionnaire is available [Appendix 12.8 Acceptability and Palatability Questionnaire for Tablets and Appendix 12.9 Acceptability and Palatability Questionnaire for Oral Suspension].

ISN/Protocol: 178-CL-204

### 7.2.7 Order of Assessments

The following order should be followed when more than 1 assessment is required at a time point with blood sampling for pharmacokinetics/metabolic profiling being collected nearest to the scheduled time point:

- 1. ECG
- 2. Vital signs
- 3. Blood collection

# 7.3 Adverse Events and Other Safety Aspects

The definitions of an AE or SAE can be found in [Appendix 12.4 Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up or Reporting].

The investigator and medically qualified designee(s) are responsible for detecting, documenting and recording events that meet the definition of an AE or SAE.

# 7.3.1 Time Period for Collecting Adverse Event and Serious Adverse Event Information

In order to identify any events that may be associated with study procedures and could lead to a change in the conduct of the study, Astellas collects AEs even if the subject has not received IP. AE collection begins after the signing of the ICF/assent and will be collected until 30 days after the final IP administration or when the subject is determined to be a screen failure.

### 7.3.2 Method of Detecting Adverse Events and Serious Adverse Events

The methods of recording, evaluating and assessing seriousness, causality and severity of AEs and SAEs are described in [Appendix 12.4 Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up or Reporting]. Care will be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and nonleading verbal questioning of the subject is the preferred method to inquire about AE occurrences.

An AE with a change in severity is recorded as a new AE.

### 7.3.3 Follow-up of Adverse Events

All AEs occurring during or after the subject has discontinued the study are to be followed up until resolved or judged to be no longer clinically significant, or until they become chronic to the extent that they can be fully characterized by the investigator.

If after the protocol-defined AE collection period (see [Section 7.3.1 Time Period for Collecting Adverse Event and Serious Adverse Event Information]), an AE progresses to an

11 Feb 2021 Astellas 


SAE, or the investigator learns of any (S)AE (serious adverse event or adverse event) including death, where he/she considers there is reasonable possibility it is related to the IP or study participation, the investigator must promptly notify the sponsor.

ISN/Protocol: 178-CL-204

### 7.3.4 Reporting of Serious Adverse Events

Prompt notification by the investigator to the sponsor of an SAE is essential, so that legal obligations and ethical responsibilities towards the safety of subjects and the safety of a study intervention under clinical investigation are met.

In the case of an SAE, the investigator must contact the sponsor by fax or email immediately (within 24 hours of awareness).

Procedures for reporting SAEs to the sponsor are described in [Appendix 12.4.5 Reporting Procedures for Serious Adverse Events].

# 7.3.5 Disease-related Events and/or Disease-related Outcomes Not Qualifying as Adverse Events or Serious Adverse Events

Under this protocol, the following event(s) will not be considered as an SAE:

- Disease progression: events including defined study endpoints that are clearly consistent with the expected pattern of progression of the underlying disease are not to be recorded as AEs. These data will be captured as efficacy assessment data as outlined in [Section 7.1 Efficacy Assessments]. If there is any uncertainty as to whether an event is due to anticipated disease progression and/or if there is evidence suggesting a causal relationship between the IP and the event, it should be reported as an SAE. All deaths up to 30 days after the final IP administration must be reported as an SAE, even if attributed to disease progression.
- Preplanned and elective hospital/clinical procedures/interventions or procedures for diagnostic, therapeutic, or surgical procedures for a pre-existing condition that did not worsen during the course of the study. These procedures are collected per the electronic data source's completion guidelines.

### 7.3.6 Adverse Events of Special Interest

Adverse Events of Special Interest include:

- Increased blood pressure
- Cardiac electrophysiology (including QTc prolongation) and cardiac arrhythmia (including increased heart rate, tachycardia, atrial fibrillation and palpitations)
- Hypersensitivity reactions
- Urinary retention
- Hepatotoxicity
- Seizure/syncope

AEs (serious or nonserious) of special interest are to be collected via the SAE worksheet and reported within 24 hours as described in [Appendix 12.4.5 Reporting Procedures for Serious Adverse Events].


ponsor: APGD ISN/Protocol: 178-CL-204

### 7.3.7 Special Situations

Certain special situations observed in association with the IP, such as incorrect administration (e.g., wrong dose of IP or background therapy) are collected in the electronic data source, as protocol deviation per [Section 10.3 Major Protocol Deviations] or may require special reporting, as described below. These special situations are not considered AEs, but do require to be communicated to Astellas as per the timelines defined below.

If a special situation is associated with, or results in, an AE, the AE is to be assessed separately from the special situation and captured as an AE in the electronic data source. If the AE meets the definition of an SAE, the SAE is to be reported as described in [Appendix 12.4.5 Reporting Procedures for Serious Adverse Events] and the details of the associated special situation are to be included in the clinical description on the SAE worksheet.

The special situations are:

- Pregnancy
- Medication error/overdose
- Misuse/abuse
- Occupational exposure
- Suspected drug-drug interaction

Instructions and procedures for reporting special situations are provided in [Appendix 12.4.6 Reporting Procedures for Special Situations].

### 7.3.8 Supply of New Information Affecting the Conduct of the Study

When new information becomes available that is necessary for conducting the study properly, the sponsor will inform all investigators involved in the study as well as the appropriate regulatory authorities. Investigators should inform the IRB/IEC of such information when needed.

The investigator will also inform the subjects, who will be required to sign an updated ICF/assent in order to continue in the study.

### 7.3.9 Urgent Safety Measures

An urgent safety measure (USM) is an intervention that is not defined by the protocol and can be put in place with immediate effect without needing to gain prior approval by the sponsor, relevant competent authorities and IRB/IEC, where applicable, in order to protect subjects from any immediate hazard to their health and/or safety. Either the investigator or the sponsor can initiate a USM. The cause of a USM can be safety-, product- or procedure-related.

### 7.3.10 Reporting Urgent Safety Measures

In the event of a potential USM, the investigator must contact the study physician (within 24 hours of awareness). Full details of the potential USM are to be recorded in the subject's


medical records. The sponsor may request additional information related to the event to support their evaluation.

ISN/Protocol: 178-CL-204

If the event is confirmed to be a USM, the sponsor will take appropriate action to ensure the safety and welfare of the subjects. These actions may include but are not limited to a change in study procedures or study treatment, halting further enrollment in the study, or stopping the study in its entirety. The sponsor or sponsor's designee will notify the relevant competent authorities and concerned ethics committee within the timelines required per current local regulations, and will inform the investigators, as required. When required, investigators must notify their IRB/IEC within timelines set by regional regulations.

### 7.4 Pharmacokinetics

Blood samples for the analysis of mirabegron in plasma will be collected as indicated in the Schedule of Assessments [Table 1] for the evaluation of pharmacokinetics.

The actual date and time of each blood sample collection will be documented. Sample collection, handling and storage will be described in the laboratory manual. Bioanalysis of mirabegron will be performed using a validated method.

A topical anesthetic cream or plaster must be offered at the point of venipuncture to minimize distress of the subject. For sampling the arm opposite to the arm used for blood pressure measurements should be used (i.e., preferably the left arm). Blood sampling should occur after vital signs and ECG measurements.

The pharmacokinetic parameters that will be calculated as part of the secondary pharmacokinetic endpoint are steady-state C<sub>max</sub>, AUC<sub>tau</sub>, C<sub>trough</sub>, T<sub>max</sub>, CL/F and V<sub>z</sub>/F. Additional parameters may be calculated based on the population pharmacokinetic model used.

# 7.5 Pharmacodynamics | Immunogenicity

Not applicable.

### 7.6 Electronic Clinical Outcome Assessment

For this study, it has been decided that there are justifiable scientific reasons (i.e., recall bias) to limit subject reported changes to changes reported by the subject to the site within 1 business day of its entry, as changes outside of this window could potentially impact the data integrity of the study. The data that will be under this rule are all subject/guardian/parent-entered primary and secondary endpoints data. However, the site/investigator can remove/inactivate any data that they determine to be in error at any time with source documentation to support the change including subject confirmation. Data will never be deleted from the electronic database by the electronic clinical outcome assessment (eCOA) service provider, but will be removed logically as per investigator's request and approval. All data changes are audit trailed showing the original entries alongside all changes including who requested the change, why it was requested, who made the change and when it was


made. Audit trails are reviewed by the sponsor/clinical research organization (CRO) to ensure adherence to the protocol and appropriate source exists at site to substantiate the change.

ISN/Protocol: 178-CL-204

Subject bladder diaries, questionnaires and other data will be completed by the subject or the subject's parent(s)/legal guardian(s)/caregiver(s) on an electronic device (e-diary). The information on the electronic device will be automatically uploaded to a central website. The investigator or site designee should review the diaries and questionnaire data on the website to ensure completion and protocol compliance before each planned visit of the subject (on site visit or TC) and discuss the results or retrain the subject and/or subject's parent(s)/legal guardian(s)/caregiver(s), if applicable. In case clinically relevant adverse changes are noticed during review of the e-diary, these will be recorded as an AE [Appendix 12.4.1 Definition of Adverse Events].

The bladder e-diary, questionnaire results and other data collected in the e-diary will be transferred electronically to the sponsor or designee at predefined intervals during the study. The vendor will provide the sponsor or designee with a complete and clean copy of the study data. The ownership of this data is with the investigator and subsequently any changes requested to these subject-reported or nonsubject reported data will be made using the vendor's established process (e.g., a data clarification form to the vendor). The requested change must be supported by documented evidence at study site.

For this study the following information will be collected and entered by the subject or subject's parent(s)/legal guardian(s) in the e-diary (see [Sections 7.2.6 Acceptability and Palatability Questionnaire and 7.2.3.2 Self-measurement of Vital Signs] for detailed information per visit):

- Bladder e-diary:
  - Each day on weekend prior to week -2: volume measurements
  - Each day for 7 days before visit 3/week 0: micturition frequency
  - Each day for 7 days before visit 3/week 0: incontinence episodes
  - On the 2-day weekend period: volume measurements
- SBPM (blood pressure and pulse):
  - Each day of the 2-day weekend period: twice per day
  - On 2 consecutive weekend days at around 1 and 2 weeks after start of dosing with PED25 (day 1) and after up-titration to PED50, if not already covered by the scheduled SBPM
- Acceptability and Palatability Questionnaire:
  - On 1 weekend day preceding visit 7/week 12 (EoT)

The investigator must guide the subject and subject's parent(s)/legal guardian(s) to ensure that on the evening before and during the 2-day weekend period collection of volume, the subject's fluid intake should be regulated (as per investigator guidance) to an appropriate level considering, e.g., age, sex and subject's condition into account. The intake must remain as consistent as possible on these volume collecting days throughout the entire study.


### 7.7 Other Assessments

Acceptability and palatability questionnaire will be completed on 1 weekend day preceding Visit 7/Week 12 (EoT). For each formulation a separate questionnaire is available, please see Appendices 12.8 Acceptability and Palatability Questionnaire for Tablets and 12.9 Acceptability and Palatability Questionnaire for Oral Suspension.

ISN/Protocol: 178-CL-204

Questionnaires are to be completed by the subject or the subject's parent(s)/caregiver(s) in the local language and provided via the e-diary. Results will be directly entered in the e-diary by the subject or subject's parent(s)/caregiver(s).

### 7.8 Total Amount of Blood

The total amount of blood for each subject will vary depending on the course of their disease, duration on treatment and central laboratory requirements. At any time during the study, if any laboratory abnormalities are found for a subject, additional blood may be drawn for safety monitoring.

The maximum blood volume to be collected within 24 hours is approximately 9.5 mL per subject on pharmacokinetic sampling days at visit 5/week 4 and visit 7/week 12 (EoT).

The total blood volume to be collected will be as follows

Table 8 Total Blood Volume per Subject over the Entire Study Period

| Sample Type | Number of Samples | Sample Volume (mL) | Total Volume (mL) |
|---|---|---|---|
| Pharmacokinetics | 2 | 5.0 | 10.0 |
| Clinical Laboratory Tests†<br>Biochemistry/hematology | 3 | 4.5‡ | 13.5 |
| Total | 23.5 | | |

<sup>†</sup> Additional hematology and biochemistry tests of approximately 4.5 mL total will be performed at visit 3/week 0 (baseline) and visit 8/week 14 (EoS) only if an adverse event related to hematology or biochemistry parameters occurred since the previous visit or at the discretion of the investigator. The total amount of blood drawn from subjects who require additional hematology and biochemistry tests due to AEs could be up to 32.5 mL.

### 8 DISCONTINUATION

# 8.1 Discontinuation of Individual Subject(s) From Study Treatment(s)

A discontinuation from treatment is defined as a subject who is randomized and for whom study treatment is permanently discontinued for any reason.

The subject is free to withdraw from the study treatment and/or study for any reason and at any time without giving reason for doing so and without penalty or prejudice. The investigator is also free to discontinue the participant from study treatment or to terminate a subject's involvement in the study at any time if the subject's clinical condition warrants it.

The reason for discontinuation from study treatment must be documented in the subject's medical records.

<sup>‡</sup> Volume does not take any unscheduled visits or repeat tests into account (e.g., follow up of adverse events).

Sponsor: APGD ISN/Protocol: 178-CL-204

A subject must discontinue study treatment for any of the following reasons:

- Subject requests to stop treatment.
- Any clinical AEs, laboratory abnormality or intercurrent illness, in the opinion of the investigator, indicates continued treatment is not in the best interest of the subject.
- If signs or symptoms of hypersensitivity to mirabegron are observed (e.g., anaphylactic reaction, erythema multiforme or exfoliative dermatitis).
- ALT or AST  $> 8 \times ULN$ .
- ALT or AST  $> 5 \times ULN$  for more than 2 weeks.
- ALT or AST >  $3 \times \text{ULN}$  and TBL >  $2 \times \text{ULN}$  or international normalized ratio (INR) > 1.5 (if INR testing is applicable/evaluated).
- ALT or AST  $> 3 \times$  ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash and/or eosinophilia (> 5%).
- Female subject becomes pregnant.
- Prolongation of QT > QTcF > 440 msec and/or QT interval prolongation > 30 msec versus baseline.
- Subject with (systolic blood pressure ≥ 160 mm Hg or diastolic blood pressure ≥ 100 mmHg.

If a subject discontinues treatment prematurely, the subject will be encouraged to complete all scheduled visits to record all available information.

## 8.2 Discontinuation of Individual Subject(s) From Study

All subjects who discontinue study treatment will remain in the study and must continue to be followed for protocol-specific follow-up procedures as outlined in the Schedule of Assessments [Table 1]. The subject will also be encouraged to attend all planned visits until the planned End of Study visit to provide data even if not on treatment anymore. The only exception to this is when the subject specifically withdraws consent/assent for any further contact with him/her or persons previously authorized by the subject to provide this information.

### 8.2.1 Lost to Follow-up

Every reasonable effort is to be made to contact any subject lost to follow-up during the course of the study to complete study-related assessments, record outstanding data and retrieve IP.

# 8.3 Discontinuation of the Study Site

If an investigator intends to discontinue participation in the study, the investigator must immediately inform the sponsor.

# 8.4 Discontinuation of the Study

The DSMB will review safety data periodically and provide a recommendation to the sponsor if the study should continue or be stopped due to safety concerns. The sponsor may terminate this study prematurely, either in its entirety or at any study site, for reasonable cause provided

Sponsor: APGD ISN/Protocol: 178-CL-204 EudraCT number 2016-001767-37


that written notice is submitted in advance of the intended termination. Advance notice is not required if the study is stopped due to safety concerns. If the sponsor terminates the study for safety reasons, the sponsor will immediately notify the investigator and subsequently provide written instructions for study termination. The study may also be stopped as a result of the outcome of the interim analysis [Section 9.10 Interim Analysis and Early Discontinuation of the Study].

### 9 STATISTICAL METHODOLOGY

A statistical analysis plan (SAP) will be written to provide details of the analysis, along with specifications for tables, listings and figures to be produced. The SAP will be finalized before database hardlock. Changes from the planned analyses planned in the final SAP that impact the statistical analyses will be justified in the clinical study report (CSR).

In general, all data will be summarized with descriptive statistics frequency and percentage for categorical data. Data will be summarized by age group, treatment group and visit unless otherwise stated.

# 9.1 Sample Size

Efficacy of mirabegron in children will be based on both primary and secondary endpoints. Given the clinical hurdle to demonstrate efficacy in a population challenging to recruit, an alpha-level of 10% would appear reasonable and justified. In a study with propiverine in children, Marschall-Kehrel (2009) showed a difference in mean number of micturition episodes/24 hours of 0.8 between propiverine and placebo, with a SD between 2.2 and 2.3. Assuming at least similar efficacy of mirabegron, with a treatment effect of 0.9 micturitions per day between mirabegron and placebo and a common SD of 2.3, a sample size of 82 evaluable subjects (children) per treatment group is assumed per treatment group would provide a power of 80%.

These assumptions, together with levels for Type-1 error and power were agreed upon with Pediatric Committee in the current Pediatric Investigation Plan.

Under the assumption that after randomization about 10% of the subjects will not be evaluable for the analysis of the primary endpoint (i.e., not fulfilling the criteria for inclusion in full analysis set [FAS]), at least 184 children (5 to < 12 years of age) must be randomized in order to have at least 164 evaluable children for the analysis of the primary efficacy endpoint.

For adolescents, no formal sample size will be calculated; at least 32 adolescents (12 to < 18 years of age) must be randomized, yielding at least 16 adolescents on mirabegron. Further assuming a 50% screen failure rate, approximately 368 children have to be enrolled to achieve 184 children (5 to < 12 years of age) randomized and approximately 64 adolescents will be enrolled to achieve at least 32 adolescents (12 to < 18 years of age) randomized (at least 92 children and 16 adolescents must be randomized to mirabegron).

Recruitment will continue until the minimum number to be randomized in both children and adolescents have been achieved.

11 Feb 2021 Astellas 

ISN/Protocol: 178-CL-204

#### 9.2 **Analysis Sets**

Detailed criteria for analysis sets will be laid out in classification specifications and the allocation of subjects to analysis sets will be determined prior to database hardlock.

#### 9.2.1 **Full Analysis Set**

The FAS will consist of all subjects who are randomized and receive at least 1 dose of IP and have at least 1 post baseline measurement for mean number of micturitions per 24 hours. The FAS will be analyzed by treatment arm as randomized (i.e., treatment arm based on randomization assignment). This will be the primary analysis set for efficacy analyses. Selected demographic and baseline characteristics will also be summarized for the FAS.

#### 9.2.2 Per Protocol Set

The per protocol set (PPS) will consist of all subjects who are randomized and receive at least 1 dose of IP and have at least 1 post baseline measurement for mean number of micturitions per 24 hours, and who do not meet criteria for PPS exclusion. These criteria are to capture relevant nonadherence to the protocol and will be defined in the SAP. Further criteria may be defined in the SAP. The PPS will be a secondary analysis set for efficacy analyses.

Selected demographic and baseline characteristics may also be summarized for the PPS.

#### 9.2.3 Safety Analysis Set

The safety analysis set (SAF) will consist of all subjects who took at least 1 dose of IP. The safety set will be analyzed by treatment arm as treated (i.e., based on the treatment the subject actually received rather than the treatment to which the subject was randomized). The SAF will be used for all summaries of demographic and baseline characteristics and all safety- and tolerability-related variables.

#### 9.2.4 **Pharmacokinetics Analysis Set**

The pharmacokinetics analysis set (PKAS) will consist of all subjects who took at least 1 dose of IP for whom sufficient plasma concentration data are available to facilitate derivation of at least 1 pharmacokinetic parameter and for whom the time of dosing on the day before sampling. Additional subjects may be excluded from the PKAS at the discretion of the pharmacokineticist. Any formal definitions for exclusion of subjects or time points from the PKAS will be documented in the classification specifications and be determined at the classification meeting.

#### 9.2.5 Pharmacodynamic Analysis Set

Not applicable.

#### 9.3 **Demographics and Baseline Characteristics**

The summaries to be provided for demographics and baseline characteristics will be described here.

#### ISN/Protocol: 178-CL-204

### 9.3.1 Demographics

The demographic summary will include age, sex, race, ethnicity, body weight, height, body mass index (BMI) (at screening) and EBC. Baseline characteristics will include, among others, medical history, OAB diagnosis and history. Selected demographic and baseline characteristics will be summarized at least for the SAF and FAS.

Demographic data will be listed.

### 9.3.2 Subject Disposition

The number and percentage of subjects who completed and discontinued treatment and reasons for treatment discontinuation will be presented for all randomized subjects and for subjects in the SAF by age group, treatment group and overall. Similar tables for screening disposition, investigational period disposition and follow-up disposition will also be presented for all enrolled subjects by age group and overall. All disposition details and dates of first and last evaluations for each subject will be listed.

# 9.3.3 Previous and Concomitant Treatment (Medication and Nonmedication Therapy)

Previous and concomitant medications will be coded with WHO-Drug Dictionary (WHO-DD), and will be summarized by therapeutic subgroup (Anatomical Therapeutic Chemical [ATC] Classification System 2<sup>nd</sup> level), chemical subgroup (ATC 4<sup>th</sup> level) and preferred WHO name for the SAF. Subjects taking the same medication multiple times will be counted once per ATC level. A medication which can be classified into several chemical and/or therapeutic subgroups will be presented in all chemical and therapeutic subgroups.

A listing of previous and concomitant medications with ATC codes by WHO preferred name will be provided for all screened subjects.

### 9.3.4 Medical History

Medical history will be coded in MedDRA and will be summarized by SOC and preferred term (PT) for the SAF. Subjects will only be counted once per MedDRA level.

Medical history for each subject will be listed.

### 9.3.5 Investigational Product Exposure

Descriptive statistics for cumulative amount of the IP the subject was exposed to and average daily dose.

Duration of exposure will be summarized in the following by descriptive statistics.

Exposure time will be categorized according to the following categories for the treatment period:

- < 14 days
- At least 14 days, < 28 days
- At least 28 days, < 56 days
- At least 56 days

11 Feb 2021 Astellas 


### Unknown

All IP exposure data will be listed.

## 9.4 Analysis of Efficacy

Efficacy analysis will be conducted on the FAS and PPS, and interpretation of results from statistical tests in children (5 to < 12 years of age) will be based on the FAS. The PPS will be used to assess the robustness of the results from the statistical tests based on the FAS. Efficacy analysis in adolescents will only be exploratory.

ISN/Protocol: 178-CL-204

### 9.4.1 Analysis of Primary Endpoint

### 9.4.1.1 Primary Analysis

The primary estimator for the primary estimand as defined in [Section 3.1 Estimand] will be calculated according to the evaluation of the primary efficacy endpoint. The primary efficacy endpoint change from baseline to week 12/EoT in mean micturitions per 24 hours (in children [5 to < 12 years of age]), will be analyzed using an analysis of covariance (ANCOVA). The ANCOVA model will include treatment group, sex and geographical region as fixed effects and the mean number of micturitions per 24 hours at baseline as covariate. This analysis will be performed and once with imputation of missing week 12 data using the last observation carried forward (LOCF) method.

The hypothesis for comparisons is given as follows:

H0: The adjusted mean change from baseline at week 12 in mean number of micturitions per 24 hours for mirabegron and placebo are the same.

H1: The adjusted mean change from baseline at week 12 in mean number of micturitions per 24 hours for mirabegron and placebo are not the same.

Statistical testing will be done at a 2-sided 0.1 significance level. A 90% CI for the treatment difference (mirabegron – placebo) will be provided. The primary analysis will use the FAS. The plausibility of the underlying assumption of missing at random for the primary estimator will be evaluated, and; therefore, the estimation of the treatment effect. Sensitivity analyses under alternative assumptions for missing data mechanisms such as missing not at random to show robustness of the estimates will be further specified in the SAP.

### 9.4.1.2 Secondary Analysis

The same analysis of the primary endpoint as described in [Section 9.4.1.1 Primary Analysis] will be conducted using the PPS, and without imputation using FAS.

The change from visit 3/week 0 (baseline) to visit 7/week 12 (EoT) in mean number of micturitions per 24 hours in children (5 to < 12 years of age) will be analyzed. The primary analysis for the primary endpoint will be using a repeated measures ANCOVA model with treatment group, visits (week 4, 8 and 12), sex, geographical region and the interaction between treatment group and visit as fixed effects and mean number of micturitions per 24 hours at baseline as covariate. Mirabegron will be compared to placebo using a linear

Sponsor: APGD ISN/Protocol: 178-CL-204

contrast within the repeated measures ANCOVA model, with 2-sided significance level of alpha = 0.1 and 90% CI. This analysis will be conducted using the FAS.

In addition to the parametric ANCOVA, a nonparametric ANCOVA will also be performed: (stratified) rank ANCOVA. This analysis will be conducted using the FAS.

### 9.4.1.3 Subgroup Analysis

For the primary efficacy endpoint, descriptive statistics (n, mean, 95% confidence interval around the mean, SD, minimum, median, maximum) will be calculated for mean change from baseline at each visit by sex, race, ethnicity, geographical region, formulation (tablets vs. oral suspension), prior OAB treatment and symptomatic UTI.

### 9.4.2 Analysis of Secondary Endpoints

The same analysis (ANCOVA) as for the primary endpoint will be applied to change from baseline at the end of the 12-week treatment period in children (5 to  $\leq$  12 years of age) for:

- Mean volume voided per 24 hours
- Maximum volume voided
- Mean number of daytime incontinence episodes per 24 hours
- Mean number of nighttime incontinence episodes per 24 hours
- Mean number of daytime micturitions per 24 hours

Change from baseline in the number of dry (incontinence free) days per 7 days at the end of the 12-week treatment period will be analyzed with a negative binomial regression model including treatment group, sex, geographical region as factors and the log baseline rate of number of dry days (e.g., the log of the number of dry days divided by number of diary days at baseline) as covariate.

### 9.4.3 Analysis of Exploratory Endpoints

All efficacy endpoints for adolescents will be analyzed descriptively.

Data of the following explorative endpoints will be summarized, separately, for pediatric subjects:

- Percentage of subjects with a reduction in daytime incontinence episodes (< 50% reduction [nonresponder], 50% [partial responder] and 100% [responder])
- Improvement from baseline in worst incontinence grading
- Change from baseline at the end of the 12-week treatment period adjusted for fluid intake:
  - Mean number of micturitions per 24 hours
- Change from baseline at the end of the 12-week treatment period (adolescents only):
  - Mean number of micturitions per 24 hours
  - Mean number of daytime micturitions per 24 hours
  - Mean volume voided per 24 hours
  - Mean number of incontinence episodes per 24 hours


• Number of dry (incontinence-free) days per 7 days at the end of the 12-week treatment period (adolescents only)

ISN/Protocol: 178-CL-204

Mean number of daytime grade 3 or 4 (Patient Perception of Intensity of Urgency Scale [PPIUS]) urgency episodes per 24 hours (adolescents only) will be summarized.

Correlations between the primary endpoint and mean volume voided, as well as incontinence episodes, will be explored.

Scatter plots will be presented to access the correlation between the primary end point, and mean volume voided and number of incontinence episodes at week 12.

## 9.5 Analysis of Safety

Safety analysis will be conducted on the SAF and conducted separately for children, adolescents and overall. Safety endpoints will be summarized using descriptive statistics.

#### 9.5.1 Adverse Events

AEs will be coded using MedDRA. A TEAE is defined as an AE observed after starting administration of the IP and 30 days after the final administration of IP. An IP-related TEAE is defined as any TEAE with a causal relationship assessed as "yes" by the investigator.

The number and percentage of TEAEs, drug-related TEAEs, serious TEAEs, drug-related serious TEAEs, TEAEs leading to leading to withdrawal of treatment and drug-related TEAEs leading to leading to withdrawal of treatment will be summarized by SOC, preferred term, age group and treatment group. The number and percentage of TEAEs by severity will also be summarized. The worst severity will be summarized if the same AE is recorded more than once for a subject.

AE data will be listed.

### 9.5.2 Laboratory Assessments

For quantitative clinical laboratory measurements (hematology, biochemistry and urinalysis), descriptive statistics will be used to summarize results and change from baseline by treatment group and within treatment group and across age group.

Shifts relative to normal ranges from baseline to each visit during the treatment period in clinical laboratory tests will be tabulated.

Laboratory data will be listed.

The laboratory parameters that will be assessed during the conduct of the study are listed in [Appendix 12.7 Laboratory Assessments].

In cases where laboratory evaluations are conducted locally, the values obtained will be adjusted to values obtained by the central laboratory. Details will be described in the SAP.

### 9.5.3 Vital Signs

Descriptive statistics will be used to summarize vital sign results and changes from baseline by treatment group and within treatment group and across age group. For clinic


ISN/Protocol: 178-CL-204

measurements Z-scores and percentiles for SBP and DBP will be calculated and summarized based on a comparison with age and height norms supplied by the Center for Disease Control and Prevention. Details to calculate Z-scores and percentiles will be provided in the SAP.

Z-scores and percentiles for pulse rate will be calculated and summarized based on a comparison with age norms based on Fleming [Fleming et al, 2011]. Details to calculate Z-scores and percentiles will be provided in the SAP.

Vital signs data will be listed.

#### 9.5.4 **Physical Examination**

Abnormal findings/conditions identified during the physical examinations will be listed as part of the medical history for the screening visit, or as AEs at later visits.

#### 9.5.5 Electrocardiogram

The routine 12-lead ECG results will be summarized separately for children (5 to < 12 years of age) and adolescents (12 to < 18 years of age) by treatment group and visit. ECGs will be recorded prior to blood draw.

#### 9.5.6 Post Void Residual Volume

The PVR volume data and change from baseline data will be summarized by treatment group and within treatment group and across age.

#### 9.5.7 **Acceptability and Palatability Questionnaire**

Results from the acceptability and palatability questionnaire for tablets [Appendix 12.8 Acceptability and Palatability Questionnaire for Tablets] and for oral suspension [Appendix 12.9 Acceptability and Palatability Questionnaire for Oral Suspension] will be summarized at week 12/EoT by age group and treatment group.

#### 9.6 **Analysis of Pharmacokinetics**

Pharmacokinetic analysis will be conducted on the PKAS and conducted separately for children, adolescents and overall. Descriptive statistics (n, mean, SD, minimum, median, maximum, coefficient of variation (CV), geometric mean and geometric CV) will be used to summarize plasma concentrations of mirabegron by visit and time point. Further details will be specified in the SAP.

#### 9.6.1 **Estimation of Pharmacokinetic Parameters**

The plasma concentrations will be analyzed with nonlinear mixed effects modeling (population pharmacokinetics) using Non-Linear Mixed Effects Modeling (NONMEM) software (version 7.3 or higher, ICON Development Solutions, Ellicott City, MD, US) to estimate the pharmacokinetic parameters. Results will be reported separately.

#### 9.7 **Analysis of Pharmacodynamics | Immunogenicity**

Not applicable.

ISN/Protocol: 178-CL-204

## 9.8 Other Analyses

Not applicable.

# 9.9 Major Protocol Deviations

Major protocol deviations as defined in [Section 10.3 Major Protocol Deviations] will be summarized for all randomized subjects by study site, treatment group and overall separately for children (5 to < 12 years of age) and adolescents (12 to < 18 years of age).

Major protocol deviation data will be listed by study site and subject.

The major protocol deviation criteria will be uniquely identified in the summary table and listing.

# 9.10 Interim Analysis (and Early Discontinuation of the Study)

A blinded interim analysis will be performed after 50% of children planned to be randomized have had their week 12/EoT assessment. The interim analysis will determine if the chance of a positive study with respect to the primary endpoint at the EoS is high enough to justify continuation of the study; otherwise, the study will be stopped for futility.

Given the data at the interim analysis, the independent data analysis center (IDAC) will calculate the predictive probability of a positive study. A positive study is defined as the final 1-sided p-value  $\leq 0.05$  when comparing Mirabegron vs. placebo in the primary efficacy analysis (in children [5 to  $\leq$  12 years of age]). If the predictive probability is  $\leq$  5% at this interim evaluation, the study will be recommended to stop for futility. Otherwise, the study will continue.

Detailed information on the decision rule of futility and simulations illustrating the operating characteristics of futility criterion will be presented in the SAP.

### 9.11 Additional Conventions

Missing data for efficacy endpoints will be imputed as EoT values, details will be described in the SAP. Handling of incomplete dates will also be described in the SAP.

Geographical regions that do not enroll sufficient subjects to allow estimation of the geographical effect will be pooled for analyses by geographical region. The pooling decisions will be made and documented prior to study hardlock.

### 10 OPERATIONAL CONSIDERATIONS

### 10.1 Data Collection

The investigator or site designee will enter data collected using an electronic data capture system. In the interest of collecting data in the most efficient manner, the investigator or designee should record data (including clinical laboratory values, if applicable) in the electronic case report form within 5 days after the subject's visit.


The monitor should verify the data in the electronic case report forms with the source and confirm that there are no inconsistencies among them.

ISN/Protocol: 178-CL-204

Clinical laboratory tests are performed at central laboratory. Central laboratory data will be transferred electronically to the sponsor or designee at predefined intervals during the study. The central laboratory will provide the sponsor or designee with a complete and clean copy of the data

Subject bladder e-diaries and questionnaires as described in [Section 7.6 Electronic Clinical Outcome Assessment] will be completed by the subject on an electronic device and the collected electronic data source will be hosted at the vendor.

The investigator or designee will review the diaries and questionnaire data throughout the study to ensure completion and protocol compliance.

## **10.2** Demographics and Baseline Characteristics

### 10.2.1 Demographics

Demographics and baseline characteristics will be collected as indicated in the Schedule of Assessments [Table 1]. This will include age, sex, race, ethnicity, body weight and height.

### 10.2.2 Medical History

A complete medical history will be collected as indicated in the Schedule of Assessments [Table 1].

### 10.2.3 Diagnosis of the Target Disease, Severity and Duration of Disease

A detailed OAB history for each subject will be collected at visit 1/screening. This history includes the underlying condition, comorbidities associated with OAB and treatment history for OAB.

# **10.3** Major Protocol Deviations

A protocol deviation is generally an unplanned excursion from the protocol that is not implemented or intended as a systematic change. All deviations from the protocol are to be recorded. A protocol waiver is a documented prospective approval of a request from an investigator to deviate from the protocol. Protocol waivers are strictly prohibited.

The investigator is responsible for ensuring the study is conducted in accordance with the procedures and evaluations described in this protocol and must protect the rights, safety and well-being of subjects. The investigator should not implement any deviation from, or changes of, the protocol, unless it is necessary to eliminate an immediate hazard to subjects.

A major protocol deviation is 1 that may potentially impact the completeness, accuracy or reliability of data contributing to the primary endpoint or affect the rights, safety or well-being of a subject. Major protocol deviations will have additional reporting requirements.

When a major deviation from the protocol is identified for an individual subject, the investigator or designee must ensure the sponsor is notified. The sponsor will follow up with


the investigator, as applicable, to assess the deviation and the possible impact to the safety and/or efficacy of the subject to determine subject continuation in the study.

ISN/Protocol: 178-CL-204

The major protocol deviation criteria that will be summarized at the EoS are as follows:

- PD1 Entered into the study even though the subject did not satisfy entry criteria
- PD2 Developed withdrawal criteria during the study and was not withdrawn
- PD3 Received wrong treatment or incorrect dose
- PD4 Received excluded concomitant treatment

The investigator will also assure that deviations meeting IRB/IEC and appropriate regulatory authorities' criteria are documented and communicated appropriately. All documentation and communications to the IRB/IEC and appropriate regulatory authorities will be provided to the sponsor and maintained within the Trial Master File.

### 10.4 Study Organization

### 10.4.1 Data and Safety Monitoring Board

A DSMB will be implemented to act in an advisory capacity to the sponsor to monitor participant safety and data quality.

Subject safety overviews will be prepared by the IDAC and will be reviewed on a regular basis by the DSMB, who will advise the sponsor on appropriate steps to protect study participants, which may include the early termination of the study.

A separate charter will describe the responsibilities, remit and timing of DSMB meetings.

### 10.4.2 Independent Data Analysis Center

An IDAC for this study will serve the 2 purposes: (1) to generate periodic safety overviews for the DSMB and (2) to calculate the futility analysis. The statistical member of the DSMB may also serve as the IDAC statistician, as described in the DSMB charter. A SAP describing the details of the periodic safety review of outputs will be developed with input from the DSMB members.

### **10.4.3** Other Study Organization

Not applicable.

## ponsor: APGD ISN/Protocol: 178-CL-204

### 11 REFERENCES

- Austin PF, Bauer SB, Bower W, Chase J, Franco I, Hoebeke P, et al. The standardization of terminology of lower urinary tract function in children and adolescents: update report from the Standardization Committee of the International Children's Continence Society. J. Urol. 2014;191:1863-5.
- BETANIS® (prescribing information). Northbrook, Illinois: Astellas Pharma US, Inc.; Jun 2012.
- BETMIGA® (prescribing information). Northbrook, Illinois: Astellas Pharma US, Inc.; Apr 2018.
- Derweesh IH, Wheeler MA, Weiss RM. Alterations in G-proteins and β-adrenergic responsive adenylyl cyclase in rat urinary bladder during aging. J Pharmacol Exp Therap. 2000;294:969-74.
- Drossman DA, Hasler WL. Rome IV functional gastrointestinal disorders: disorders of gut-brain interaction. Gastroenterology. 2016;150:1257-61. Available at: https://www.gastrojournal.org/article/S0016-5085(16)30048-8/fulltext. Accessed 21 Jun 2019.
- Fleming S, Thompson M, Stevens R, Heneghan C, Plüddemann A, Maconochie I, et al. Normal ranges of heart rate and respiratory rate in children from birth to 18 years of age: a systematic review of observational studies. Lancet. 2011;377:1011-18.
- Flynn JT, Kaelbar DC, Baker-Smith CM, Blowey D, Carroll AE, Daniels SR, et al. Clinical practice guideline for screening and management of high blood pressure in children and adolescents. Pediatrics. 2017;140(3):e20171904.
- Investigator's Brochure Mirabegron (YM178), Astellas.
- Marschall-Kehrel D, Feustel C, Persson de Geeter C, Stehr M, Radmayr C, Sillén U, et al. Treatment with propiverine in children suffering from nonneurogenic overactive bladder and urinary incontinence: results of a randomized placebo-controlled phase 3 clinical trial. Eur Urol. 2009;55:729-36.
- McDowell MA, Fryar CD, Ogden CL, Flegal KM. Anthropometric reference data for children and adults: United States, 2003–2006. Natl Health Stat Report. 2008;22(10):1-48.
- Momper JD, Mulugeta Y, Green DJ, Karesh A, Krudys KM, Sachs HC, et al. Adolescent Dosing and Labeling Since the Food and Drug Administration Amendments Act of 2007. JAMA Pediatr. 2013;167:926-932.
- MYRBETRIQ® (prescribing information). Northbrook, Illinois: Astellas Pharma US, Inc.; Jun 2012.
- Nevéus T, von Gontard A, Hoebeke P et al. The standardization of terminology of lower urinary tract function in children and adolescents: report from the standardisation committee of the international children's continence society. J Urol. 2006; 176; 314 324.
- Schwartz GJ, Muñoz A, Schneider MF, Mak RH, Kaskel F, Warady BA, et al. New Equations to Estimate GFR in Children with CKD. J Am Soc Nephrol. 2009;20:629-37.
- Temple R. Hy's law: predicting serious hepatotoxicity. Pharmacoepidemiol Drug Saf. 2006;15:241-3.


ISN/Protocol: 178-CL-204

#### 12 **APPENDICES**

#### 12.1 **Ethical, Regulatory and Study Oversight Considerations**

#### 12.1.1 **Ethical Conduct of the Study**

The study will be conducted in accordance with the protocol, ICH guidelines, applicable regulations and guidelines governing study conduct and the ethical principles that have their origin in the Declaration of Helsinki.

#### 12.1.2 Institutional Review Board/Independent Ethics Committee/Competent **Authorities**

GCP requires that the protocol, any protocol amendments, Investigator's Brochure, ICF/assent and all other forms of subject information related to the study (e.g., advertisements used to recruit subjects) and any other necessary documents be reviewed by an IRB/IEC. The IRB/IEC will review the ethical, scientific and medical appropriateness of the study before it is conducted. IRB/IEC approval of the protocol, ICF/assent and subject information and/or advertising, as relevant, will be obtained prior to initiation of any studyspecific procedures.

Any substantial amendments to the protocol will require competent authority and IRB/IEC approval before implementation, except for changes necessary to eliminate an immediate hazard to subjects.

The investigator will be responsible for the following:

- Providing written summaries of the status of the study to the IRB/IEC annually or more frequently in accordance with the requirements, policies and procedures established by the IRB/IEC
- Notifying the IRB/IEC of SAEs or other significant safety findings as required by IRB/IEC procedures
- Providing oversight of the conduct of the study at the study site and adherence to requirements of 21 CFR, ICH guidelines, the IRB/IEC, EU Regulation No. 536/2014 for studies (if applicable), and all other applicable local regulations

### Protocol Amendment and/or Revision

Any changes to the study that arise after approval of the protocol must be documented as protocol amendments: substantial amendments and/or nonsubstantial amendments. Depending on the nature of the amendment, either IRB/IEC or competent authority approval or notification may be required. The changes will become effective only after the approval of the sponsor, investigator, IRB/IEC and appropriate regulatory authorities.

Amendments to this protocol must be signed by the sponsor and investigator. Written verification of IRB/IEC approval will be obtained before any amendment is implemented. Modifications to the protocol that are administrative in nature do not require IRB/IEC approval, but will be submitted to the IRB/IEC for their information, if required by local regulations.

11 Feb 2021 Astellas  Sponsor: APGD EudraCT number 2016-001767-37 - CONFIDENTIAL -

Sponsor: APGD ISN/Protocol: 178-CL-204

If there are changes to the ICF/assent, written verification of IRB/IEC approval must be forwarded to the sponsor. An approved copy of the new ICF/assent must also be forwarded to the sponsor.

### 12.1.4 Financial Disclosure

Investigators and subinvestigator(s) will provide the sponsor with sufficient, accurate financial information as requested to allow the sponsor to submit complete and accurate financial certification or disclosure statements to the appropriate regulatory authorities. Investigators are responsible for providing information on financial interests during the course of the study and for 1 year after completion of the study.

### 12.1.5 Informed Consent/Assent of Subjects

### 12.1.5.1 Subject Information and Consent/Assent

For this pediatric study in subjects aged 5 to < 18 years of age, in addition to information sheets and consent forms/assent for subjects (according to applicable local regulations), parent/legal guardian information sheets and consent forms/assent will also be prepared.

The investigator or his/her representative will explain the nature of the study to the subject and his/her parent(s)/legal guardian(s) and answer all questions regarding this study. Prior to any study-related screening procedures being performed on the subject, the ICF/assent will be reviewed, signed and dated by the subject or his/her parent(s)/legal guardian(s), the person who administered the ICF/assent and any other signatories according to local requirements. A copy of the signed ICF/assent will be given to the subject and the original will be placed in the subject's medical record. An entry must also be made in the subject's dated source documents to confirm that the ICF/assent was signed prior to any study-related procedures and that the subject received a signed copy of the ICF/assent.

The following general rules apply but these may vary by local regulations for pediatric studies:

- The investigator/subinvestigator(s) is responsible for explaining the nature and purpose of the study as well as other study-related matters to subjects and their parent(s)/legal guardian(s), using the written information, and for obtaining the child's assent and the parent(s)'/guardian(s)' full understanding and written consent/assent to participate in the study of their own free will.
- In cases where there might be an explicit wish of a minor or an incapacitated adult, who is capable of forming an opinion and assessing this information, to refuse to participate or to be withdrawn from the clinical study at any time, this will have to be considered by the investigator, even if consent/assent is given by the parent(s)/legal guardian(s). Every effort should be made to understand and respect differences of opinion between the subject and their parent(s)/legal guardian(s). Strong and definitive objections from the child should be respected.
- The investigator or other responsible personnel who provided explanations (including collaborators who gave supportive information, if applicable) and the subject and

Sponsor: APGD ISN/Protocol: 178-CL-204

EudraCT number 2016-001767-37


parent(s)/legal guardian(s) should sign and date the written information, or write down his/her name, and date the form.

- Informed consent/assent must be obtained prior to any study-related procedures (including discontinuation of prohibited medication, if applicable). Consent/assent should be obtained from the subject and his/her parent(s)/legal guardian(s), before start of pre-investigational period. Consent/assent will be obtained per local regulations.
- The investigator or other responsible personnel must give a copy of the signed consent/assent form to the subject and parent(s)/legal guardian(s) and store the original appropriately in accordance with the rules at the study site concerned.
- The investigator or other responsible personnel should note the following when obtaining consent/assent from subjects and parent(s)/legal guardian(s):
  - No subject may be subjected to undue influence, such as compulsory enrollment into a study.
  - The language and expressions used in the written information should be as plain and understandable as possible. Subjects and their parent(s)/legal guardian(s) should be given the opportunity to ask questions and receive satisfactory answers to the inquiry and should have adequate time to decide whether or not to participate in the study. Written information should not contain any language or contents that causes the subject to waive or appears to waive any legal rights, or that releases/mitigates or appears to release/mitigate the study site, the investigator/subinvestigator(s), collaborators, or the sponsor from liability for negligence.

The signed ICFs/assents will be retained by the investigator and made available (for review only) to the study monitor, auditor and appropriate regulatory authorities and other applicable individuals upon request.

# 12.1.5.2 Supply of New and Important Information Influencing the Subject's Consent/Assent and Revision of the Written Information

- 1. The investigator or his/her representative will immediately inform the subject verbally whenever new information becomes available that may be relevant to the subject's consent/assent or may influence the subject's willingness to continue participating in the study (e.g., report of serious adverse drug reaction). The communication must be documented in the subject's medical records and whether the subject is willing to remain in the study or not must be confirmed and documented.
- 2. The investigator must update the subject's ICF/assent and submit it for approval to the IRB/IEC. The investigator or his/her representative must obtain written informed consent/assent from the subject on all updated ICFs/assents throughout their participation in the study. The investigator or his/her designee must reconsent subjects with the updated ICF/assent even if relevant information was provided verbally. The investigator or his/her representative who obtained the written informed consent/assent and the subject should sign and date the ICF/assent. A copy of the signed ICF/assent will be given to the subject and the original will be placed in the subject's medical record. An entry must be made in the subject's records documenting the reconsent process.


Sponsor: APGD ISN/Protocol: 178-CL-204

### 12.1.6 Source Documents

1. Source data must be available at the study site to document the existence of the subjects and to substantiate the integrity of study data collected. Source data must include the original documents relating to the study, as well as the medical treatment and medical history of the subject.

- 2. The investigator must maintain accurate documentation (source data) that supports the information entered in the CRF.
- 3. The investigator is responsible for ensuring the source data are attributable, legible, contemporaneous, original, accurate and complete whether the data are handwritten on paper or entered electronically. If source data are created (first entered), modified, maintained, achieved, retrieved or transmitted electronically via computerized systems (and/or other kind of electronic devices) as part of regulated study activities, such systems must be compliant with all applicable laws and regulations governing use of electronic records and/or electronic signatures. Such systems may include, but are not limited to, electronic medical/health records, protocol-related assessments, AE tracking, electronic clinical outcome assessment eCOA and/or drug accountability.
- 4. Paper records from electronic systems used in place of electronic format must be certified copies. A certified copy must be an exact copy and must have all the same attributes and information as the original. Certified copies must include signature and date of the individual completing the certification. Certified copies must be a complete and chronological set of study records (including notes, attachments, and audit trail information, if applicable). All printed records must be kept in the subject file and be available for archiving.
- 5. Study monitors will perform ongoing source data review to confirm that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP and all applicable regulatory requirements.

#### 12.1.7 Record Retention

The investigator will archive all study data (e.g., subject identification code list, source data electronic data source and investigator's file) and relevant correspondence. These documents are to be kept on file for the appropriate term determined by local regulation. The sponsor will notify the study site/investigator if the European Medicines Agency (EMA) is approved or if the IND/investigational medicinal product dossier is discontinued. The investigator agrees to obtain the sponsor's agreement prior to disposal, moving or transferring of any study-related records. The sponsor will archive and retain all documents pertaining to the study according to local regulations.

Data generated by the methods described in the protocol will be recorded in the subject's medical records and/or study progress notes.

The documents of the efficacy and safety evaluation committee (minutes and SOPs and others) and the judgment committee outside the study sites (minutes and SOPs and others) shall be retained by the sponsor.
ponsor: APGD ISN/Protocol: 178-CL-204

## 12.1.8 Subject Confidentiality and Privacy

Individual subject medical information obtained as a result of this study is considered confidential and disclosure to third parties is prohibited unless the subject provides written consent/assent or approval. Additional medical information may be given only after approval of the subject to the investigator or to other appropriate medical personnel responsible for the subject's well-being.

The sponsor shall not disclose any confidential information on subjects obtained during the performance of their duties in the study without justifiable reasons.

Even though any individuals involved in the study, including the study monitors and auditors, may get to know matters related to a subject's privacy due to direct access to source documents, or from other sources, they may not disclose the content to third parties.

The sponsor affirms the subject's right to protection against invasion of privacy. Only a subject identification number will identify subject data retrieved by the sponsor. However, the sponsor requires the investigator to permit the sponsor, sponsor's representative(s), the IRB/IEC and when necessary, representatives of the regulatory health authorities to review and/or to copy any medical records relevant to the study.

The sponsor agrees to comply and process personal data in accordance with all applicable privacy laws and regulations, including, without limitation, the Personal Information Protection Law in Japan and privacy laws in the US. If the services will involve the collection or processing of personal data (as defined by applicable data protection legislation) within the European Economic Area (EEA), then the sponsor shall serve as the controller of such data, as defined by the EU Data Protection Directive (DPD), and investigator and/or third party shall act only under the instructions of the sponsor in regard to personal data. If the sponsor is not based in the EEA, the sponsor must appoint a third party to act as its local data protection representative or arrange for a co-controller established in the EU for data protection purposes in order to comply with the DPD.

#### 12.1.9 Arrangement for Use of Information and Publication of the Study

Information concerning the test product, patent applications, processes, unpublished scientific data, the Investigator's Brochure and other pertinent information is confidential and remains the property of the sponsor. Details should be disclosed only to the persons involved in the approval or conduct of the study. The investigator may use this information for the purpose of the study only. It is understood by the investigator that the sponsor will use the information obtained during the study in connection with the development of the drug and therefore may disclose it as required to other clinical investigators or to regulatory agencies. In order to allow for the use of the information derived from this study, the investigator understands that he/she has an obligation to provide the sponsor with all data obtained during the study.

Publication of the study results is discussed in the study agreement.

Sponsor: APGD EudraCT number 2016-001767-37


## 12.1.10 Insurance of Subjects and Others

The sponsor has covered this study by means of an insurance of the study according to national requirements. The name and address of the relevant insurance company, the certificate of insurance, the policy number and the sum insured are provided in the investigator's file.

ISN/Protocol: 178-CL-204

#### 12.1.11 Signatory Investigator for Clinical Study Report

ICH E3 guidelines recommend and EU Directive 2001/83/EC requires that a final CSR that forms part of a marketing authorization application, be signed by the representative for the coordinating investigator(s) or the principal investigator(s). The representative for the coordinating investigator(s) or the principal investigator(s) will have the responsibility to review the final study results to confirm to the best of his/her knowledge it accurately describes the conduct and results of the study. The representative for the coordinating investigator(s) or the principal investigator(s) will be selected from the participating investigators by the sponsor prior to database hardlock.

#### 12.2 **Procedure for Study Quality Control**

#### 12.2.1 **Study Monitoring**

The sponsor is responsible for monitoring the study to ensure that the rights, safety and wellbeing of subjects are protected, the study is properly conducted in adherence to the current protocol and GCP. The sponsor is responsible for assigning the study monitor(s) to this study for proper monitoring. They will monitor the study in accordance with planned monitoring procedures.

#### 12.2.2 **Direct Access to Source Data/Documents**

The investigator and the study site must accept monitoring and auditing by the sponsor, as well as inspections from the IRB/IEC and appropriate regulatory authorities. In these instances, they must provide all study-related records including source documents when they are requested by the sponsor monitors and auditors, the CRO, the IRB/IEC or appropriate regulatory authorities. The confidentiality of the subject's identity shall be well protected consistent with local and national regulations when the source documents are subject to direct access

## 12.2.3 Data Management

Data management will be coordinated by the Data Science department or designee of the sponsor in accordance with the SOPs for data management. All study-specific processes and definitions will be documented by data management. Electronic data source completion will be described in the electronic data source instructions. Coding of medical terms and medications will be performed using MedDRA and the WHO Drug Dictionary, respectively. Data management is accountable for eCOA.

#### ISN/Protocol: 178-CL-204


## 12.2.4 Quality Assurance

The sponsor is implementing and maintaining quality assurance (QA) and quality control (QC) systems with written SOPs to ensure that studies are conducted and data are generated, documented, recorded, and reported in compliance with the protocol, GCP and applicable regulatory requirement(s). Where applicable, the QA and QC systems and written SOPs of the CRO will be applied.

The sponsor or sponsor's designee may arrange to audit the study at any or all study sites and facilities. The audit may include on-site review of regulatory documents, CRFs and source documents. Direct access to these documents will be required by the auditors.

To support quality around subject safety and reliability of study results, quality tolerance limits (QTLs) are defined and monitored. QTLs represent the acceptable variation of study data, taking into consideration the current state of medical and statistical knowledge about the variables to be analyzed as well as the statistical design of the study. It is a level, point, or value associated with a parameter that should trigger an evaluation if a deviation is detected to determine if there is a possible systematic issue (i.e., a trend has occurred). The QTLs defined for this study are provided below.

**Table 9 Quality Tolerance Limit** 

| Tuble 5 Quality Tolerance Zimit | | |
|---|---|---|
| QTL #: Name and Parameter | Definition | Parameter Justification |
| Subject ePRO diary completion: | Proportion (%) of randomized | If subject diaries are not completed |
| Proportion (%) of randomized | subject with missing number | accurately or are discrepant with |
| subjects who provide the number of | of micturitions in 7 days of | source data, there is a risk of |
| micturitions in 7 days of ePRO diary | diary data at week 4, week 8 | inaccurate data which may impact |
| data at week 4, week 8 and week 12. | and week 12. | primary endpoint. |
| Subject ePRO diary completion: | Proportion (%) of randomized | If subject diaries are not completed |
| Proportion (%) of randomized | subjects with missing urine | accurately or are discrepant with |
| subjects who provide urine volume | volume voided data over | source data, there is a risk of |
| voided data over 2 days of ePRO | 2 days of diary data at week 4, | inaccurate data which may impact |
| diary data at week 4, week 8 and | week 8 and week 12. | secondary endpoints. |
| week 12. | | |
| Subject ePRO diary completion: | Proportion (%) of randomized | If subject diaries are not completed |
| Proportion (%) of randomized | subjects with missing number | accurately or are discrepant with |
| subjects who provide number of dry | of dry days and number of wet | source data, there is a risk of |
| days and number of wet days for | days for 7 days of diary data at | inaccurate data which may impact |
| 7 days of ePRO diary data at week 4, | week 4, week 8 and week 12. | secondary endpoints. |
| week 8 and week 12. | | |
| Subject ePRO diary completion: | Proportion (%) of randomized | A high number of missing |
| Proportion (%) of randomized | subjects with missing | acceptability and palatability |
| subjects with missing acceptability | acceptability and palatability | questionnaire will have a negative |
| and palatability questionnaire at | questionnaire at week 12. | impact on the interpretation of the |
| week 12. | | secondary endpoints. |
| Pharmacokinetic sample results: | Proportion (%) of overall | A high number of missing |
| Proportion (%) missing week 4 and | planned sampling time points | pharmacokinetic sample results can |
| week 12 pharmacokinetic sample | with a missing result due to | have a negative impact on |
| results. | any reason, such as missed | interpretation of secondary endpoints. |
| | collection, lost or mishandled. | |

ePRO: electronic patient-reported outcome; QTL: quality tolerance limit

#### **QTL Management Activities:**

For control of risks associated with QTLs, refer to the Study Monitoring Plan.

# ponsor: APGD ISN/Protocol: 178-CL-204

## 12.3 Contraception Requirements

## **Contraception for Pediatric Male Subjects of Reproductive Potential**

Male children/adolescents in the following categories are not considered of reproductive potential:

- 1. Tanner stage 1 development
- 2. Documented surgically sterile

Documentation from the site personnel's review of the male subject's medical records, medical exam and medical history interview is necessary.

## Contraception guidance for male children/adolescents of reproductive potential:

- Male children/adolescents of reproductive potential (Tanner Stage 2 and above) receiving non-genotoxic agents should use a condom during treatment and for 3 weeks + 5 × half-life of drug after last dose.
- Male children/adolescents of reproductive potential receiving genotoxic agents should use a condom during treatment and for 90 days + 5 × half-life of drug after last dose.
- Male participants should inform their female partners that they are participating in a clinical trial and effective methods of contraception should be used.
- Female partners of male subjects who have not undergone bilateral orchiectomy should consider use of highly effective methods of contraception until the end of relevant systemic exposure, as defined above.

#### Contraception for Pediatric Female Subjects of Childbearing Potential

# Female children/adolescents in the following categories are not considered of childbearing potential:

- 1. Pre-menarchal
- 2. Documented surgically sterile (hysterectomy, bilateral salpingectomy, bilateral oophorectomy)

Documentation from the site personnel's review of the female subject's medical records, medical exam and medical history interview is necessary.

## Contraception guidance for female children/adolescents of childbearing potential:

- Female children/adolescents of childbearing potential receiving non-genotoxic agents should use highly effective contraception during treatment and for 30 days after last dose.
- Female children/adolescents of childbearing potential receiving genotoxic agents should use contraception during treatment and for 180 days + 5 × half-life of drug after last dose.
- Pregnancy testing for female children/adolescents of childbearing potential
  - o At all on-site visits and 30 days after end of relevant systemic exposure

Sponsor: APGD - CONFIDENTIAL -

EudraCT number 2016-001767-37

One of the highly effective methods of contraception listed below is required at the time of informed consent and until the end of relevant systemic exposure as defined above.

ISN/Protocol: 178-CL-204

## Highly Effective Birth Control Methods-failure rate < 1%/year

- 1. Combined estrogen and progestogen containing hormonal contraception
  - a. Oral
  - b. Intravaginal
  - c. Transdermal-Patch
  - d. Injectable-Cyclofem, Mesigyna
  - e. Intrauterine device
  - f. Intrauterine hormone-releasing system
- 2. Progestogen-only hormonal contraception
  - a. Oral
  - b. Injectable-DMPA-IM or -SC
  - c. Implantable-Norplant
- 3. Bilateral tubal occlusion
- 4. Vasectomized male partner
- True abstinence\*

\*True abstinence: When this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drug. It is not necessary to use any other method of contraception when complete abstinence is elected.

## Birth control methods considered unacceptable:

- 1. Periodic abstinence (calendar, symptothermal, post-ovulation methods)
- Withdrawal (coitus interruptus)
- 3. Spermicides only
- 4. Lactational amenorrhea

APGD ISN/Protocol: 178-CL-204

# 12.4 Adverse Events: Definitions and Procedures for Recording, Evaluating, Follow-up and Reporting

#### 12.4.1 Definition of Adverse Events

An AE is any untoward medical occurrence in a subject administered an IP, and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP whether or not considered related to the IP.

## 12.4.1.1 Abnormal Laboratory Findings

Any abnormal laboratory test result (e.g., hematology, biochemistry or urinalysis dipstick) or other safety assessment (e.g., vital signs, physical examination, ECGs or radiographic scans), including those that worsen from baseline should be considered to be reported as an (S)AE.

Any abnormal laboratory finding or other abnormal safety assessment, which is associated with the underlying disease or with concomitant medication, will not be considered an AE unless judged by the investigator to be more severe than expected for the subject's condition or not associated with the known side effects of the concomitant medication. Additionally, minor laboratory deviations or fluctuations outside of normal ranges of preexisting disease(s) or condition(s) present or detected at the start of the study that do not worsen and/or that are not reproducible with re-testing will not to be considered an AE.

Repeating an abnormal laboratory test or other safety assessment, in the absence of any of the above criteria, does not constitute an AE. Any abnormal test result that is determined to be an error does not require reporting as an AE.

## 12.4.1.2 Potential Cases of Drug-induced Liver Injury

Refer to [Appendix 12.5 Liver Safety Monitoring and Assessment] for detailed instructions on drug induced liver injury. Abnormal values in AST and/or ALT concurrent or with abnormal elevations in TBL that meet the criteria outlined in [Appendix 12.5 Liver Safety Monitoring and Assessment], in the absence of other causes of liver injury, are considered potential cases of drug-induced liver injury (potential Hy's Law cases) and are always to be considered important medical events and reported per [Appendix 12.4.5 Reporting Procedures for Serious Adverse Events].

#### 12.4.2 Definition of Serious Adverse Events

An AE is considered "serious" if, in the view of either the investigator or sponsor, the event:

- Results in death
- Is life-threatening (An AE is considered "life-threatening" if, in the view of either the investigator or sponsor, its occurrence places the subject at immediate risk of death; it does not include an AE that, had it occurred in a more severe form, might have caused death)

ISN/Protocol: 178-CL-204

- Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions
- Results in congenital anomaly, or birth defect
- Requires inpatient hospitalization (except for planned procedures as allowed per study) or leads to prolongation of hospitalization (except if prolongation of planned hospitalization is not caused by an AE)
- Other medically important events (defined in paragraph below)

Medical and scientific judgment should be exercised in deciding whether expedited reporting is appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalization, but may jeopardize the subject or may require intervention to prevent 1 of the other outcomes listed in the definition above. These events, including those that may result in disability/incapacity, usually are considered serious. Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

## 12.4.3 Criteria for Causal Relationship to Investigational Product

A medically qualified investigator is obligated to assess the relationship between IP and each occurrence of each (S)AE. This investigator will use medical judgment as well as the reference safety information [Section 2.1.3 Summary of Key Safety Information for Investigational Product(s)] to determine the relationship. The causality assessment is 1 of the criteria used when determining regulatory reporting requirements.

The investigator is requested to provide an explanation for the causality assessment for each (S)AE and must document in the medical notes that he/she has reviewed the (S)AE and has provided an assessment of causality.

Following a review of the relevant data, the causal relationship between the IP and each (S)AE will be assessed by answering "yes" or "no" to the question "Do you consider that there is a reasonable possibility that the event may have been caused by the IP?"

When making an assessment of causality, the following factors are to be considered when deciding if there is evidence and/or arguments to suggest there is a "reasonable possibility" that an (S)AE may have been caused by the IP (rather than a relationship cannot be ruled out) or if there is evidence to reasonably deny a causal relationship:

- Has the subject been administered IP?
- Plausibility (i.e., could the event have been caused by the suspect drug? Consider biologic and/or pharmacologic mechanism, half-life, literature evidence, drug class, preclinical and study data, etc.)
- Dechallenge/dose reduction/rechallenge:
  - Dechallenge: did the (S)AE resolve or improve after only stopping the dose of the suspect drug without any treatment?
  - Dose reduction: did the (S)AE resolve or improve after reducing the dose of the suspect drug?

Sponsor: APGD ISN/Protocol: 178-CL-204 EudraCT number 2016-001767-37


• Rechallenge: did the (S)AE reoccur if the suspected drug was reintroduced after having been stopped?

- Laboratory or other test results: a specific lab investigation supports the assessment of the relationship between the (S)AE and the IP (e.g., based on values pre-, during and post-treatment)
- Available alternative explanations independent of IP exposure; such as other concomitant drugs, past medical history, concurrent or underlying disease, risk factors including medical and family history, season, location, etc., and strength of the alternative explanation
- Finally, judging which are more likely based on all the above contents, factors of reasonable possibility or confounding factors, comprehensive judgment of plausible temporal relationship between exposure to the IP and (S)AE onset and/or resolution will be provided. Did the (S)AE occur in a reasonable temporal relationship to the administration of the IP?

There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report to the sponsor. However, it is very important that the investigator always assesses causality for every event before the initial transmission of the SAE data to the sponsor. With limited or insufficient information about the event to make an informed medical judgment and in absence of any indication or evidence to establish a causal relationship, a causality assessment of "no" is to be considered. In such instance, the investigator is expected to obtain additional information regarding the event as soon as possible and to re-evaluate the causality upon receipt of additional information. The medically qualified investigator may revise his/her assessment of causality in light of new information regarding the SAE and shall send an SAE follow-up report and update the electronic data source with the new information and updated causality assessment.

#### 12.4.4 Criteria for Defining the Severity of an Adverse Event

The investigator will use the following definitions to rate the severity of each AE:

- Mild: No disruption of normal daily activities
- Moderate: Affects normal daily activities
- Severe: Inability to perform daily activities

## 12.4.5 Reporting Procedures for Serious Adverse Events

The investigator must complete and submit an SAE worksheet containing all information that is required by local and/or regional regulations to the sponsor by fax or email immediately (within 24 hours of awareness).

The SAE worksheet must be signed by a medically qualified investigator (as identified on delegation of authority log). Signature confirms accuracy and completeness of the SAE data as well as the investigator causality assessment including the explanation for the causality assessment.

If the SAE is associated with emergency unblinding by the investigator as outlined in [Section 6.3.4 Breaking the Treatment Code for Emergency], this is to be recorded on the 11 Feb 2021 Astellas 

Sponsor: APGD EudraCT number 2016-001767-37


SAE worksheet. On the SAE worksheet, the investigator is to include when unblinding took place in association with the SAE.

ISN/Protocol: 178-CL-204

For contact details, see [Contact Details of sponsor's Key Personnel]. Fax or email the SAE/special situations worksheet to:

Astellas Pharma Global Development Inc.
US Pharmacovigilance
North America fax number: +1-888-396-3750
North America alternate fax number: +1-847-317-1241
International fax number: +44 800 471 5263
Email: safety-us@astellas.com

If there are any questions, or if clarification is needed regarding the SAE, please contact the sponsor's medical monitor/study physician or their designee [Contact Details of Sponsor's Key Personnel].

Follow-up information for the event should be sent promptly (as soon as available but no longer than within 7 days of the initial notification).

Full details of the SAE should be recorded on the medical records, SAE/special situation worksheet and on the electronic data source.

The following minimum information is required:

- International study number/study number
- Subject number, sex and age
- Date of report
- Description of the SAE (event and seriousness criteria)
- Causal relationship to the IP (including reason)
- Blinded regimen

The sponsor or sponsor's designee will medically evaluate the SAE and determine if the report meets the requirements for expedited reporting based on seriousness, causality, and expectedness of the events (e.g., SUSAR reporting) according to current local/regional regulatory requirements. The sponsor or sponsor's designee will submit expedited safety reports to competent authorities and concerned ethics committee per current local regulations and will inform the investigators of such regulatory reports as required. Investigators must submit safety reports as required by their IRB/IEC within timelines set by regional regulations (e.g., EMA, FDA) where required. Documentation of the submission to and receipt by the IRB/IEC of expedited safety reports should be retained by the study site. In the US, FDA expedited IND reporting guidelines will be followed.

The sponsor will notify all investigators responsible for ongoing clinical studies with the test product of all SUSARs, which require submission per local requirements IRB/IEC.

The investigators should provide written documentation of IRB/IEC notification for each report to the sponsor.

ISN/Protocol: 178-CL-204

The investigator may contact the sponsor's medical monitor/study physician for any other problem related to the rights, safety or well-being of the subject.

### 12.4.6 Reporting Procedures for Special Situations

## **12.4.6.1 Pregnancy**

If a female subject becomes pregnant during the study dosing period or within 30 days from the discontinuation of dosing, the investigator is to report the information to the sponsor according to the timelines in [Appendix 12.4.5 Reporting Procedures for Serious Adverse Events using the SAE worksheet as a special situation and in the electronic data source.

The investigator will attempt to collect pregnancy information on any female partner of a male subject who becomes pregnant during the study dosing period or within 30 days from the discontinuation of dosing and report the information to the sponsor according to the timelines in [Appendix 12.4.5 Reporting Procedures for Serious Adverse Events] using the SAE worksheet as a special situation.

The expected date of delivery or expected date of the end of the pregnancy, last menstruation, estimated conception date, pregnancy result and neonatal data, etc., should be included in this information.

While pregnancy itself is not considered to be an AE or SAE, any pregnancy complication or termination (including elective termination) of a pregnancy is to be reported for a female subject as an AE in the electronic data source or SAE per [Appendix 12.4.5 Reporting Procedures for Serious Adverse Events]. For (S)AEs experienced by a female partner of a male subject, (S)AEs are to be reported via the SAE worksheet.

Additional information regarding the outcome of a pregnancy when also categorized as an SAE is mentioned below:

- "Spontaneous abortion" includes miscarriage, abortion and missed abortion
- Death of a newborn or infant within 1 month after birth is to be reported as an SAE regardless of its relationship with the IP
- If an infant die more than 1 month after the birth, it is to be reported if a relationship between the death and intrauterine exposure to the IP is judged as "possible" by the investigator
- Congenital anomaly (including anomaly in miscarried fetus)

Unless a congenital anomaly is identified prior to spontaneous abortion or miscarriage, the embryo or fetus should be assessed for congenital defects by visual examination or other means as appropriate. (S)AEs experienced by the newborn/infant should be reported via the pregnancy reporting form. Generally, follow up will be no longer than 6 to 8 weeks following the estimated delivery date.

#### 12.4.6.2 Lack of Efficacy

Not applicable.

Sponsor: APGD ISN/Protocol: 178-CL-204

## 12.4.6.3 Medication Error, Overdose and "Off-label Use"

If a medication error (defined as an unintended failure in the treatment process that leads to, or has the potential to lead to, harm to the subject), overdose or "off-label use" (i.e., use outside of what is stated in the protocol) is suspected, refer to [Section 10.3 Major Protocol Deviations]. Any associated (S)AEs are to be reported in the electronic data source. If the AE meets the definition of an SAE, the SAE is also to be reported as described in [Appendix 12.4.5 Reporting Procedures for Serious Adverse Events] together with the details of the medication error, overdose and/or "off-label use."

In the event of suspected overdose, refer to the approved package insert, summary of product characteristics, or local product information supplied by the manufacturer for each IP.

## 12.4.6.4 Misuse/Abuse

Definition of misuse: Situations where the IP is/are intentionally and inappropriately used not in accordance with the intended use as defined in the protocol.

Definition of abuse: Persistent or sporadic, intentional excessive use of medicinal products which is accompanied by harmful physical or psychological effects.

If misuse or abuse of the IP is suspected, the investigator must forward the special situation worksheet to the sponsor by fax or email immediately (within 24 hours of awareness). Any associated (S)AEs are to be reported in the electronic data source. If the AE meets the definition of an SAE, the SAE is also to be reported as described in [Appendix 12.4.5 Reporting Procedures for Serious Adverse Events] together with details of the misuse or abuse of the IP.

## 12.4.6.5 Occupational Exposure

If occupational exposure (e.g., inadvertent exposure to the IP of study site personnel while preparing it for administration to the subject) to the IP occurs, the investigator must forward the special situation worksheet to the sponsor by fax or email immediately (within 24 hours of awareness). Any associated (S)AEs occurring to the individual associated with or resulting from the special situation are to be reported on the special situations worksheet.

## 12.4.6.6 (Suspicion of) Transmission of Infectious Agent

Not applicable.

#### 12.4.6.7 Suspected Drug-drug Interaction

If a drug-drug interaction associated with the IP is suspected, the investigator must forward the special situation worksheet to the sponsor by fax or email immediately (within 24 hours of awareness). Any associated (S)AEs are to be reported in the electronic data source. If the AE meets the definition of an SAE, the SAE is also to be reported as described in [Appendix 12.4.5 Reporting Procedures for Serious Adverse Events] together with details of the suspected drug-drug interaction.

## Sponsor: APGD ISN/Protocol: 178-CL-204

## 12.5 Liver Safety Monitoring and Assessment

The purpose of this appendix is to provide guidance for the monitoring of drug-induced liver injury during the course of the study. It should be noted that this section does not specify the EoS analyses of liver enzymes. The EoS liver enzymes analyses will be described in the SAP. Any subject enrolled in a study with active drug therapy and reveals an increase of serum aminotransferases (AT) to  $> 3 \times \text{ULN}$  or bilirubin  $> 2 \times \text{ULN}$  should undergo detailed testing for liver enzymes (including at least alkaline phosphatase [ALP], ALT, AST and TBL). Testing should be repeated within 72 hours of notification of the test results. For studies for which a central laboratory is used, alerts will be generated by the central laboratory regarding moderate and severe liver abnormality to inform the investigator and study team. Subjects should be asked if they have any symptoms suggestive of hepatobiliary dysfunction.

## **Definition of Liver Abnormalities**

Confirmed abnormalities will be characterized as moderate and severe where ULN is as shown below.

**Table 10** Moderate and Severe Liver Abnormalities

| | ALT or AST | | TBL |
|----------|------------|------|-----------|
| Moderate | > 3 × ULN | or | > 2 × ULN |
| Severe | > 3 × ULN | and† | > 2 × ULN |

ALT: alanine aminotransferase; AST: aspartate aminotransferase; TBL: total bilirubin; ULN: upper limit of normal

In addition, the subject should be considered to have severe hepatic abnormalities for any of the following:

- ALT or AST  $> 8 \times ULN$
- ALT or AST  $> 5 \times$  ULN for more than 2 weeks
- ALT or AST >  $3 \times \text{ULN}$  and  $\dagger$  and TBL >  $2 \times \text{ULN}$  or international normalized ratio (INR) > 1.5 (if INR testing is applicable/evaluated)
- ALT or AST  $> 3 \times$  ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash and/or eosinophilia (> 5%)
- † Samples taken simultaneously or within a maximum of 24 hours.

The investigator may determine that abnormal liver function results, other than as described above, may qualify as moderate or severe abnormalities and require additional monitoring and follow-up.

## **Follow-up Procedures**

Confirmed moderate and severe abnormalities in hepatic functions should be thoroughly characterized by obtaining appropriate expert consultations, detailed pertinent history, physical examination and clinical laboratory tests. The study site personnel are to complete the liver abnormality case report form (LA-CRF). Subjects with confirmed abnormal liver function testing should be followed as described below.

11 Feb 2021 Astellas 

<sup>†</sup> Samples taken simultaneously or within maximum 24 hours.

Sponsor: APGD ISN/Protocol: 178-CL-204

Confirmed moderately abnormal liver function tests should be repeated 2 to 3 times weekly, and then weekly or less if abnormalities stabilize or the IP has been discontinued and the subject is asymptomatic.

Severe hepatic liver function abnormalities as defined above, in the absence of another etiology, may be considered an important medical event and may be reported as a SAE. The sponsor should be contacted and informed of all subjects for whom severe hepatic liver function abnormalities possibly attributable to IP are observed.

To further assess abnormal hepatic laboratory findings, the investigator is expected to:

- Obtain a more detailed history of symptoms and prior or concurrent diseases. Symptoms and new-onset diseases are to be recorded as "AEs" within the electronic data source. Illnesses and conditions such as hypotensive events and decompensated cardiac disease that may lead to secondary liver abnormalities should be noted. Nonalcoholic steatohepatitis is seen in obese hyperlipoproteinemic and/or diabetic subjects and may be associated with fluctuating AT levels. The investigator should ensure that the medical history form captures any illness that predates study enrollment that may be relevant in assessing hepatic function.
- Obtain a history of concomitant drug use (including nonprescription medication, complementary and alternative medications), alcohol use, recreational drug use and special diets. Medications are to be entered in the electronic data source. Information on alcohol, other substance use and diet should be entered on the LA-CRF or an appropriate document.
- Obtain a history of exposure to environmental chemical agents.
- Based on the subject's history, other testing may be appropriate including:
  - Acute viral hepatitis (A, B, C, D, E or other infectious agents)
  - Ultrasound or other imaging to assess biliary tract disease
  - Other clinical laboratory tests, including INR and direct bilirubin
- Consider gastroenterology or hepatology consultations.
- Submit results for any additional testing and possible etiology on the LA-CRF or an appropriate document.

#### **Study Treatment Discontinuation**

In the absence of an explanation for increased liver function tests, such as viral hepatitis, preexisting or acute liver disease, or exposure to other agents associated with liver injury, the subject may be discontinued from study treatment. The investigator may determine that it is not in the subject's best interest to continue study treatment. Discontinuation of study treatment should be considered if:

- ALT or AST  $> 8 \times ULN$
- ALT or AST  $> 5 \times ULN$  for more than 2 weeks
- ALT or AST >  $3 \times \text{ULN}$  and † TBL >  $2 \times \text{ULN}$  or INR > 1.5) (if INR testing is applicable/evaluated)

Sponsor: APGD ISN/Protocol: 178-CL-204 EudraCT number 2016-001767-37


• ALT or AST  $> 3 \times$  ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash and/or eosinophilia (> 5%)

† Samples taken simultaneously or within a maximum of 24 hours.

In addition, if close monitoring for a subject with moderate or severe hepatic laboratory tests is not possible, study treatment should be discontinued.

Hy's Law definition: Drug-induced jaundice caused by hepatocellular injury, without a significant obstructive component, has a high rate of bad outcomes, from 10% to 50% mortality (or transplant).

The 2 "requirements" for Hy's Law are:

- 1. Evidence that a drug can cause hepatocellular-type injury, generally shown by an increase in AT elevations > 3 × ULN ("2 × ULN elevations are too common in treated and untreated subjects to be discriminating").
- 2. Cases of increased TBL (at least 2 × ULN) with concurrent AT elevations at least 3 × ULN and no evidence of intra- or extra-hepatic bilirubin obstruction (elevated ALP) or Gilbert's syndrome [Temple, 2006].

FDA Guidance for Industry titled, "Drug-induced Liver Injury: Premarketing Clinical Evaluation" issued by the FDA on July 2009:

- 1. The drug causes hepatocellular injury, generally shown by a higher incidence of 3-fold or greater elevations above the ULN of ALT or AST than the (nonhepatotoxic) control drug or placebo.
- 2. Among subjects showing such AT elevations, often with ATs much greater than  $3 \times \text{ULN}$ , 1 or more also show elevation of serum TBL to  $> 2 \times \text{ULN}$ , without initial findings of cholestasis (elevated serum ALP).
- 3. No other reason can be found to explain the combination of increased AT and TBL, such as viral hepatitis A, B or C; preexisting or acute liver disease; or another drug capable of causing the observed injury.

## References

Temple R. Hy's Law: Predicting Serious Hepatotoxicity. Pharmacoepidemiol Drug Saf. 2006; 15:241-3.

ISN/Protocol: 178-CL-204

## 12.6 List of Excluded Concomitant Medications

Any medication used for the management of OAB (including tricyclic antidepressants, 1<sup>st</sup> generation H1-antagonists and alpha-blockers) and any drugs that are sensitive CYP2D6 substrates with a narrow therapeutic index and sensitive P-gp substrates.

Use of these medications is not permitted during the study phase. This list is <u>not exhaustive</u>. In case of doubt, the investigator should contact the local study monitor.

| Anticholinergics/antimuscarinics | Tricyclic/heterocyclic antidepressants | 1 <sup>st</sup> generation H1-antagonists† |
|---|---|---|
| Darifenacin | Alimemazine /Trimipramine | Tripelennamine |
| Dicyclomine/Dicycloverine | Amitriptyline | Dimenhydrinate |
| Fesoterodine | Amoxapine | Clemastine |
| Flavoxate | Clomipramine | Bromazine |
| Isopropamide | Desipramine | Orphenadrine |
| Oxybutynin | Dosulepin/Dothiepin | Doxylamine |
| Oxyphencyclimine | Doxepine | Carbinoxamine |
| Propantheline | Imipramine | Diphenhydramine |
| Propiverine | Lofepramine | Cyclizine |
| Tolterodine | Maprotiline | Chlorcyclizine |
| Trospium | Mianserin | Hydroxyzine |
| Solifenacin | Mirtazapine | Meclizine |
| | Nortriptyline | |
| | Protriptyline | |
| Alpha-blockers | CYP2D6 with narrow therapeutic index | Sensitive P-gp substrates |
| Tamsulosin | Thioridazine | Digoxin |
| Alfuzosin | Flecainide | Dabigatran |
| Doxazosin | Propafenone | |
| Terazosin | Imipramine | |
| Silodosin | Desipramine | |
| Moderate CYP3A4 inhibitors | Strong CYP3A4 inhibitors | Moderate CYP3A4 inducers |
| Fluconazole | Itraconazole | Cenobamate |
| Ciprofloxacin | Ketoconazole | Tipranavir |
| Erythromycin | Ritonavir | Ritonavir |
| Clotrimazole | Clarthromycin | Thioridazine |
| Fluvoxamine | Voriconazole | Rifabutin |
| Verapamil | Posaconazole | Nafeillin |
| Dronedarone | Troleandomycin | Lopinavir |
| Cimetidine | Telithromycin | Modafinil |
| Grapefruit Juice | | Phenobarbital |
| Table continued on next page | | |

Sponsor: APGD ISN/Protocol: 178-CL-204 EudraCT number 2016-001767-37


| Strong CYP3A4 inducers | P-gp inhibitors‡ | P-gp Inducers‡ |
|---|---|---|
| Rifampin | Amiodarone | Rifampin |
| Rifapentine | Carvedilol | Carbamazepine |
| Phenytoin | Clarithromycin | Dexamethasone |
| Carbamazepine | Dronedarone | Phenobarbital |
| St. John's wort | Itraconazole | Phenytoin |
| | Lopinavir, Ritonavir | Rifampicin |
| | Quinidine | St. John's wort |
| | Verapamil | Trazodone |
| QT prolongating medications | Other | |
| Amiodarone | Mirabegron (except for study drug) | |
| Sotalol | Botulinum toxin | |
| Quinidine | Opioids | |
| Levofloxacin, Ciprofloxacin | | |
| Clarithromycin, Erythromycin | | |
| Ketoconazole, Itraconazole | | |
| Amitriptyline, Fluoxetine | | |
| Haloperidol, Droperidol | | |
| Cisapride | | |
| Sumatriptan, Zolmitriptan | | |

P-gp: P-glycoprotein

 $<sup>\</sup>dagger$  Incidental use for motion sickness is accepted.

<sup>‡</sup> Moderate or strong not specified.

Sponsor: APGD EudraCT number 2016-001767-37


# 12.7 Laboratory Assessments

Laboratory tests will be performed according to the schedule of assessments and sent to a central laboratory for analysis.

ISN/Protocol: 178-CL-204

**Table 11** Clinical Laboratory Tests

| Panel/Assessments | Parameters to be Analyzed |
|-------------------|-------------------------------------------|
| Hematology | Hematocrit |
| | Hemoglobin |
| | Mean corpuscular volume |
| | Mean corpuscular hemoglobin |
| | Mean corpuscular hemoglobin concentration |
| | Platelets |
| | Red blood cell count |
| | White blood cell count |
| | White blood cell count differential |
| Biochemistry | Albumin |
| | Alanine aminotransferase |
| | Alkaline phosphatase |
| | Aspartate aminotransferase |
| | Bicarbonate |
| | Blood urea nitrogen |
| | Calcium |
| | Chloride |
| | Corrected serum calcium |
| | Creatinine |
| | Creatinine kinase |
| | Glucose |
| | Lactate dehydrogenase |
| | Magnesium |
| | Phosphate |
| | Potassium |
| | Serum hCG for female subjects |
| | Sodium |
| | Total bilirubin (total and direct) |
| | Total protein |
| Urinalysis | Leukocyte esterase |
| | Nitrites |
| | рН |
| | Protein |
| | Red blood cells |

hCG: human chorionic gonadotropin

# 12.8 Acceptability and Palatability Questionnaire for Tablets

| | | Questions | | |
|---|---|---|---|---|
| 1. How was t | 1. How was the <u>TASTE</u> of the study drug? | | | |
| 0 | 1 | 2 | 3 | 4 |
| Really bad | Bad | Not bad, not<br>good | Good | Really good |
| 2. How was i | t to <u>SWALLOV</u> | $\underline{\mathbf{V}}$ the study drug? | | |
| 0 | 1 | 2 | 3 | 4 |
| | $(\widetilde{})$ | $\left(\frac{3}{2}\right)$ | $(\mathbb{Z})$ | |
| Really difficult | Difficult | Not difficult,<br>not easy | Easy | Really easy |
| | | not easy | | |

# 12.9 Acceptability and Palatability Questionnaire for Oral Suspension

| | | Questions | Questions | |
|---|---|---|---|---|
| 1. How was t | the <u>TASTE</u> of th | e study drug? | | |
| 0 | 1 | 2 | 3 | 4 |
| | | | | $\odot$ |
| Really bad | Bad | Not bad, not<br>good | Good | Really good |
| 2. How was t | he <u>SMELL</u> of tl | ne study drug? | | |
| 0 | 1 | 2 | 3 | 4 |
| Really bad | Bad | Not bad, not | Good | Really Good |
| | | good | | |
| 3. How was i | t to <u>TAKE</u> the s | tudy drug? | | |
| 0 | 1 | 2 | 3 | 4 |
| Really difficult | Difficult | Not difficult, not easy | Easy | Really easy |
| | | not easy | | |

ISN/Protocol: 178-CL-204

Sponsor: APGD EudraCT number 2016-001767-37


| 4. How was it to PREPARE the study drug? | | | | |
|---|---|---|---|---|
| 0 | 1 | 2 | 3 | 4 |
| Really difficult | Difficult | Not difficult,<br>not easy | Easy | Really easy |

# 12.10 Centiles of Heart Rate for Normal Children from Birth to 18 Years of Age



# 12.11 Centers for Disease Control and Prevention Data Table of Stature for Age Chart for Males

## Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 24 | 79.91084 | 80.72977 | 81.99171 | 84.10289 | 86.4522 | 88.80525 | 90.92619 | 92.19688 | 93.02265 |
| 24.5 | 80.26037 | 81.08868 | 82.36401 | 84.49471 | 86.86161 | 89.22805 | 91.35753 | 92.63177 | 93.45923 |
| 25.5 | 81.00529 | 81.83445 | 83.11387 | 85.25888 | 87.65247 | 90.05675 | 92.22966 | 93.53407 | 94.38278 |
| 26.5 | 81.73416 | 82.56406 | 83.84716 | 86.00517 | 88.42326 | 90.8626 | 93.07608 | 94.40885 | 95.27762 |
| 27.5 | 82.44846 | 83.27899 | 84.56534 | 86.73507 | 89.17549 | 91.64711 | 93.89827 | 95.25754 | 96.14512 |
| 28.5 | 83.14945 | 83.98045 | 85.26962 | 87.44977 | 89.91041 | 92.41159 | 94.69757 | 96.08149 | 96.98663 |
| 29.5 | 83.83819 | 84.66948 | 85.96098 | 88.15028 | 90.62908 | 93.15719 | 95.47522 | 96.88198 | 97.80345 |
| 30.5 | 84.51558 | 85.34694 | 86.64027 | 88.83745 | 91.33242 | 93.88496 | 96.23239 | 97.66027 | 98.59691 |
| 31.5 | 85.18238 | 86.01357 | 87.3082 | 89.51202 | 92.02127 | 94.59585 | 96.97022 | 98.41758 | 99.36828 |
| 32.5 | 85.83925 | 86.66999 | 87.9654 | 90.17464 | 92.69638 | 95.2908 | 97.68978 | 99.15514 | 100.1189 |
| 33.5 | 86.48678 | 87.3168 | 88.61244 | 90.82592 | 93.35847 | 95.97068 | 98.39218 | 99.87416 | 100.8501 |
| 34.5 | 87.12552 | 87.95452 | 89.24986 | 91.46645 | 94.00823 | 96.63637 | 99.07848 | 100.5759 | 101.5631 |
| 35.5 | 87.75597 | 88.58366 | 89.87816 | 92.0968 | 94.64637 | 97.28875 | 99.74979 | 101.2615 | 102.2593 |
| 36.5 | 88.37864 | 89.20473 | 90.49789 | 92.71756 | 95.27359 | 97.9287 | 100.4072 | 101.9324 | 102.9402 |
| 37.5 | 88.93297 | 89.77301 | 91.08608 | 93.3344 | 95.91475 | 98.58525 | 101.069 | 102.593 | 103.5983 |
| 38.5 | 89.47916 | 90.33306 | 91.66589 | 93.94268 | 96.54734 | 99.23358 | 101.7234 | 103.247 | 104.2503 |
| 39.5 | 90.01766 | 90.88532 | 92.23779 | 94.54291 | 97.17191 | 99.87426 | 102.3709 | 103.8948 | 104.8967 |
| 40.5 | 90.54891 | 91.43025 | 92.80225 | 95.13557 | 97.78898 | 100.5078 | 103.012 | 104.537 | 105.538 |
| 41.5 | 91.07337 | 91.96832 | 93.35972 | 95.72115 | 98.39903 | 101.1348 | 103.6473 | 105.1739 | 106.1747 |
| 42.5 | 91.59152 | 92.49999 | 93.91068 | 96.30009 | 99.00254 | 101.7556 | 104.2771 | 105.8061 | 106.8071 |
| 43.5 | 92.10382 | 93.0257 | 94.45556 | 96.87286 | 99.59998 | 102.3708 | 104.9021 | 106.434 | 107.4357 |
| 44.5 | 92.61073 | 93.54592 | 94.99482 | 97.43989 | 100.1918 | 102.9807 | 105.5225 | 107.0579 | 108.0609 |
| 45.5 | 93.11271 | 94.06109 | 95.52888 | 98.00159 | 100.7783 | 103.5858 | 106.1387 | 107.6784 | 108.683 |
| 46.5 | 93.61022 | 94.57166 | 96.05817 | 98.55838 | 101.36 | 104.1865 | 106.7513 | 108.2956 | 109.3024 |
| 47.5 | 94.10371 | 95.07806 | 96.5831 | 99.11064 | 101.9373 | 104.7831 | 107.3604 | 108.9101 | 109.9193 |
| 48.5 | 94.59361 | 95.5807 | 97.10407 | 99.65875 | 102.5105 | 105.3759 | 107.9665 | 109.522 | 110.5342 |
| 49.5 | 95.08035 | 96.08 | 97.62147 | 100.2031 | 103.0799 | 105.9654 | 108.5698 | 110.1317 | 111.1473 |
| 50.5 | 95.56435 | 96.57635 | 98.13566 | 100.7439 | 103.6459 | 106.5518 | 109.1706 | 110.7394 | 111.7588 |
| 51.5 | 96.046 | 97.07013 | 98.64701 | 101.2817 | 104.2087 | 107.1354 | 109.7693 | 111.3454 | 112.369 |
| 52.5 | 96.52568 | 97.5617 | 99.15585 | 101.8166 | 104.7687 | 107.7165 | 110.366 | 111.95 | 112.9781 |
| 53.5 | 97.00376 | 98.05141 | 99.6625 | 102.3491 | 105.3262 | 108.2953 | 110.9609 | 112.5533 | 113.5863 |
| 54.5 | 97.48058 | 98.53958 | 100.1673 | 102.8792 | 105.8813 | 108.872 | 111.5543 | 113.1555 | 114.1937 |
| 55.5 | 97.95648 | 99.02654 | 100.6705 | 103.4074 | 106.4343 | 109.4469 | 112.1464 | 113.7568 | 114.8006 |

## Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 56.5 | 98.43175 | 99.51256 | 101.1723 | 103.9339 | 106.9855 | 110.0201 | 112.7374 | 114.3574 | 115.4072 |
| 57.5 | 98.90667 | 99.99791 | 101.6731 | 104.4588 | 107.535 | 110.5919 | 113.3273 | 114.9575 | 116.0134 |
| 58.5 | 99.38151 | 100.4828 | 102.173 | 104.9825 | 108.083 | 111.1623 | 113.9164 | 115.557 | 116.6194 |
| 59.5 | 99.8565 | 100.9676 | 102.6723 | 105.505 | 108.6296 | 111.7316 | 114.5047 | 116.1561 | 117.2254 |
| 60.5 | 100.3318 | 101.4523 | 103.1712 | 106.0265 | 109.1751 | 112.2998 | 115.0924 | 116.755 | 117.8314 |
| 61.5 | 100.8077 | 101.9372 | 103.6697 | 106.5472 | 109.7196 | 112.8671 | 115.6795 | 117.3536 | 118.4374 |
| 62.5 | 101.2843 | 102.4225 | 104.1682 | 107.0673 | 110.2631 | 113.4335 | 116.2661 | 117.9521 | 119.0435 |
| 63.5 | 101.7618 | 102.9082 | 104.6666 | 107.5868 | 110.8058 | 113.9992 | 116.8522 | 118.5505 | 119.6498 |
| 64.5 | 102.2401 | 103.3945 | 105.1651 | 108.1058 | 111.3477 | 114.5641 | 117.438 | 119.1487 | 120.2562 |
| 65.5 | 102.7195 | 103.8814 | 105.6638 | 108.6244 | 111.889 | 115.1284 | 118.0234 | 119.7469 | 120.8627 |
| 66.5 | 103.2 | 104.369 | 106.1627 | 109.1427 | 112.4296 | 115.6921 | 118.6084 | 120.345 | 121.4694 |
| 67.5 | 103.6815 | | 106.6619 | 109.6607 | 112.9696 | 116.2551 | 119.1931 | 120.943 | 122.0761 |
| 68.5 | 104.1642 | 105.3466 | 107.1614 | 110.1785 | 113.509 | 116.8176 | 119.7774 | 121.5408 | 122.6829 |
| 69.5 | 104.6479 | 105.8364 | 107.6611 | 110.696 | 114.0479 | 117.3794 | 120.3613 | 122.1384 | 123.2897 |
| 70.5 | 105.1326 | 106.327 | 108.1612 | 111.2132 | 114.5861 | 117.9407 | 120.9447 | 122.7359 | 123.8965 |
| 71.5 | 105.6183 | 106.8182 | 108.6614 | 111.7302 | 115.1238 | 118.5012 | 121.5277 | 123.333 | 124.5031 |
| 72.5 | 106.1048 | 107.3099 | 109.1619 | 112.2469 | 115.6609 | 119.0611 | 122.1101 | 123.9297 | 125.1095 |
| 73.5 | 106.5921 | 107.8021 | 109.6624 | 112.7631 | 116.1973 | 119.6203 | 122.6918 | 124.526 | 125.7156 |
| 74.5 | 107.0799 | 108.2946 | 110.1629 | 113.2789 | 116.7329 | 120.1786 | 123.2729 | 125.1217 | 126.3212 |
| 75.5 | 107.5682 | 108.7873 | 110.6633 | 113.7942 | 117.2678 | 120.7361 | 123.8532 | 125.7168 | 126.9263 |
| 76.5 | 108.0566 | 109.2801 | 111.1634 | 114.3089 | 117.8018 | 121.2926 | 124.4327 | 126.3111 | 127.5307 |
| 77.5 | 108.5451 | 109.7727 | 111.6631 | 114.8229 | 118.3348 | 121.848 | 125.0111 | 126.9045 | 128.1344 |
| 78.5 | 109.0335 | 110.2649 | 112.1623 | 115.336 | 118.8668 | 122.4024 | 125.5884 | 127.4969 | 128.7371 |
| 79.5 | 109.5214 | 110.7566 | 112.6608 | 115.8481 | 119.3977 | 122.9555 | 126.1646 | 128.0882 | 129.3387 |
| 80.5 | 110.0086 | 111.2476 | 113.1583 | 116.3592 | 119.9272 | 123.5073 | 126.7394 | 128.6782 | 129.9391 |
| 81.5 | 110.495 | 111.7375 | 113.6548 | 116.869 | 120.4554 | 124.0576 | 127.3128 | 129.2668 | 130.5381 |
| 82.5 | 110.9801 | 112.2263 | 114.1499 | 117.3774 | 120.9821 | 124.6064 | 127.8846 | 129.8538 | 131.1356 |
| 83.5 | 111.4638 | 112.7135 | 114.6436 | 117.8842 | 121.5072 | 125.1535 | 128.4547 | 130.4392 | 131.7314 |
| 84.5 | 111.9459 | 113.1991 | 115.1356 | 118.3893 | 122.0305 | 125.6987 | 129.023 | 131.0226 | 132.3253 |
| 85.5 | 112.4259 | 113.6827 | 115.6257 | 118.8926 | 122.552 | 126.2421 | 129.5893 | 131.6041 | 132.9172 |
| 86.5 | 112.9036 | 114.1642 | 116.1136 | 119.3938 | 123.0714 | 126.7834 | 130.1535 | 132.1834 | 133.507 |
| 87.5 | 113.3789 | 114.6431 | 116.5992 | 119.8927 | 123.5886 | 127.3225 | 130.7154 | 132.7605 | 134.0943 |
| 88.5 | 113.8513 | 115.1194 | 117.0822 | 120.3893 | 124.1035 | 127.8594 | 131.275 | 133.335 | 134.6792 |

## Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 89.5 | 114.3206 | 115.5927 | 117.5625 | 120.8833 | 124.616 | 128.3937 | 131.8321 | 133.907 | 135.2615 |
| 90.5 | 114.7867 | 116.0629 | 118.0398 | 121.3746 | 125.1259 | 128.9256 | 132.3865 | 134.4763 | 135.8409 |
| 91.5 | 115.2491 | 116.5297 | 118.5139 | 121.863 | 125.6331 | 129.4547 | 132.9381 | 135.0426 | 136.4173 |
| 92.5 | 115.7077 | 116.9928 | 118.9847 | 122.3483 | 126.1374 | 129.981 | 133.4868 | 135.606 | 136.9906 |
| 93.5 | 116.1623 | 117.4521 | 119.4519 | 122.8305 | 126.6388 | 130.5044 | 134.0325 | 136.1662 | 137.5607 |
| 94.5 | 116.6127 | | 119.9153 | 123.3092 | 127.137 | 131.0247 | 134.5751 | 136.7231 | 138.1274 |
| 95.5 | 117.0587 | 118.3585 | 120.3749 | 123.7845 | 127.632 | 131.5419 | 135.1144 | 137.2767 | 138.6906 |
| 96.5 | 117.5 | 118.8053 | 120.8305 | 124.2562 | 128.1237 | 132.0559 | 135.6504 | 137.8267 | 139.2502 |
| 97.5 | 117.9366 | 119.2475 | 121.2819 | 124.7242 | 128.6119 | 132.5664 | 136.1829 | 138.3731 | 139.2302 |
| 98.5 | 118.3683 | 119.6851 | 121.729 | 125.1882 | 129.0966 | 133.0736 | 136.7118 | 138.9159 | 140.358 |
| 99.5 | 118.7949 | 120.1179 | | | | | | | |
| | | | 122.1716 | 125.6484 | 129.5777 | 133.5771 | 137.2371 | 139.4548 | 140.9062 |
| 100.5 | 119.2165 | 120.5459 | 122.6099 | 126.1045 | 130.055 | 134.0771 | 137.7587 | 139.9899 | 141.4503 |
| 101.5 | 119.633 | 120.969 | 123.0435 | 126.5565 | 130.5286 | 134.5734 | 138.2765 | 140.5211 | 141.9904 |
| 102.5 | 120.0442 | | 123.4726 | 127.0044 | 130.9983 | 135.066 | 138.7905 | 141.0484 | 142.5263 |
| 103.5 | 120.4502 | 121.8004 | 123.897 | 127.4481 | 131.4641 | 135.5548 | 139.3006 | 141.5716 | 143.0582 |
| 104.5 | 120.851 | 122.2086 | 124.3168 | 127.8876 | 131.926 | 136.0397 | 139.8069 | 142.0908 | 143.586 |
| 105.5 | 121.2467 | 122.6119 | 124.7319 | 128.3228 | 132.384 | 136.5209 | 140.3093 | 142.6061 | 144.1096 |
| 106.5 | 121.6372 | 123.0103 | 125.1425 | 128.7539 | 132.8381 | 136.9982 | 140.8077 | 143.1173 | 144.6291 |
| 107.5 | 122.0228 | 123.4039 | 125.5485 | 129.1807 | 133.2882 | 137.4717 | 141.3023 | 143.6245 | 145.1445 |
| 108.5 | 122.4034 | 123.7928 | 125.9501 | 129.6035 | 133.7345 | 137.9414 | 141.793 | 144.1278 | 145.656 |
| 109.5 | 122.7793 | 124.1771 | 126.3473 | 130.0222 | 134.1769 | 138.4073 | 142.28 | 144.6272 | 146.1634 |
| 110.5 | 123.1506 | 124.5569 | 126.7402 | 130.4369 | 134.6155 | 138.8696 | 142.7632 | 145.1228 | 146.6671 |
| 111.5 | 123.5175 | 124.9325 | 127.1291 | 130.8477 | 135.0504 | 139.3282 | 143.2428 | 145.6148 | 147.167 |
| 112.5 | 123.8803 | 125.304 | 127.514 | 131.2548 | 135.4818 | 139.7833 | 143.7188 | 146.1032 | 147.6633 |
| 113.5 | 124.2391 | | 127.8953 | 131.6584 | 135.9097 | 140.235 | 144.1915 | 146.5882 | 148.1562 |
| 114.5 | 124.5943 | 126.0358 | 128.273 | 132.0585 | 136.3343 | 140.6835 | 144.661 | 147.0699 | 148.6459 |
| 115.5 | 124.9462 | 126.3966 | 128.6474 | 132.4555 | 136.7557 | 141.1289 | 145.1273 | 147.5486 | 149.1325 |
| 220.0 | 125.295 | 126.7544 | 129.0189 | 132.8495 | 137.1742 | 141.5713 | 145.5909 | 148.0245 | 149.6163 |
| 117.5 | 125.6413 | 127.1096 | 129.3876 | 133.2407 | 137.5899 | 142.0111 | 146.0518 | 148.4979 | 150.0977 |
| 118.5 | 125.9852 | 127.4624 | 129.754 | 133.6295 | 138.0032 | 142.4484 | 146.5103 | 148.9689 | 150.5767 |
| 119.5 | 126.3272 | 127.8132 | 130.1183 | 134.0161 | 138.4143 | 142.8835 | 146.9668 | 149.438 | 151.0539 |
| | 126.6678 | 128.1625 | 130.4809 | 134.4008 | 138.8234 | 143.3168 | 147.4214 | 149.9053 | 151.5294 |
| 121.5 | 127.0073 | 128.5106 | 130.8422 | 134.7841 | 139.231 | 143.7484 | 147.8747 | 150.3714 | 152.0038 |

## Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 122.5 | 127.3462 | 128.8579 | 131.2026 | 135.1663 | 139.6373 | 144.1789 | 148.3268 | 150.8365 | 152.4773 |
| 123.5 | 127.6851 | 129.2051 | 131.5625 | 135.5477 | 140.0427 | 144.6085 | 148.7782 | 151.301 | 152.9504 |
| 124.5 | 128.0243 | 129.5524 | 131.9224 | 135.9288 | 140.4477 | 145.0377 | 149.2294 | 151.7655 | 153.4235 |
| 125.5 | 128.3643 | 129.9004 | 132.2828 | 136.3101 | 140.8527 | 145.4669 | 149.6808 | 152.2303 | 153.8972 |
| 126.5 | 128.7058 | 130.2496 | 132.6441 | 136.692 | 141.2582 | 145.8965 | 150.1329 | 152.696 | 154.3718 |
| 127.5 | 129.0491 | 130.6005 | 133.0068 | 137.075 | 141.6646 | 146.3272 | 150.5861 | 153.1631 | 154.848 |
| 128.5 | 129.3949 | 130.9536 | 133.3714 | 137.4597 | 142.0725 | 146.7593 | 151.041 | 153.6321 | 155.3263 |
| 129.5 | 129.7436 | 131.3094 | 133.7386 | 137.8466 | 142.4824 | 147.1936 | 151.4982 | 154.1035 | 155.8072 |
| 130.5 | 130.0958 | 131.6686 | 134.1089 | 138.2362 | 142.8949 | 147.6305 | 151.9583 | 154.578 | 156.2913 |
| 131.5 | 130.452 | 132.0316 | 134.4828 | 138.6292 | 143.3107 | 148.0707 | 152.4218 | 155.0562 | 156.7792 |
| 132.5 | 130.8127 | 132.399 | 134.8608 | 139.0262 | 143.7304 | 148.5147 | 152.8894 | 155.5386 | 157.2715 |
| 133.5 | 131.1785 | 132.7714 | 135.2437 | 139.4278 | 144.1545 | 148.9633 | 153.3617 | 156.0258 | 157.7688 |
| 134.5 | 131.5498 | 133.1491 | 135.6318 | 139.8346 | 144.5838 | 149.4172 | 153.8394 | 156.5186 | 158.2717 |
| 135.5 | 131.9272 | 133.5329 | 136.026 | 140.2472 | 145.019 | 149.8769 | 154.323 | 157.0174 | 158.7806 |
| 136.5 | 132.311 | 133.9232 | 136.4266 | 140.6664 | 145.4607 | 150.3433 | 154.8133 | 157.5229 | 159.2964 |
| 137.5 | 132.7018 | 134.3205 | 136.8343 | 141.0928 | 145.9097 | 150.8169 | 155.3109 | 158.0356 | 159.8193 |
| 138.5 | 133.1 | 134.7252 | 137.2496 | 141.5269 | 146.3665 | 151.2984 | 155.8164 | 158.5562 | 160.35 |
| 139.5 | 133.5059 | 135.1378 | 137.673 | 141.9694 | 146.832 | 151.7885 | 156.3303 | 159.0851 | 160.889 |
| 140.5 | 133.9199 | 135.5588 | 138.105 | 142.4209 | 147.3066 | 152.2878 | 156.8532 | 159.6228 | 161.4365 |
| 141.5 | 134.3423 | 135.9885 | 138.5461 | 142.882 | 147.7911 | 152.7969 | 157.3857 | 160.1697 | 161.993 |
| 142.5 | 134.7733 | 136.4271 | 138.9968 | 143.3532 | 148.2859 | 153.3164 | 157.928 | 160.7262 | 162.5588 |
| 143.5 | 135.2132 | 136.8751 | 139.4573 | 143.835 | 148.7917 | 153.8466 | 158.4807 | 161.2924 | 163.1339 |
| 144.5 | 135.6621 | 137.3326 | 139.928 | 144.3277 | 149.3088 | 154.3881 | 159.0439 | 161.8686 | 163.7185 |
| 145.5 | 136.1202 | 137.7998 | 140.4091 | 144.8317 | 149.8376 | 154.941 | 159.6179 | 162.4549 | 164.3126 |
| 146.5 | 136.5875 | 138.2769 | 140.9009 | 145.3473 | 150.3784 | 155.5056 | 160.2026 | 163.0511 | 164.916 |
| 147.5 | 137.064 | 138.7638 | 141.4034 | 145.8746 | 150.9313 | 156.0819 | 160.7981 | 163.6571 | 165.5285 |
| 148.5 | 137.5496 | 139.2605 | 141.9167 | 146.4137 | 151.4964 | 156.6699 | 161.4041 | 164.2726 | 166.1497 |
| 149.5 | 138.0442 | 139.767 | 142.4407 | 146.9645 | 152.0735 | 157.2694 | 162.0203 | 164.8972 | 166.7791 |
| 150.5 | 138.5477 | 140.2831 | 142.9752 | 147.5269 | 152.6624 | 157.88 | 162.6462 | 165.5302 | 167.416 |
| 151.5 | 139.0597 | 140.8085 | 143.52 | 148.1005 | 153.2627 | 158.5012 | 163.2811 | 166.1711 | 168.0596 |
| 152.5 | 139.5799 | 141.3429 | 144.0746 | 148.6849 | 153.8738 | 159.1324 | 163.9243 | 166.8187 | 168.7091 |
| 153.5 | 140.108 | 141.8859 | 144.6388 | 149.2795 | 154.4951 | 159.7725 | 164.5748 | 167.4723 | 169.3634 |
| 154.5 | 140.6435 | 142.4369 | 145.2117 | 149.8836 | 155.1255 | 160.4207 | 165.2314 | 168.1305 | 170.0213 |

## Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 155.5 | 141.1858 | 142.9955 | 145.7928 | 150.4962 | 155.7642 | 161.0758 | 165.893 | 168.7923 | 170.6817 |
| 156.5 | 141.7345 | 143.5608 | 146.3813 | 151.1165 | 156.4099 | 161.7364 | 166.5581 | 169.4561 | 171.343 |
| 157.5 | 142.2889 | 144.1322 | 146.9763 | 151.7433 | 157.0612 | 162.401 | 167.2253 | 170.1205 | 172.004 |
| 158.5 | 142.8482 | 144.7089 | 147.5767 | 152.3754 | 157.7168 | 163.0682 | 167.8929 | 170.784 | 172.663 |
| 159.5 | 143.4118 | 145.29 | 148.1815 | 153.0113 | 158.3751 | 163.7363 | 168.5594 | 171.445 | 173.3186 |
| 160.5 | 143.9788 | 145.8746 | 148.7896 | 153.6498 | 159.0344 | 164.4035 | 169.2231 | 172.1018 | 173.9691 |
| 161.5 | 144.5483 | 146.4615 | 149.3998 | 154.2892 | 159.6931 | 165.0681 | 169.8822 | 172.7528 | 174.6131 |
| 162.5 | 145.1196 | 147.0498 | 150.0107 | 154.928 | 160.3493 | 165.7283 | 170.535 | 173.3965 | 175.249 |
| 163.5 | 145.6915 | 147.6385 | 150.621 | 155.5647 | 161.0015 | 166.3823 | 171.1798 | 174.0312 | 175.8753 |
| 164.5 | 146.2633 | 148.2262 | 151.2295 | 156.1977 | 161.6478 | 167.0284 | 171.8151 | 174.6554 | 176.4906 |
| 165.5 | 146.8339 | 148.812 | 151.8348 | 156.8253 | 162.2865 | 167.665 | 172.4393 | 175.2677 | 177.0935 |
| 166.5 | 147.4023 | 149.3947 | 152.4355 | 157.4462 | 162.9161 | 168.2905 | 173.0509 | 175.8668 | 177.6829 |
| 167.5 | 147.9674 | 149.9731 | 153.0304 | 158.0587 | 163.535 | 168.9033 | 173.6486 | 176.4515 | 178.2575 |
| 168.5 | 148.5284 | 150.5461 | 153.6181 | 158.6615 | 164.1418 | 169.5022 | 174.2313 | 177.0206 | 178.8165 |
| 169.5 | 149.0842 | 151.1127 | 154.1975 | 159.2532 | 164.7352 | 170.0859 | 174.7978 | 177.5733 | 179.3589 |
| 170.5 | 149.6338 | 151.6717 | 154.7674 | 159.8327 | 165.314 | 170.6535 | 175.3473 | 178.1088 | 179.884 |
| 171.5 | 150.1763 | 152.2221 | 155.3268 | 160.3988 | 165.8771 | 171.2039 | 175.879 | 178.6264 | 180.3913 |
| 172.5 | 150.7107 | 152.763 | 155.8746 | 160.9506 | 166.4236 | 171.7364 | 176.3923 | 179.1256 | 180.8804 |
| 173.5 | 151.2363 | 153.2935 | 156.4099 | 161.4872 | 166.9528 | 172.2504 | 176.8868 | 179.6061 | 181.3509 |
| 174.5 | 151.7521 | 153.8127 | 156.9319 | 162.0078 | 167.4641 | 172.7455 | 177.3622 | 180.0676 | 181.8027 |
| 175.5 | 152.2575 | 154.32 | 157.4399 | 162.5118 | 167.9571 | 173.2213 | 177.8183 | 180.5102 | 182.2358 |
| 176.5 | 152.7517 | 154.8147 | 157.9334 | 162.9988 | 168.4313 | 173.6778 | 178.2551 | 180.9338 | 182.6503 |
| 177.5 | 153.2342 | 155.2961 | 158.4118 | 163.4685 | 168.8867 | 174.1148 | 178.6727 | 181.3385 | 183.0463 |
| 178.5 | 153.7043 | 155.7638 | 158.8747 | 163.9205 | 169.3231 | 174.5324 | 179.0712 | 181.7247 | 183.4242 |
| 179.5 | 154.1615 | 156.2174 | 159.3218 | 164.3547 | 169.7405 | 174.9309 | 179.451 | 182.0927 | 183.7842 |
| 180.5 | 154.6056 | 156.6566 | 159.7529 | 164.7713 | 170.1393 | 175.3105 | 179.8124 | 182.4429 | 184.127 |
| 181.5 | 155.036 | 157.0811 | 160.168 | 165.1701 | 170.5195 | 175.6716 | 180.1559 | 182.7757 | 184.4528 |
| 182.5 | 155.4526 | 157.4907 | 160.5669 | 165.5514 | 170.8815 | 176.0146 | 180.482 | 183.0918 | 184.7624 |
| 183.5 | 155.8552 | 157.8853 | 160.9498 | 165.9154 | 171.2257 | 176.34 | 180.7912 | 183.3916 | 185.0562 |
| 184.5 | 156.2436 | 158.265 | 161.3167 | 166.2625 | 171.5525 | 176.6483 | 181.0841 | 183.6757 | 185.3349 |
| 185.5 | 156.6178 | 158.6298 | 161.6679 | 166.5929 | 171.8626 | 176.9402 | 181.3614 | 183.9449 | 185.599 |
| 186.5 | 156.9777 | 158.9798 | 162.0035 | 166.9072 | 172.1563 | 177.2163 | 181.6236 | 184.1997 | 185.8493 |
| 187.5 | 157.3235 | 159.315 | 162.3239 | 167.2057 | 172.4343 | 177.4771 | 181.8715 | 184.4408 | 186.0863 |

# Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 188.5 | 157.6551 | 159.6359 | 162.6294 | 167.489 | 172.6972 | 177.7234 | 182.1056 | 184.6687 | 186.3107 |
| 189.5 | 157.9729 | 159.9425 | 162.9204 | 167.7576 | 172.9456 | 177.9558 | 182.3267 | 184.8843 | 186.5231 |
| 190.5 | 158.277 | 160.2352 | 163.1973 | 168.012 | 173.1801 | 178.175 | 182.5353 | 185.0879 | 186.724 |
| 191.5 | 158.5676 | 160.5143 | 163.4605 | 168.2528 | 173.4014 | 178.3815 | 182.7322 | 185.2804 | 186.9142 |
| 192.5 | 158.845 | 160.7802 | 163.7104 | 168.4805 | 173.6101 | 178.5762 | 182.9179 | 185.4623 | 187.0941 |
| 193.5 | 159.1095 | 161.0332 | 163.9476 | 168.6958 | 173.8067 | 178.7595 | 183.0931 | 185.6341 | 187.2643 |
| 194.5 | 159.3614 | 161.2738 | 164.1725 | 168.8991 | 173.992 | 178.9321 | 183.2583 | 185.7965 | 187.4254 |
| 195.5 | 159.6011 | 161.5023 | 164.3856 | 169.0911 | 174.1665 | 179.0946 | 183.414 | 185.9498 | 187.5779 |
| 196.5 | 159.829 | 161.7191 | 164.5873 | 169.2722 | 174.3308 | 179.2476 | 183.5609 | 186.0948 | 187.7222 |
| 197.5 | 160.0455 | 161.9247 | 164.7782 | 169.4431 | 174.4854 | 179.3915 | 183.6995 | 186.2318 | 187.8588 |
| 198.5 | 160.2508 | 162.1196 | 164.9587 | 169.6041 | 174.631 | 179.5271 | 183.8302 | 186.3613 | 187.9881 |
| 199.5 | 160.4456 | 162.3041 | 165.1292 | 169.756 | 174.768 | 179.6547 | 183.9535 | 186.4837 | 188.1106 |
| 200.5 | 160.63 | 162.4786 | 165.2903 | 169.8991 | 174.8969 | 179.7748 | 184.0699 | 186.5995 | 188.2267 |
| 201.5 | 160.8046 | 162.6437 | 165.4424 | 170.0339 | 175.0182 | 179.888 | 184.1797 | 186.7091 | 188.3368 |
| 202.5 | 160.9697 | 162.7997 | 165.586 | 170.1608 | 175.1323 | 179.9946 | 184.2835 | 186.8128 | 188.4411 |
| 203.5 | 161.1258 | 162.947 | 165.7214 | 170.2804 | 175.2398 | 180.095 | 184.3815 | 186.911 | 188.54 |
| 204.5 | 161.2733 | 163.086 | 165.8491 | 170.3931 | 175.341 | 180.1896 | 184.4741 | 187.004 | 188.6338 |
| 205.5 | 161.4125 | 163.2172 | 165.9694 | 170.4991 | 175.4362 | 180.2789 | 184.5617 | 187.0922 | 188.7229 |
| 206.5 | 161.5438 | 163.3409 | 166.0828 | 170.599 | 175.5259 | 180.3631 | 184.6446 | 187.1757 | 188.8075 |
| 207.5 | 161.6676 | 163.4575 | 166.1897 | 170.693 | 175.6104 | 180.4426 | 184.723 | 187.255 | 188.8878 |
| 208.5 | 161.7843 | 163.5673 | 166.2903 | 170.7816 | 175.6901 | 180.5176 | 184.7972 | 187.3302 | 188.9642 |
| 209.5 | 161.8942 | 163.6708 | 166.3851 | 170.865 | 175.7652 | 180.5885 | 184.8676 | 187.4016 | 189.0368 |
| 210.5 | 161.9977 | 163.7682 | 166.4743 | 170.9436 | 175.836 | 180.6555 | 184.9343 | 187.4694 | 189.1058 |
| 211.5 | 162.0951 | 163.8598 | 166.5583 | 171.0176 | 175.9028 | 180.7189 | 184.9975 | 187.5338 | 189.1715 |
| 212.5 | 162.1866 | 163.9461 | 166.6373 | 171.0873 | 175.9658 | 180.7789 | 185.0576 | 187.5951 | 189.234 |
| 213.5 | 162.2727 | 164.0272 | 166.7116 | 171.1529 | 176.0254 | 180.8357 | 185.1146 | 187.6534 | 189.2936 |
| 214.5 | 162.3537 | 164.1034 | 166.7816 | 171.2148 | 176.0816 | 180.8895 | 185.1687 | 187.7088 | 189.3503 |
| 215.5 | 162.4297 | 164.1751 | 166.8474 | 171.2732 | 176.1348 | 180.9405 | 185.2202 | 187.7617 | 189.4044 |
| 216.5 | 162.5011 | 164.2424 | 166.9094 | 171.3282 | 176.185 | 180.9889 | 185.2692 | 187.812 | 189.456 |
| 217.5 | 162.5681 | 164.3057 | 166.9676 | 171.3801 | 176.2326 | 181.0348 | 185.3159 | 187.86 | 189.5052 |
| 218.5 | 162.631 | 164.3651 | 167.0224 | 171.429 | 176.2776 | 181.0784 | 185.3603 | 187.9057 | 189.5522 |
| 219.5 | 162.69 | 164.4209 | 167.074 | 171.4752 | 176.3202 | 181.1199 | 185.4026 | 187.9494 | 189.5971 |
| 220.5 | 162.7453 | 164.4733 | 167.1224 | 171.5188 | 176.3606 | 181.1593 | 185.443 | 187.9911 | 189.6399 |

EudraCT number 2016-001767-37 - CONFIDENTIAL -

# Males, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 221.5 | 162.7972 | 164.5224 | 167.168 | 171.5599 | 176.3989 | 181.1968 | 185.4815 | 188.0309 | 189.6809 |
| 222.5 | 162.8458 | 164.5686 | 167.2109 | 171.5988 | 176.4352 | 181.2325 | 185.5182 | 188.069 | 189.7201 |
| 223.5 | 162.8914 | 164.6119 | 167.2513 | 171.6355 | 176.4697 | 181.2666 | 185.5534 | 188.1054 | 189.7575 |
| 224.5 | 162.9341 | 164.6526 | 167.2892 | 171.6701 | 176.5024 | 181.299 | 185.5869 | 188.1402 | 189.7934 |
| 225.5 | 162.9741 | 164.6907 | 167.325 | 171.7029 | 176.5335 | 181.33 | 185.619 | 188.1736 | 189.8277 |
| 226.5 | 163.0115 | 164.7265 | 167.3585 | 171.7339 | 176.563 | 181.3595 | 185.6497 | 188.2055 | 189.8606 |
| 227.5 | 163.0465 | 164.76 | 167.3902 | 171.7632 | 176.5911 | 181.3877 | 185.6791 | 188.236 | 189.8922 |
| 228.5 | 163.0793 | 164.7915 | 167.4199 | 171.791 | 176.6179 | 181.4147 | 185.7073 | 188.2653 | 189.9224 |
| 229.5 | 163.11 | 164.821 | 167.4479 | 171.8172 | 176.6433 | 181.4405 | 185.7343 | 188.2934 | 189.9513 |
| 230.5 | 163.1387 | 164.8487 | 167.4742 | 171.8421 | 176.6676 | 181.4651 | 185.7601 | 188.3204 | 189.9791 |
| 231.5 | 163.1656 | 164.8746 | 167.499 | 171.8657 | 176.6907 | 181.4887 | 185.7849 | 188.3462 | 190.0058 |
| 232.5 | 163.1907 | 164.8989 | 167.5224 | 171.888 | 176.7127 | 181.5113 | 185.8087 | 188.3711 | 190.0314 |
| 233.5 | 163.2142 | 164.9217 | 167.5444 | 171.9091 | 176.7337 | 181.533 | 185.8316 | 188.3949 | 190.056 |
| 234.5 | 163.2361 | 164.9431 | 167.5651 | 171.9292 | 176.7538 | 181.5538 | 185.8535 | 188.4178 | 190.0797 |
| 235.5 | 163.2566 | 164.9631 | 167.5846 | 171.9483 | 176.773 | 181.5737 | 185.8746 | 188.4399 | 190.1024 |
| 236.5 | 163.2757 | 164.9819 | 167.6029 | 171.9663 | 176.7913 | 181.5928 | 185.8949 | 188.461 | 190.1242 |
| 237.5 | 163.2936 | 164.9995 | 167.6203 | 171.9835 | 176.8088 | 181.6111 | 185.9144 | 188.4814 | 190.1452 |
| 238.5 | 163.3103 | 165.016 | 167.6366 | 171.9998 | 176.8255 | 181.6287 | 185.9331 | 188.501 | 190.1654 |
| 239.5 | 163.3259 | 165.0315 | 167.6519 | 172.0153 | 176.8415 | 181.6456 | 185.9512 | 188.5198 | 190.1849 |
| 240 | 163.3333 | 165.0389 | 167.6593 | 172.0227 | 176.8492 | 181.6538 | 185.9599 | 188.529 | 190.1943 |

# 12.12 Centers for Disease Control and Prevention Data Table of Stature for Age Chart for Females

## Females, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 24 | 78.43754 | 79.25982 | 80.52476 | 82.63524 | 84.97556 | 87.31121 | 89.40951 | 90.66355 | 91.47729 |
| 24.5 | 78.82133 | 79.64777 | 80.91946 | 83.04213 | 85.39732 | 87.74918 | 89.86316 | 91.12707 | 91.94741 |
| 25.5 | 79.60198 | 80.44226 | 81.73541 | 83.8943 | 86.29026 | 88.68344 | 90.83505 | 92.12168 | 92.95685 |
| 26.5 | 80.37555 | 81.22666 | 82.53699 | 84.72592 | 87.15714 | 89.58751 | 91.77421 | 93.08254 | 93.93209 |
| 27.5 | 81.1357 | 81.9954 | 83.31968 | 85.53389 | 87.99602 | 90.46018 | 92.67969 | 94.00873 | 94.87215 |
| 28.5 | 81.87746 | 82.74411 | 84.07998 | 86.31589 | 88.80551 | 91.30065 | 93.55097 | 94.89974 | 95.77649 |
| 29.5 | 82.59712 | 83.46957 | 84.81532 | 87.07028 | 89.58477 | 92.10859 | 94.38793 | 95.75551 | 96.64505 |
| 30.5 | 83.29206 | 84.16953 | 85.52398 | 87.79609 | 90.33342 | 92.88403 | 95.19083 | 96.57635 | 97.47814 |
| 31.5 | 83.96065 | 84.84264 | 86.205 | 88.49291 | 91.05154 | 93.62741 | 95.9603 | 97.36295 | 98.27646 |
| 32.5 | 84.6021 | 85.4883 | 86.85807 | 89.16084 | 91.73964 | 94.33951 | 96.69729 | 98.11632 | 99.04107 |
| 33.5 | 85.2163 | 86.10656 | 87.48344 | 89.80045 | 92.39854 | 95.0214 | 97.40303 | 98.83778 | 99.77332 |
| 34.5 | 85.80379 | 86.69803 | 88.08186 | 90.4127 | 93.02945 | 95.67446 | 98.07904 | 99.52891 | 100.4748 |
| 35.5 | 86.36557 | 87.26379 | 88.6545 | 90.99891 | 93.63382 | 96.30029 | 98.72705 | 100.1915 | 101.1474 |
| 36.5 | 86.90307 | 87.80528 | 89.20285 | 91.56066 | 94.21336 | 96.90071 | 99.34899 | 100.8276 | 101.7931 |
| 37.5 | 87.43482 | 88.34236 | 89.74875 | 92.12298 | 94.79643 | 97.50724 | 99.97896 | 101.4726 | 102.4485 |
| 38.5 | 87.95945 | 88.87256 | 90.28811 | 92.67925 | 95.37392 | 98.10855 | 100.604 | 102.1129 | 103.0991 |
| 39.5 | 88.4785 | 89.39733 | 90.82228 | 93.2307 | 95.94693 | 98.70568 | 101.2251 | 102.7494 | 103.746 |
| 40.5 | 88.9933 | 89.91797 | 91.35246 | 93.7784 | 96.51645 | 99.29957 | 101.8432 | 103.383 | 104.3901 |
| 41.5 | 89.50502 | 90.43559 | 91.87972 | 94.32334 | 97.08337 | 99.89104 | 102.459 | 104.0144 | 105.032 |
| 42.5 | 90.01466 | 90.95115 | 92.40497 | 94.86634 | 97.64848 | 100.4808 | 103.0732 | 104.6444 | 105.6727 |
| 43.5 | 90.52307 | 91.46549 | 92.92901 | 95.40817 | 98.21247 | 101.0696 | 103.6866 | 105.2736 | 106.3126 |
| 44.5 | 91.031 | 91.97932 | 93.45252 | 95.94946 | 98.77593 | 101.6579 | 104.2996 | 105.9025 | 106.9523 |
| 45.5 | 91.53905 | 92.49325 | 93.97609 | 96.49076 | 99.3394 | 102.2462 | 104.9128 | 106.5316 | 107.5922 |
| 46.5 | 92.04774 | 93.00778 | 94.50021 | 97.03254 | 99.90331 | 102.835 | 105.5264 | 107.1613 | 108.2328 |
| 47.5 | 92.55748 | 93.52333 | 95.02528 | 97.57519 | 100.4681 | 103.4247 | 106.141 | 107.7919 | 108.8744 |
| 48.5 | 93.06862 | 94.04022 | 95.55164 | 98.11905 | 101.0339 | 104.0154 | 106.7567 | 108.4238 | 109.5172 |
| 49.5 | 93.58141 | 94.55872 | 96.07954 | 98.66436 | 101.6012 | 104.6075 | 107.3737 | 109.057 | 110.1614 |
| 50.5 | 94.09605 | 95.07903 | 96.60918 | 99.21132 | 102.17 | 105.2012 | 107.9924 | 109.6918 | 110.8073 |
| 51.5 | 94.61267 | 95.60128 | 97.14072 | 99.76009 | 102.7406 | 105.7965 | 108.6127 | 110.3283 | 111.4548 |
| 52.5 | 95.13134 | 96.12555 | 97.67423 | 100.3108 | 103.313 | 106.3936 | 109.2347 | 110.9665 | 112.1041 |
| 53.5 | 95.65211 | 96.65189 | 98.20976 | 100.8634 | 103.8873 | 106.9925 | 109.8585 | 111.6066 | 112.7552 |
| 54.5 | 96.17495 | 97.18029 | 98.74731 | 101.418 | 104.4635 | 107.5933 | 110.4841 | 112.2483 | 113.4079 |
| 55.5 | 96.69982 | 97.71069 | 99.28686 | 101.9745 | 105.0415 | 108.1958 | 111.1114 | 112.8917 | 114.0624 |

# Females, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 56.5 | 97.22663 | 98.24303 | 99.82832 | 102.5329 | 105.6213 | 108.8001 | 111.7404 | 113.5368 | 114.7184 |
| 57.5 | 97.75525 | 98.77719 | 100.3716 | 103.093 | 106.2029 | 109.406 | 112.3709 | 114.1833 | 115.3759 |
| 58.5 | 98.28555 | 99.31303 | 100.9165 | 103.6549 | 106.7861 | 110.0134 | 113.0028 | 114.8312 | 116.0347 |
| 59.5 | 98.81735 | 99.85039 | 101.463 | 104.2182 | 107.3707 | 110.6222 | 113.6359 | 115.4802 | 116.6945 |
| 60.5 | 99.35047 | 100.3891 | 102.0109 | 104.7829 | 107.9566 | 111.2321 | 114.2701 | 116.1301 | 117.3552 |
| 61.5 | 99.8847 | 100.9289 | 102.5599 | 105.3488 | 108.5436 | 111.8431 | 114.9052 | 116.7808 | 118.0166 |
| 62.5 | 100.4198 | 101.4696 | 103.1098 | 105.9156 | 109.1316 | 112.4548 | 115.5408 | 117.432 | 118.6783 |
| 63.5 | 100.9555 | 102.011 | 103.6604 | 106.4831 | 109.7202 | 113.0671 | 116.1768 | 118.0834 | 119.3402 |
| 64.5 | 101.4916 | 102.5529 | 104.2115 | 107.0512 | 110.3092 | 113.6797 | 116.813 | 118.7348 | 120.0019 |
| 65.5 | 102.0279 | 103.0948 | 104.7628 | 107.6194 | 110.8984 | 114.2923 | 117.449 | 119.3858 | 120.6632 |
| 66.5 | 102.564 | 103.6367 | 105.3141 | 108.1877 | 111.4876 | 114.9048 | 118.0845 | 120.0362 | 121.3238 |
| 67.5 | 103.0996 | 104.1782 | 105.865 | 108.7556 | 112.0764 | 115.5167 | 118.7193 | 120.6857 | 121.9832 |
| 68.5 | 103.6346 | 104.7191 | 106.4154 | 109.323 | 112.6646 | 116.1278 | 119.3531 | 121.334 | 122.6413 |
| 69.5 | 104.1685 | 105.259 | 106.9648 | 109.8895 | 113.2519 | 116.7379 | 119.9855 | 121.9807 | 123.2977 |
| 70.5 | 104.7012 | 105.7976 | 107.5131 | 110.4549 | 113.838 | 117.3466 | 120.6163 | 122.6256 | 123.9521 |
| 71.5 | 105.2323 | 106.3348 | 108.0599 | 111.0189 | 114.4226 | 117.9537 | 121.2452 | 123.2684 | 124.6042 |
| 72.5 | 105.7615 | 106.8701 | 108.605 | 111.5812 | 115.0055 | 118.5588 | 121.8718 | 123.9086 | 125.2536 |
| 73.5 | 106.2886 | 107.4033 | 109.148 | 112.1415 | 115.5863 | 119.1616 | 122.4959 | 124.5461 | 125.9 |
| 74.5 | 106.8132 | 107.9342 | 109.6888 | 112.6996 | 116.1648 | 119.7619 | 123.1171 | 125.1804 | 126.5432 |
| 75.5 | 107.3351 | 108.4624 | 110.227 | 113.255 | 116.7406 | 120.3594 | 123.7352 | 125.8114 | 127.1827 |
| 76.5 | 107.8541 | 108.9877 | 110.7623 | 113.8077 | 117.3136 | 120.9537 | 124.3499 | 126.4387 | 127.8184 |
| 77.5 | 108.3698 | 109.5099 | 111.2944 | 114.3572 | 117.8833 | 121.5447 | 124.9608 | 127.062 | 128.45 |
| 78.5 | 108.882 | 110.0285 | 111.8232 | 114.9034 | 118.4496 | 122.132 | 125.5678 | 127.6811 | 129.0771 |
| 79.5 | 109.3905 | 110.5435 | 112.3483 | 115.446 | 119.0123 | 122.7154 | 126.1705 | 128.2957 | 129.6996 |
| 80.5 | 109.8949 | 111.0545 | 112.8696 | 115.9847 | 119.571 | 123.2946 | 126.7688 | 128.9056 | 130.3171 |
| 81.5 | 110.3952 | 111.5613 | 113.3867 | 116.5193 | 120.1254 | 123.8695 | 127.3623 | 129.5105 | 130.9295 |
| 82.5 | 110.8909 | 112.0638 | 113.8995 | 117.0496 | 120.6755 | 124.4397 | 127.951 | 130.1103 | 131.5365 |
| 83.5 | 111.3821 | 112.5616 | 114.4077 | 117.5754 | 121.221 | 125.0051 | 128.5345 | 130.7047 | 132.138 |
| 84.5 | 111.8684 | 113.0546 | 114.9112 | 118.0964 | 121.7617 | 125.5655 | 129.1127 | 131.2936 | 132.7338 |
| 85.5 | 112.3496 | 113.5427 | 115.4097 | 118.6125 | 122.2974 | 126.1207 | 129.6855 | 131.8768 | 133.3238 |
| 86.5 | 112.8257 | 114.0256 | 115.9031 | 119.1235 | 122.8279 | 126.6706 | 130.2526 | 132.4542 | 133.9077 |
| 87.5 | 113.2963 | 114.5031 | 116.3913 | 119.6293 | 123.3531 | 127.215 | 130.814 | 133.0256 | 134.4857 |
| 88.5 | 113.7615 | 114.9752 | 116.874 | 120.1297 | 123.8728 | 127.7539 | 131.3696 | 133.5911 | 135.0574 |

## Females, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 89.5 | 114.2211 | 115.4418 | 117.3512 | 120.6246 | 124.387 | 128.287 | 131.9194 | 134.1505 | 135.623 |
| 90.5 | 114.6749 | 115.9026 | 117.8228 | 121.1138 | 124.8956 | 128.8144 | 132.4631 | 134.7038 | 136.1824 |
| 91.5 | 115.123 | 116.3577 | 118.2886 | 121.5974 | 125.3985 | 129.3359 | 133.0009 | 135.251 | 136.7356 |
| 92.5 | 115.5651 | 116.8069 | 118.7486 | 122.0753 | 125.8956 | 129.8516 | 133.5328 | 135.7922 | 137.2826 |
| 93.5 | 116.0012 | 117.2502 | 119.2028 | 122.5473 | 126.3869 | 130.3615 | 134.0587 | 136.3273 | 137.8236 |
| 94.5 | 116.4314 | 117.6875 | 119.6511 | 123.0135 | 126.8724 | 130.8656 | 134.5787 | 136.8565 | 138.3585 |
| 95.5 | 116.8555 | 118.1189 | 120.0935 | 123.4739 | 127.3522 | 131.364 | 135.093 | 137.3798 | 138.8876 |
| 96.5 | 117.2737 | 118.5443 | 120.53 | 123.9285 | 127.8263 | 131.8567 | 135.6015 | 137.8975 | 139.411 |
| 97.5 | 117.6858 | 118.9638 | 120.9607 | 124.3774 | 128.2947 | 132.3438 | 136.1046 | 138.4097 | 139.9289 |
| 98.5 | 118.092 | 119.3774 | 121.3855 | 124.8207 | 128.7576 | 132.8255 | 136.6024 | 138.9166 | 140.4415 |
| 99.5 | 118.4924 | 119.7852 | 121.8047 | 125.2584 | 129.2152 | 133.302 | 137.095 | 139.4184 | 140.9492 |
| 100.5 | 118.8869 | 120.1873 | 122.2182 | 125.6906 | 129.6675 | 133.7734 | 137.5828 | 139.9155 | 141.4521 |
| 101.5 | 119.2757 | 120.5838 | 122.6263 | 126.1177 | 130.1148 | 134.2401 | 138.066 | 140.4082 | 141.9507 |
| 102.5 | 119.659 | 120.9748 | 123.0291 | 126.5396 | 130.5574 | 134.7023 | 138.545 | 140.8968 | 142.4454 |
| 103.5 | 120.037 | 121.3606 | 123.4268 | 126.9568 | 130.9954 | 135.1604 | 139.0201 | 141.3817 | 142.9364 |
| 104.5 | 120.4097 | 121.7413 | 123.8196 | 127.3694 | 131.4293 | 135.6146 | 139.4918 | 141.8633 | 143.4244 |
| 105.5 | 120.7775 | 122.1171 | 124.2078 | 127.7777 | 131.8593 | 136.0654 | 139.9604 | 142.3422 | 143.9098 |
| 106.5 | 121.1405 | 122.4884 | 124.5916 | 128.1822 | 132.2859 | 136.5132 | 140.4265 | 142.8188 | 144.393 |
| 107.5 | 121.4991 | 122.8555 | 124.9715 | 128.5831 | 132.7094 | 136.9585 | 140.8906 | 143.2937 | 144.8747 |
| 108.5 | 121.8537 | 123.2186 | 125.3478 | 128.9808 | 133.1304 | 137.4018 | 141.3532 | 143.7674 | 145.3555 |
| 109.5 | 122.2044 | 123.5782 | 125.7208 | 129.3759 | 133.5493 | 137.8437 | 141.8149 | 144.2406 | 145.8359 |
| 110.5 | 122.5518 | 123.9347 | 126.0911 | 129.7689 | 133.9667 | 138.2847 | 142.2764 | 144.7139 | 146.3167 |
| 111.5 | 122.8963 | 124.2885 | 126.4592 | 130.1603 | 134.3832 | 138.7256 | 142.7382 | 145.1879 | 146.7984 |
| 112.5 | 123.2384 | 124.6402 | 126.8255 | 130.5506 | 134.7995 | 139.1669 | 143.2012 | 145.6634 | 147.2818 |
| 113.5 | 123.5785 | 124.9902 | 127.1907 | 130.9406 | 135.2163 | 139.6094 | 143.666 | 146.141 | 147.7676 |
| 114.5 | 123.9173 | 125.3393 | 127.5554 | 131.3309 | 135.6342 | 140.0538 | 144.1333 | 146.6215 | 148.2564 |
| 115.5 | 124.2553 | 125.688 | 127.9203 | 131.7223 | 136.054 | 140.501 | 144.6039 | 147.1056 | 148.7491 |
| 116.5 | 124.5933 | 126.0371 | 128.2861 | 132.1156 | 136.4766 | 140.9516 | 145.0785 | 147.594 | 149.2461 |
| 117.5 | 124.932 | 126.3872 | 128.6537 | 132.5115 | 136.9027 | 141.4065 | 145.5579 | 148.0874 | 149.7484 |
| 118.5 | 125.2721 | 126.7392 | 129.0238 | 132.9109 | 137.3333 | 141.8665 | 146.0429 | 148.5865 | 150.2564 |
| 119.5 | 125.6144 | 127.094 | 129.3973 | 133.3147 | 137.7691 | 142.3324 | 146.5341 | 149.092 | 150.7707 |
| 120.5 | 125.9599 | 127.4524 | 129.7752 | 133.7239 | 138.2112 | 142.8051 | 147.0322 | 149.6044 | 151.292 |
| 121.5 | 126.3095 | 127.8154 | 130.1584 | 134.1394 | 138.6602 | 143.2852 | 147.5379 | 150.1242 | 151.8205 |

## Females, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 122.5 | 126.6641 | 128.184 | 130.5479 | 134.562 | 139.1172 | 143.7735 | 148.0517 | 150.652 | 152.3568 |
| 123.5 | 127.0248 | 128.5591 | 130.9446 | 134.9929 | 139.5829 | 144.2707 | 148.5741 | 151.188 | 152.9011 |
| 124.5 | 127.3926 | 128.9419 | 131.3496 | 135.4328 | 140.0581 | 144.7773 | 149.1054 | 151.7325 | 153.4534 |
| 125.5 | 127.7687 | 129.3334 | 131.7639 | 135.8826 | 140.5435 | 145.2938 | 149.646 | 152.2856 | 154.0139 |
| 126.5 | 128.1541 | 129.7346 | 132.1885 | 136.3433 | 141.0397 | 145.8206 | 150.196 | 152.8473 | 154.5824 |
| 127.5 | 128.5499 | 130.1467 | 132.6243 | 136.8154 | 141.5472 | 146.3579 | 150.7552 | 153.4174 | 155.1586 |
| 128.5 | 128.9573 | 130.5705 | 133.0721 | 137.2997 | 142.0664 | 146.9059 | 151.3236 | 153.9955 | 155.742 |
| 129.5 | 129.3772 | 131.0071 | 133.5329 | 137.7967 | 142.5974 | 147.4643 | 151.9008 | 154.5812 | 156.3321 |
| 130.5 | 129.8106 | 131.4573 | 134.0072 | 138.3067 | 143.1404 | 148.0329 | 152.4861 | 155.1737 | 156.928 |
| 131.5 | 130.2585 | 131.9218 | 134.4955 | 138.83 | 143.695 | 148.6111 | 153.079 | 155.7721 | 157.5288 |
| 132.5 | 130.7217 | 132.4013 | 134.9983 | 139.3664 | 144.2609 | 149.1984 | 153.6783 | 156.3755 | 158.1335 |
| 133.5 | 131.2006 | 132.8962 | 135.5157 | 139.9157 | 144.8376 | 149.7937 | 154.283 | 156.9825 | 158.7407 |
| 134.5 | 131.6958 | 133.4067 | 136.0476 | 140.4775 | 145.424 | 150.3959 | 154.8918 | 157.5918 | 159.3491 |
| 135.5 | 132.2074 | 133.9328 | 136.5937 | 141.051 | 146.0192 | 151.0036 | 155.5032 | 158.202 | 159.9571 |
| 136.5 | 132.7354 | 134.4742 | 137.1534 | 141.6352 | 146.6217 | 151.6153 | 156.1156 | 158.8115 | 160.5633 |
| 137.5 | 133.2795 | 135.0304 | 137.7259 | 142.2288 | 147.23 | 152.2293 | 156.7273 | 159.4185 | 161.166 |
| 138.5 | 133.8388 | 135.6004 | 138.31 | 142.8304 | 147.8424 | 152.8438 | 157.3365 | 160.0213 | 161.7634 |
| 139.5 | 134.4125 | 136.1831 | 138.9043 | 143.4381 | 148.4569 | 153.4568 | 157.9413 | 160.6182 | 162.3541 |
| 140.5 | 134.9993 | 136.7769 | 139.507 | 144.0501 | 149.0714 | 154.0662 | 158.5398 | 161.2075 | 162.9363 |
| 141.5 | 135.5973 | 137.3801 | 140.1161 | 144.6641 | 149.6839 | 154.67 | 159.1302 | 161.7874 | 163.5084 |
| 142.5 | 136.2047 | 137.9905 | 140.7295 | 145.278 | 150.292 | 155.2663 | 159.7107 | 162.3564 | 164.069 |
| 143.5 | 136.8191 | 138.6058 | 141.3448 | 145.8893 | 150.8936 | 155.8529 | 160.2796 | 162.9129 | 164.6167 |
| 144.5 | 137.4381 | 139.2236 | 141.9594 | 146.4958 | 151.4866 | 156.428 | 160.8353 | 163.4555 | 165.1503 |
| 145.5 | 138.0588 | 139.841 | 142.5709 | 147.0949 | 152.0687 | 156.9899 | 161.3764 | 163.983 | 165.6685 |
| 146.5 | 138.6784 | 140.4554 | 143.1767 | 147.6845 | 152.6381 | 157.5369 | 161.9016 | 164.4943 | 166.1706 |
| 147.5 | 139.2941 | 141.064 | 143.7741 | 148.2623 | 153.193 | 158.0677 | 162.4097 | 164.9885 | 166.6555 |
| 148.5 | 139.9028 | 141.6641 | 144.3607 | 148.8263 | 153.7317 | 158.581 | 162.8999 | 165.4648 | 167.1228 |
| 149.5 | 140.5019 | 142.253 | 144.9342 | 149.3747 | 154.2529 | 159.0758 | 163.3715 | 165.9227 | 167.572 |
| 150.5 | 141.0885 | 142.8283 | 145.4925 | 149.9059 | 154.7555 | 159.5513 | 163.8239 | 166.3618 | 168.0027 |
| 151.5 | 141.6602 | 143.3877 | 146.0338 | 150.4184 | 155.2385 | 160.007 | 164.2568 | 166.7819 | 168.4147 |
| 152.5 | 142.2148 | 143.9294 | 146.5564 | 150.9113 | 155.7012 | 160.4425 | 164.6701 | 167.1829 | 168.808 |
| 153.5 | 142.7504 | 144.4516 | 147.059 | 151.3835 | 156.1432 | 160.8576 | 165.0637 | 167.5648 | 169.1827 |
| 154.5 | 143.2654 | 144.953 | 147.5405 | 151.8346 | 156.5643 | 161.2524 | 165.4378 | 167.9278 | 169.5391 |

## Females, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 155.5 | 143.7584 | 145.4325 | 148.0002 | 152.2642 | 156.9644 | 161.627 | 165.7928 | 168.2723 | 169.8773 |
| 156.5 | 144.2287 | 145.8894 | 148.4376 | 152.6721 | 157.3437 | 161.9818 | 166.1289 | 168.5987 | 170.1979 |
| 157.5 | 144.6756 | 146.3232 | 148.8525 | 153.0584 | 157.7025 | 162.3172 | 166.4466 | 168.9074 | 170.5013 |
| 158.5 | 145.0987 | 146.7338 | 149.2449 | 153.4234 | 158.0411 | 162.6338 | 166.7467 | 169.199 | 170.7881 |
| 159.5 | 145.4981 | 147.1213 | 149.615 | 153.7674 | 158.3603 | 162.9321 | 167.0296 | 169.4742 | 171.0587 |
| 160.5 | 145.874 | 147.4859 | 149.9633 | 154.0911 | 158.6606 | 163.2129 | 167.2961 | 169.7335 | 171.314 |
| 161.5 | 146.2269 | 147.8281 | 150.2902 | 154.3951 | 158.9427 | 163.477 | 167.5469 | 169.9777 | 171.5544 |
| 162.5 | 146.5573 | 148.1487 | 150.5966 | 154.6801 | 159.2075 | 163.725 | 167.7826 | 170.2074 | 171.7807 |
| 163.5 | 146.866 | 148.4483 | 150.8831 | 154.947 | 159.4557 | 163.9577 | 168.0042 | 170.4234 | 171.9935 |
| 164.5 | 147.1539 | 148.7279 | 151.1507 | 155.1966 | 159.6882 | 164.1761 | 168.2122 | 170.6263 | 172.1936 |
| 165.5 | 147.4219 | 148.9885 | 151.4003 | 155.4298 | 159.9058 | 164.3808 | 168.4075 | 170.817 | 172.3816 |
| 166.5 | 147.6712 | 149.2309 | 151.6329 | 155.6475 | 160.1094 | 164.5726 | 168.5907 | 170.9959 | 172.5582 |
| 167.5 | 147.9026 | 149.4562 | 151.8494 | 155.8507 | 160.2997 | 164.7523 | 168.7626 | 171.1639 | 172.7239 |
| 168.5 | 148.1173 | 149.6655 | 152.0508 | 156.0401 | 160.4777 | 164.9206 | 168.9239 | 171.3216 | 172.8796 |
| 169.5 | 148.3164 | 149.8598 | 152.2381 | 156.2167 | 160.6441 | 165.0783 | 169.0751 | 171.4696 | 173.0257 |
| 170.5 | 148.5009 | 150.04 | 152.4121 | 156.3813 | 160.7995 | 165.226 | 169.217 | 171.6085 | 173.1628 |
| 171.5 | 148.6717 | 150.2072 | 152.5738 | 156.5348 | 160.9449 | 165.3644 | 169.3501 | 171.7388 | 173.2915 |
| 172.5 | 148.8299 | 150.3621 | 152.7241 | 156.6778 | 161.0808 | 165.4941 | 169.4749 | 171.8611 | 173.4124 |
| 173.5 | 148.9764 | 150.5059 | 152.8638 | 156.8112 | 161.2079 | 165.6157 | 169.5921 | 171.976 | 173.5258 |
| 174.5 | 149.1121 | 150.6392 | 152.9936 | 156.9356 | 161.3268 | 165.7297 | 169.7022 | 172.0839 | 173.6324 |
| 175.5 | 149.2377 | 150.7629 | 153.1143 | 157.0517 | 161.4381 | 165.8366 | 169.8055 | 172.1853 | 173.7326 |
| 176.5 | 149.3542 | 150.8777 | 153.2266 | 157.16 | 161.5423 | 165.9369 | 169.9026 | 172.2806 | 173.8267 |
| 177.5 | 149.4622 | 150.9843 | 153.3312 | 157.2612 | 161.6399 | 166.0312 | 169.9939 | 172.3701 | 173.9152 |
| 178.5 | 149.5623 | 151.0833 | 153.4286 | 157.3558 | 161.7315 | 166.1197 | 170.0798 | 172.4544 | 173.9984 |
| 179.5 | 149.6553 | 151.1754 | 153.5193 | 157.4443 | 161.8174 | 166.2029 | 170.1606 | 172.5337 | 174.0768 |
| 180.5 | 149.7416 | 151.2611 | 153.604 | 157.5271 | 161.898 | 166.2812 | 170.2366 | 172.6084 | 174.1505 |
| 181.5 | 149.8219 | 151.341 | 153.683 | 157.6047 | 161.9738 | 166.3549 | 170.3083 | 172.6787 | 174.22 |
| 182.5 | 149.8967 | 151.4154 | 153.7569 | 157.6775 | 162.045 | 166.4244 | 170.3759 | 172.7451 | 174.2855 |
| 183.5 | 149.9663 | 151.4848 | 153.826 | 157.7458 | 162.112 | 166.4898 | 170.4396 | 172.8076 | 174.3472 |
| 184.5 | 150.0312 | 151.5497 | 153.8907 | 157.8099 | 162.1752 | 166.5516 | 170.4997 | 172.8667 | 174.4055 |
| 185.5 | 150.0918 | 151.6103 | 153.9513 | 157.8702 | 162.2347 | 166.6099 | 170.5566 | 172.9225 | 174.4606 |
| 186.5 | 150.1484 | 151.6671 | 154.0082 | 157.927 | 162.2908 | 166.6649 | 170.6103 | 172.9752 | 174.5125 |
| 187.5 | 150.2014 | 151.7203 | 154.0616 | 157.9804 | 162.3439 | 166.717 | 170.6611 | 173.025 | 174.5617 |

http://www.cdc.gov/growthcharts/html charts/statage.htm/#females


## Females, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 188.5 | 150.251 | 151.7702 | 154.1119 | 158.0308 | 162.394 | 166.7663 | 170.7091 | 173.0722 | 174.6082 |
| 189.5 | 150.2975 | 151.8171 | 154.1592 | 158.0784 | 162.4414 | 166.8129 | 170.7546 | 173.1168 | 174.6522 |
| 190.5 | 150.3412 | 151.8612 | 154.2037 | 158.1234 | 162.4862 | 166.8571 | 170.7978 | 173.1591 | 174.6938 |
| 191.5 | 150.3823 | 151.9027 | 154.2457 | 158.1659 | 162.5287 | 166.899 | 170.8387 | 173.1992 | 174.7333 |
| 192.5 | 150.4209 | 151.9418 | 154.2854 | 158.2061 | 162.569 | 166.9388 | 170.8775 | 173.2373 | 174.7708 |
| 193.5 | 150.4573 | 151.9787 | 154.3229 | 158.2442 | 162.6072 | 166.9766 | 170.9144 | 173.2734 | 174.8063 |
| 194.5 | 150.4917 | 152.0135 | 154.3584 | 158.2803 | 162.6435 | 167.0125 | 170.9494 | 173.3077 | 174.84 |
| 195.5 | 150.5241 | 152.0465 | 154.3919 | 158.3146 | 162.6781 | 167.0466 | 170.9827 | 173.3402 | 174.8721 |
| 196.5 | 150.5547 | 152.0776 | 154.4238 | 158.3472 | 162.7109 | 167.0791 | 171.0144 | 173.3712 | 174.9025 |
| 197.5 | 150.5837 | 152.1072 | 154.454 | 158.3782 | 162.7421 | 167.11 | 171.0446 | 173.4007 | 174.9314 |
| 198.5 | 150.6111 | 152.1352 | 154.4827 | 158.4077 | 162.7719 | 167.1395 | 171.0733 | 173.4288 | 174.959 |
| 199.5 | 150.6372 | 152.1617 | 154.51 | 158.4357 | 162.8002 | 167.1676 | 171.1007 | 173.4555 | 174.9852 |
| 200.5 | 150.6619 | 152.187 | 154.5359 | 158.4625 | 162.8273 | 167.1944 | 171.1268 | 173.481 | 175.0102 |
| 201.5 | 150.6854 | 152.211 | 154.5607 | 158.4879 | 162.8531 | 167.22 | 171.1517 | 173.5053 | 175.034 |
| 202.5 | 150.7077 | 152.2339 | 154.5842 | 158.5123 | 162.8778 | 167.2444 | 171.1754 | 173.5284 | 175.0567 |
| 203.5 | 150.7289 | 152.2556 | 154.6067 | 158.5355 | 162.9013 | 167.2677 | 171.1981 | 173.5505 | 175.0783 |
| 204.5 | 150.7491 | 152.2764 | 154.6281 | 158.5577 | 162.9238 | 167.29 | 171.2198 | 173.5716 | 175.099 |
| 205.5 | 150.7684 | 152.2962 | 154.6486 | 158.5789 | 162.9454 | 167.3114 | 171.2405 | 173.5918 | 175.1187 |
| 206.5 | 150.7868 | 152.3151 | 154.6681 | 158.5992 | 162.966 | 167.3318 | 171.2604 | 173.6111 | 175.1376 |
| 207.5 | 150.8044 | 152.3332 | 154.6868 | 158.6187 | 162.9858 | 167.3514 | 171.2793 | 173.6295 | 175.1556 |
| 208.5 | 150.8211 | 152.3504 | 154.7047 | 158.6373 | 163.0047 | 167.3701 | 171.2975 | 173.6471 | 175.1728 |
| 209.5 | 150.8372 | 152.3669 | 154.7218 | 158.6551 | 163.0228 | 167.3881 | 171.3149 | 173.664 | 175.1892 |
| 210.5 | 150.8525 | 152.3827 | 154.7382 | 158.6722 | 163.0402 | 167.4053 | 171.3315 | 173.6802 | 175.205 |
| 211.5 | 150.8672 | 152.3979 | 154.754 | 158.6886 | 163.0569 | 167.4218 | 171.3475 | 173.6956 | 175.2201 |
| 212.5 | 150.8812 | 152.4124 | 154.769 | 158.7043 | 163.0729 | 167.4376 | 171.3628 | 173.7104 | 175.2345 |
| 213.5 | 150.8947 | 152.4263 | 154.7835 | 158.7194 | 163.0882 | 167.4528 | 171.3775 | 173.7246 | 175.2483 |
| 214.5 | 150.9076 | 152.4396 | 154.7974 | 158.7339 | 163.103 | 167.4674 | 171.3915 | 173.7382 | 175.2616 |
| 215.5 | 150.92 | 152.4524 | 154.8107 | 158.7478 | 163.1172 | 167.4814 | 171.405 | 173.7513 | 175.2742 |
| 216.5 | 150.9319 | 152.4647 | 154.8235 | 158.7612 | 163.1308 | 167.4948 | 171.418 | 173.7638 | 175.2864 |
| 217.5 | 150.9433 | 152.4765 | 154.8358 | 158.774 | 163.1439 | 167.5078 | 171.4304 | 173.7758 | 175.2981 |
| 218.5 | 150.9542 | 152.4878 | 154.8476 | 158.7864 | 163.1565 | 167.5202 | 171.4424 | 173.7873 | 175.3093 |
| 219.5 | 150.9647 | 152.4987 | 154.859 | 158.7983 | 163.1686 | 167.5321 | 171.4538 | 173.7984 | 175.32 |
| 220.5 | 150.9749 | 152.5092 | 154.8699 | 158.8097 | 163.1802 | 167.5436 | 171.4649 | 173.809 | 175.3303 |

http://www.cdc.gov/growthcharts/html charts/statage.htm/#females


## Females, Stature, Ages 2-20 Years

| Age (in<br>months) | 3rd<br>Percentile<br>Stature (in<br>centimeters) | 5th<br>Percentile<br>Stature (in<br>centimeters) | 10th<br>Percentile<br>Stature (in<br>centimeters) | 25th<br>Percentile<br>Stature (in<br>centimeters) | 50th<br>Percentile<br>Stature (in<br>centimeters) | 75th<br>Percentile<br>Stature (in<br>centimeters) | 90th<br>Percentile<br>Stature (in<br>centimeters) | 95th<br>Percentile<br>Stature (in<br>centimeters) | 97th<br>Percentile<br>Stature (in<br>centimeters) |
|---|---|---|---|---|---|---|---|---|---|
| 221.5 | 150.9846 | 152.5192 | 154.8804 | 158.8207 | 163.1914 | 167.5546 | 171.4755 | 173.8192 | 175.3402 |
| 222.5 | 150.9939 | 152.5289 | 154.8905 | 158.8313 | 163.2022 | 167.5653 | 171.4856 | 173.829 | 175.3497 |
| 223.5 | 151.0029 | 152.5382 | 154.9003 | 158.8415 | 163.2126 | 167.5755 | 171.4954 | 173.8384 | 175.3588 |
| 224.5 | 151.0115 | 152.5472 | 154.9096 | 158.8514 | 163.2226 | 167.5853 | 171.5049 | 173.8474 | 175.3675 |
| 225.5 | 151.0198 | 152.5558 | 154.9187 | 158.8608 | 163.2322 | 167.5948 | 171.5139 | 173.8561 | 175.376 |
| 226.5 | 151.0279 | 152.5641 | 154.9273 | 158.8699 | 163.2415 | 167.6039 | 171.5226 | 173.8645 | 175.384 |
| 227.5 | 151.0356 | 152.5721 | 154.9357 | 158.8787 | 163.2504 | 167.6127 | 171.531 | 173.8725 | 175.3918 |
| 228.5 | 151.043 | 152.5798 | 154.9438 | 158.8872 | 163.259 | 167.6211 | 171.5391 | 173.8802 | 175.3993 |
| 229.5 | 151.0501 | 152.5873 | 154.9516 | 158.8953 | 163.2673 | 167.6293 | 171.5468 | 173.8877 | 175.4064 |
| 230.5 | 151.057 | 152.5944 | 154.959 | 158.9032 | 163.2753 | 167.6371 | 171.5543 | 173.8948 | 175.4133 |
| 231.5 | 151.0636 | 152.6013 | 154.9663 | 158.9107 | 163.283 | 167.6446 | 171.5615 | 173.9017 | 175.42 |
| 232.5 | 151.07 | 152.6079 | 154.9732 | 158.918 | 163.2904 | 167.6519 | 171.5684 | 173.9083 | 175.4264 |
| 233.5 | 151.0762 | 152.6143 | 154.9799 | 158.9251 | 163.2976 | 167.6589 | 171.5751 | 173.9147 | 175.4325 |
| 234.5 | 151.0821 | 152.6205 | 154.9864 | 158.9319 | 163.3045 | 167.6657 | 171.5815 | 173.9208 | 175.4384 |
| 235.5 | 151.0879 | 152.6265 | 154.9926 | 158.9384 | 163.3111 | 167.6722 | 171.5877 | 173.9267 | 175.4441 |
| 236.5 | 151.0934 | 152.6322 | 154.9986 | 158.9447 | 163.3175 | 167.6785 | 171.5937 | 173.9324 | 175.4496 |
| 237.5 | 151.0987 | 152.6377 | 155.0044 | 158.9508 | 163.3237 | 167.6845 | 171.5994 | 173.9379 | 175.4548 |
| 238.5 | 151.1038 | 152.6431 | 155.01 | 158.9567 | 163.3297 | 167.6904 | 171.6049 | 173.9432 | 175.4599 |
| 239.5 | 151.1088 | 152.6482 | 155.0154 | 158.9624 | 163.3354 | 167.696 | 171.6103 | 173.9482 | 175.4648 |
| 240 | 151.1112 | 152.6507 | 155.0181 | 158.9651 | 163.3383 | 167.6987 | 171.6129 | 173.9507 | 175.4671 |

http://www.cdc.gov/growthcharts/html charts/statage.htm/#females


Sponsor: APGD ISN/Protocol: 178-CL-204

## 12.13 Clinical Study Continuity

#### INTRODUCTION

The purpose of this appendix is to provide acceptable alternate methods to assess safety and efficacy parameters, as appropriate, in the event the clinical study is interrupted at the country, state, site or participant level during any crisis (e.g., natural disaster, pandemic).

#### BENEFIT-RISK RATIONALE

Maintaining the safety of clinical study participants and delivering continuity of care in the clinical study setting is paramount during any crisis. The site is expected to follow the protocol and associated Schedule of Assessments [Table 1] unless the site principal investigator discusses the need with the Astellas medical monitor to implement the alternate measures.

The approach outlined within this appendix defines which assessments are required to maintain a favorable benefit/risk to the participant, to maintain overall study integrity and to provide acceptable alternate methods to complete the study required assessments and procedures if study activities are unable to be performed as described in [Section 7 Study Procedures and Assessments] due to a crisis.

#### INFORMED CONSENT

Participants who need to follow any or all of the alternate measures outlined in this Appendix will be required to provide informed consent, which explicitly informs them of the nature of and rationale for these changes, and gain their agreement to continue participation in the study prior to the implementation of any of these changes. In the event the urgency of implementing the alternate measures does not allow for the participant to provide written consent prior to implementation, the principal investigator or designee will obtain oral agreement from the subject followed by written documentation as soon as is feasible. A separate addendum to the study informed consent will be provided to document the participant's consent of the changes.

#### PARTICIPANT PROCEDURES ASSESSMENT

Sites with participants who are currently enrolled into this clinical study may consider implementing the alternate methods outlined below if one or more of the following conditions are met due to the crisis:

- Regional or local travel has been restricted, inclusive of mandatory shelter in place measures, which makes participant travel to/from the study site nearly impossible
- Site facilities have been closed for clinical study conduct
- Site has been restricted to treating patients with conditions outside of the scope of the study
- Site personnel have temporarily relocated the conduct of the study to a location that place a burden on the participant with respect to time and travel

11 Feb 2021 Astellas 
EudraCT number 2016-001767-37


Participant(s) have temporarily relocated from the current study site to an alternate study site to avoid placing a burden on the participant with respect to travel

- Participant(s) have temporarily relocated from their home location and the new distances from the site would cause undue burden with respect to time and travel
- Participant has risk factors for which traveling to the site poses an additional risk to the participant's health and safety

Adherence to the original protocol as reflected in the Schedule of Assessments [Table 1] is expected, where plausible, in the case of a crisis. The alternate measures as noted in [Table 12] below are only permissible in the event of a crisis, and after discussing the need with the Astellas medical monitor to implement the alternate measures. This is to allow for continuity of receiving IP and maintaining critical safety and efficacy assessments for patients participating in the study at a time of crisis.

If one or more of the alternate measures noted below is implemented for a participant, the site should document in the participant's source document the justification for implementing the alternate measure and the actual alternate measures that were implemented, along with the corresponding time point(s).

EudraCT number 2016-001767-37


Table 12 Alternate Schedule of Assessments in Response to a Crisis

| | | Γ | Oouble-blind | Placebo-con<br>(12 weeks) | trolled Perio | od | Follow-up Period (2 weeks) |
|---|---|---|---|---|---|---|---|
| | | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 |
| Critical Assessments | Alternate Approach(es) | Week 0<br>Baseline | Week 2<br>TC <sup>a</sup> | Week 4 | Week 8<br>TC <sup>a</sup> | Week 12<br>(EoT) <sup>b</sup> | Week 14<br>(EoS) <sup>b,c</sup> |
| | | Day -1 | Day 14 (± 3 days) | Day 28 (± 3 days) | Day 56 (± 3 days) | Day 84 (± 3 days) | Day 98<br>(+ 3 days) |
| Previous and Concomitant Medication | Remote/Virtual/Telemedicine Visits allowed. Please refer to protocol schedule of assessments. | X | X | X | X | X | X |
| Physical Examination | The exam can be done at a local clinic and the results submitted to PI. | | | X | | X | |
| Height and Body Weight | Can be obtained at a local clinic or at home | X | | | | X | |
| Dose Titration <sup>d</sup> | Courier service directly to subject. Titration to occur based on PI's evaluation via phone. For tablets: subject to take spare 25 mg tablets until 50 mg wallet is delivered via courier. | | | X | | | |
| Dispense IP <sup>e</sup> | Courier service directly to subject | X | | X | | | |
| Drug Accountability | Used product can be shipped back to site via courier. | X | | | | X | |
| Vital Signs <sup>f</sup> | Can be performed at a local clinic and results submitted to PI for evaluation OR Blood pressure and pulse collected via SBPM and temperature collected at home and reported to site (respiration rate missing). | X | | X | | X | X |
| SBPM <sup>g</sup> | Will be sent to subject's home address | X | X | X | X | X | |
| Table continued on next page | | I. | 1 | 1 | I | | 1 |

EudraCT number 2016-001767-37


| Double-blind Placebo-controlled P (12 weeks) | | | | | trolled Perio | Follow-up Period (2 weeks) | |
|---|---|---|---|---|---|---|---|
| | | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 |
| Critical Assessments | Alternate Approach(es) | Week 0<br>Baseline | Week 2<br>TC <sup>a</sup> | Week 4 | Week 8<br>TC <sup>a</sup> | Week 12<br>(EoT) <sup>b</sup> | Week 14<br>(EoS) <sup>b,c</sup> |
| | | Day -1 | Day 14 (± 3 days) | Day 28 (± 3 days) | Day 56 (± 3 days) | Day 84 (± 3 days) | Day 98<br>(+ 3 days) |
| Routine 12-lead ECG <sup>f</sup> | ECG testing can be completed at local clinic. | X | | X | | X | |
| Clinical Laboratory Tests (Hematology and Biochemistry) <sup>h</sup> | Visit collection of samples at local facility acceptable if results can be made available to investigative site. | Xi | | X | | X | X <sup>i</sup> |
| Clinical Laboratory Tests (Urinalysis) <sup>h</sup> | Visit collection of samples at local facility acceptable if results can be made available to investigative site. | Xi | | X | | X | Xi |
| Pregnancy Test <sup>i</sup> | Visit collection of samples at local facility acceptable if results can be made available to investigative site. | X | | X | | X | X |
| AEs | Remote/Virtual/Telemedicine Visits allowed. Please refer to protocol schedule of assessments. | X | X | X | X | X | X |
| Bladder e-diary | Will be sent to subject's home address | X | X | X | X | X | |
| Acceptability and Palatability Questionnaire <sup>j</sup> | To be performed remotely via e-diary. | | | | | X | |
| Pharmacokinetics <sup>k</sup> | Astellas Medical Monitor to assess. Not allowed at an alternate clinical due to special sample handling. | | | X | | X | |

AE: adverse event; ECG: electrocardiogram; e-diary: electronic diary; EoS: end of study; EoT: end of treatment; IP: investigational product; OAB: overactive bladder; PED25: pediatric equivalent dose 25 mg; PED50: pediatric equivalent dose 50 mg; PI: principal investigator; SBPM: self blood pressure monitoring; TC: telephone call *Footnotes continued on next page* 

Sponsor: APGD

EudraCT number 2016-001767-37


a. For the visits where a TC is indicated, there is no need for the subject to visit the clinic provided that the bladder e-diary data are reviewed by the investigator prior to the TC and discussed and confirmed with the subject or parent(s)/legal guardian(s) during the TC. Urotherapy is also to be discussed and confirmed with the subject or parent(s)/legal guardian(s) during each TC as indicated in Table 1.

- b. Subjects who withdraw early from the study after having received IP should complete both the EoT and EoS visits.
- c. The EoS visit (visit 8/week 14 [EoS]) should take place at least 14 days after the EoT visit (visit 7/week 12 [EoT]).
- d. Dose up-titration to PED50 to occur at visit 5/week 4 unless investigator determines OAB is adequately controlled. Dose down-titration from PED50 to PED25 can be done at any time for safety reasons.
- e. Daily IP administration will start on day 1 (i.e., the day after visit 3/week 0 [baseline]).
- f. Blood pressure, pulse, body temperature and ECGs will all be measured in single measurements. Subject to be in the sitting position (when possible, otherwise supine, but always in the same position for each procedure). Subject should have been calm and without distress for at least 5 minutes. Preferably, the right arm should be used to measure vital signs. Body temperature will be measured with an ear thermometer. Clinic measurements will be used to assess eligibility.
- g. SBPM will be measured once in the morning and evening during the 2-day weekend bladder e-diary collection period. SBPM measurements should start in the weekend prior to week -2 and be taken in the weekend prior to the indicated visit (or TC). SBPM will be measured on 2 consecutive days at 1 and 2 weeks after start of dosing with PED25 (day 1) and after up-titration to PED50, if not already covered by the scheduled SBPM. Measurements will be taken in the sitting position (when possible, otherwise supine, but always in the same position). Preferably, the right arm should be used. Subject should have been calm and without distress for at least 5 minutes. Morning measurement should be taken before IP intake and evening measurement should be taken prior to bedtime.
- h. Additional hematology, biochemistry and urinalysis (urinalysis dipstick) tests will be performed at visit 3/week 0 (baseline) and visit 8/week 14 (EoS) only if an AE related to hematology, biochemistry or urinalysis parameters occurred since the previous visit or at the discretion of the investigator.
- i. Urine pregnancy test will be performed for females of childbearing potential at all on-site visits.
- j. The acceptability and palatability questionnaire will be completed on one weekend day preceding at visit 7/week 12 (EoT).
- k. There will be 2 pharmacokinetic sampling days at visit 5/week 4 and visit 7/week 12 (EoT). Both pharmacokinetic sampling days will consist of collecting 1 predose (trough) sample. On pharmacokinetic sampling days, dosing should occur in the clinic and breakfast should be eaten at the clinic within 1 hour before dosing.


# INVESTIGATIONAL PRODUCT SUPPLY

If any of the conditions outlined above in the Participant Procedures Assessment are met, if the following mitigating strategy will be employed, as needed, to ensure continuity of IP supply to the participants:

• Increase stock of IP on site to reduce number of shipments required, if site space will allow.

ISN/Protocol: 178-CL-204

• Direct-to-subject shipments of IP from the site to the subject's home.

# DATA COLLECTION REQUIREMENTS

Additional data may be collected in order to indicate how participation in the study may have been affected by a crisis and to accommodate data collection resulting from alternate measures implemented to manage the conduct of the study and participant safety.

• Critical assessments for safety and efficacy based on study endpoints to be identified as missing or altered (performed virtually, at alternative locations, out of window, or other modifications) due to the crisis.

12.14 List of Abbreviations and Definition of Key Study Terms

# **List of Abbreviations**

| Abbreviation | Description |
|---|---|
| APEB | Astellas Pharma Europe B.V. |
| APGD | Astellas Pharma Global Development Inc. |
| AE | adverse event |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| AR | adrenergic receptor |
| AST | aspartate aminotransferase |
| AT | aminotransferases |
| ATC | Anatomical Therapeutic Chemical |
| AUC | area under the concentration-time curve |
| AUC <sub>24</sub> | area under the concentration-time curve from time zero to 24 hours |
| AUCtau | area under concentration-time curve over dosing interval |
| AUC <sub>inf</sub> | area under the concentration-time curve from the time of dosing extrapolated to |
| ALIC | time infinity area under the concentration-time curve from the time of dosing to the last |
| $AUC_{last}$ | E |
| DMI | measurable concentration |
| BMI | body mass index |
| CDE | maximum drug concentration |
| CRF | case report form |
| CRO | contract research organization |
| CSR | clinical study report |
| CV | coefficient of variation |
| CY | cytochrome |
| DBP | diastolic blood pressure |
| DPD | Data Protection Directive |
| DSMB | Data and Safety Monitoring Board |
| EBC | expected bladder capacity |
| ECG | electrocardiogram |
| eCOA | electronic clinical outcome assessment |
| e-diary | electronic diary |
| EEA | European Economic Area |
| EMA | European Medicines Agency |
| EMG | electromyography |
| EoS | end of study |
| ЕоТ | end of treatment |
| FAO | Food and Agricultural Organization |
| FAS | full analysis set |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| hCG | human chorionic gonadotropin |
| ICCS | International Children's Continence Society |
| ICF | informed consent form |
| ICH | International Council for Harmonisation of Technical Requirements for |
| | Pharmaceuticals for Human Use |


| Abbussistics | Description |
|-------------------|--------------------------------------------------|
| Abbreviation IDAC | Description in description |
| | independent data analysis center |
| IEC | Independent Ethics Committee |
| INR | international normalized ratio |
| IP | investigational product |
| IRB | Institutional Review Board |
| IRT | interactive response technology |
| ISN | international study number |
| LA-CRF | liver abnormality case report form |
| LOCF | last observation carried forward |
| LQTS | long QT syndrome |
| LS | least squares |
| NDO | neurogenic detrusor overactivity |
| NONMEM | non-linear mixed effects modeling |
| OAB | overactive bladder |
| OCAS | oral-controlled absorption system |
| PED | pediatric equivalent dose |
| P-gp | P-glycoprotein |
| PIP | pediatric investigational plan |
| PKAS | pharmacokinetic analysis set |
| PPIUS | Patient perception of intensity of urgency scale |
| PPS | per protocol set |
| PVR | post void residual |
| QA | quality assurance |
| QC | quality control |
| QTL | quality tolerance limit |
| SAE | serious adverse event |
| SAF | safety analysis set |
| SAP | statistical analysis plan |
| SBP | systolic blood pressure |
| SBPM | self-blood pressure measurement |
| SOP | standard operating procedure |
| SUSAR | serious unexpected serious adverse reaction |
| TEAE | treatment-emergent adverse event |
| TBL | total bilirubin |
| TC | telephone call |
| USM | urgent safety measure |
| ULN | upper limit of normal |
| UTI | urinary tract infection |
| WHO-DD | WHO-Drug Dictionary |
| ,,110 DD | 1110 Diag Dictionary |

EudraCT number 2016-001767-37


# **Definition of Key Study Terms**

| Terms | Definition of Terms |
|---|---|
| Baseline | Assessments of subjects as they enter a study before they receive any treatment. |
| Endpoint | Variable that pertains to the efficacy or safety evaluations of a study. |
| | Note: Not all endpoints are themselves assessments since certain endpoints might apply to populations or emerge from analysis of results. That is, endpoints might be facts about assessments (e.g., prolongation of survival). |
| Enroll | To register or enter a subject into a study. Note: Once a subject has received the IP or placebo, the protocol applies to the subject. |
| Intervention | The drug, device, therapy or process under investigation in a study that is believed to have an effect on outcomes of interest in a study (e.g., health-related quality of life, efficacy, safety and pharmacokinetics). |
| Investigational period | Period of time where major interests of protocol objectives are observed, and where the test product or comparative drug (sometimes without randomization) is given to a subject and continues until the last assessment after completing administration of the test product or comparative drug. |
| Post investigational period | Period of time after the last assessment of the protocol. Follow-up observations for sustained adverse events and/or survival are done in this period. |
| Randomization | The process of assigning subjects to treatment or control groups using an element of chance to determine assignments in order to reduce bias. |
| | NOTE: Unequal randomization is used to allocate subjects into groups at a differential rate; for example, three subjects may be assigned to a treatment group for everyone assigned to the control group. |
| Screening | A process of active consideration of potential subjects for randomization in a study. |
| Screen failure | Potential subject who signed the ICF/assent but did not meet 1 or more criteria required for participation in the study and was not randomized. |
| Screening period | Period of time before entering the investigational period, usually from the time when a subject signs the consent/assent form until just before the test product or comparative drug (sometimes without randomization) is given to a subject. |
| Study period | Period of time from the first study site initiation date to the last study site completing the study. |
| Variable | Any quantity that varies; any attribute, phenomenon or event that can have different qualitative or quantitative values. |

Sponsor: APGD EudraCT number 2016-001767-37 - CONFIDENTIAL - ISN/Protocol: 178-CL-204

# 13 ATTACHMENT 1: SUBSTANTIAL AMENDMENT 1

# I. The purpose of this amendment is:

# **Substantial Changes**

# 1. Update Schedule of Assessments

# **DESCRIPTION OF CHANGE:**

The schedule of assessments is updated with the following changes:

- Physical examination is added to visit 5 (week 4).
- Height and body weight measurement is added to visit 7 (week 12).
- Clinical Laboratory Tests (Hematology and Biochemistry) footnote is removed from visit 5 (week 4)
- Self-blood pressure measurement (SBPM) is added visit 2 (week -2) and removed from visit 8 (week 14).
- Pregnancy tests are added to visit 3 (week 0), visit 5 (week 4) and visit 7 (week 12).
- Additional text is added to footnote h to explain that the SBPM should be done during the weekend preceding the study visit.
- Footnote i is revised to remove visit 5 (week 4).
- Footnote j is revised to clarify that urine pregnancy tests will be performed for females of childbearing potential at all on-site visits.

#### RATIONALE:

This is a combination of regulatory commitments to include additional pregnancy testing and laboratory testing, as well as fixing some errors for clarification.

Footnote i was removed from the Clinical Laboratory Tests at visit 5 (week 4), because this visit is now required.

# 2. Update Subject Weight Range

# **DESCRIPTION OF CHANGE:**

The minimum weight of subjects is changed from 11 kg to 13 kg. This is updated in the dose rationale and Inclusion Criterion #4.

# **RATIONALE:**

This study should only include children and adolescents from 5 years to 18 years; therefore, the lower weight limit was revised.

#### 3. Delete Exclusion Criterion #11

# **DESCRIPTION OF CHANGE:**

A criterion (#11) that subjects must have a pulse of  $> 99^{th}$  percentile for age at Screening is deleted.

11 Feb 2021 Astellas 

EudraCT number 2016-001767-37


# RATIONALE:

This criterion is the same as exclusion criterion #33 because the criterion was originally checked at screening <u>and</u> baseline. The criterion itself still applies to subjects, but is only needed at baseline.

# 4. Update Exclusion Criterion #13

# DESCRIPTION OF CHANGE:

Text is added to allow the option that the subject is currently taking medication known to prolong the QT interval.

# RATIONALE:

This revision is made for consistency with Table 21 in the Investigator's Brochure.

# 5. Update Exclusion Criterion #18

# **DESCRIPTION OF CHANGE:**

The criterion is updated to exclude subjects who use moderate or strong cytochrome CYP3A4/5 or P-gp inhibitors or inducers.

# RATIONALE:

This revision is made per a Regulatory request.

# **Nonsubstantial Changes**

# 1. Update Key Sponsor Personnel

# DESCRIPTION OF CHANGE:

Contact details for medical monitor are updated.

#### RATIONALE:

Contact details of medical monitor are updated based on changes to study personnel.

# 2. Update Compound Name

# **DESCRIPTION OF CHANGE:**

The compound name has been updated to YM178 (from ED178).

#### RATIONALE:

This revision is made to correct an error. ED178 is the project name for pediatric.

EudraCT number 2016-001767-37


# 3. Update Planned Study Period

# **DESCRIPTION OF CHANGE:**

The planned completion date is extended to 2Q2023 (from 3Q2022).

#### RATIONALE:

This revision is made based on current enrollment projections.

# 4. Update Background

# **DESCRIPTION OF CHANGE:**

Text regarding mirabegron mechanism of action is added to the Background section.

#### RATIONALE:

This revision is made for consistency with the current Mirabegron Investigator's Brochure.

# 5. Updated Total Number and Location of Study Sites

# **DESCRIPTION OF CHANGE:**

The number of planned study sites is increased to 65 (from 50) and North America is added as a study site location.

# RATIONALE:

The planned number of study sites is increased to account for the current number of approved sites. The revision to study location is made to correct an error. During development of the statistical analysis plan, it was noted that North America was not listed in the protocol.

# 6. Update Study Objectives and Endpoints

# DESCRIPTION OF CHANGE:

Text is added to note that primary and secondary objectives and endpoints apply to children only; exploratory objectives and endpoints also apply to adolescents. Subject age is added to the exploratory objective. Mean number of micturitions per 24 hours is added as an exploratory endpoint.

# RATIONALE:

These revisions are made for clarification. To ensure mean micturitions is analyzed for adolescents. The mean number of micturitions endpoint is added ensure mean micturitions is analyzed for adolescents.

# 7. Clarify Exclusion Criterion #19

# **DESCRIPTION OF CHANGE:**

The criterion is updated to add the text 'and cannot be discontinued.'

11 Feb 2021 Astellas 

EudraCT number 2016-001767-37


# RATIONALE:

This revision is made to for clarification. If the prohibited medication can be discontinued, the subject may be enrolled in the study.

# 8. Clarify Reference for Investigational Products (IP)

# **DESCRIPTION OF CHANGE:**

Section 6.1.1 is updated to clarify that detailed information on mirabegron granules for oral suspension is located in the Investigator's Brochure and Investigational Medicinal Product Dossier.

# RATIONALE:

The original protocol stated where to locate additional information for tablets only, so text is added on where to find additional information for the granules.

# 9. Update Subject Compliance

# **DESCRIPTION OF CHANGE:**

Weighing is added a method for assessing compliance of subject compliance with IP.

# **RATIONALE:**

This revision is made for clarification. Tablets will be counted and granules for oral suspension will be weighed.

# 10. Expand Urotherapy Information in Section 6.4.2

# **DESCRIPTION OF CHANGE:**

Additional information about urotherapy is added to Section 6.4.2.

#### RATIONALE:

This revision is made for clarification.

# 11. Update Concomitant Medications

# DESCRIPTION OF CHANGE:

Medications that prolong the QT interval, and medications that are moderate or strong cytochrome CYP3A4/5 or P-gp inhibitors, are added to the list of prohibited concomitant medications. Examples of medications used for the treatment of overactive bladder are added.

EudraCT number 2016-001767-37


#### RATIONALE:

In accordance with Section 6.5.3 of the Investigator's Brochure, these medications are added on the list of concomitant medications excluded from the protocol.

# 12. Update Description of Physical Examination

# **DESCRIPTION OF CHANGE:**

Additional details of the physical examination are added to Section 7.2.4.

#### RATIONALE:

This revision is made for clarification.

# 13. Update Total Amount of Blood

# **DESCRIPTION OF CHANGE:**

The number of clinical laboratory samples and total blood volume are updated.

# RATIONALE:

This revision is made since visit 5 (week 4) is now mandatory. The blood volumes are updated to account for the clinical laboratory tests at this visit.

# 14. Define Pharmacokinetic Parameters

# DESCRIPTION OF CHANGE:

The pharmacokinetic parameters that will be calculated as part of the secondary pharmacokinetic endpoint are defined.

# RATIONALE:

The specific pharmacokinetic parameters to be calculated were not previously defined.

# 15. Clarify Electronic Clinical Outcome Assessments

# **DESCRIPTION OF CHANGE:**

Section 7.6, Electronic Clinical Outcome Assessment, is updated to provide additional information about the integrity of the data. Additional text from the latest Global Protocol Format (GPF) is added.

# RATIONALE:

These revisions are made to describe how the integrity of the data is ensured, especially the data subjects enter into electronic forms.

11 Feb 2021 Astellas 

EudraCT number 2016-001767-37


# 16. Update Subject Discontinuation Criteria

# **DESCRIPTION OF CHANGE:**

The following criteria are added as reasons that a subject may be discontinued from study treatment:

- Pregnancy
- Prolongation of QT > QTcF > 440 msec and/or QT interval prolongation > 30 msec
- Systolic blood pressure ≥ 160 mm Hg or diastolic blood pressure ≥ 100 mmHg

Follow-up for prolongation of QT intervals is added to Section 9.5.5.

#### RATIONALE:

These revisions are made due to regulatory agency feedback/request.

# 17. Update Rationale for Sample Size

# **DESCRIPTION OF CHANGE:**

Text is added to state that the assumptions about sample size, in addition to the levels for Type-1 error and power, were agreed upon with Pediatric Committee in the current Pediatric Investigation Plan.

# RATIONALE:

This revision is made for clarification of assumptions.

# 18. Clarify Local Laboratory Evaluations

# **DESCRIPTION OF CHANGE:**

Text is added to clarify that when local laboratory evaluations are conducted, the values obtained will be adjusted to values obtained by the central laboratory. A reference is made to the statistical analysis plan.

#### RATIONALE:

This revision is made to indicate how the local lab values will be analyzed when the modified schedule of assessments is utilized.

#### 19. Add Section for Independent Data Analysis Center (IDAC)

# **DESCRIPTION OF CHANGE:**

A new section is added to Section 10, Operational Considerations, to describe the purpose of the IDAC and its members.

# RATIONALE:

This revision is made to clarify the role of the IDAC and the interactions between the IDAC and the Data and Safety Monitoring Board.

11 Feb 2021 Astellas 

EudraCT number 2016-001767-37


# 20. Update Source Documents

# **DESCRIPTION OF CHANGE:**

Appendix 12.1.6, Source Documents, is updated with compulsory text from the latest GPF.

#### RATIONALE:

This revision is made to align the study protocol with the current GPF and to add additional information for ensuring integrity of data.

#### 21. Remove Source Data Verification

#### **DESCRIPTION OF CHANGE:**

Information about source data verification is removed from Section 10.1, *Data Collection* and 12.2.1, *Study Monitoring*. Information about source data review is added to Appendix 12.1.6, *Source Documents*.

# RATIONALE:

This revision is made to comply with the European guidelines published by the European Commission regarding the remote source data verification during the COVID-19 pandemic.

# 22. Update Contraception Requirements

# DESCRIPTION OF CHANGE:

Appendix 12.3 is updated with standard text from the latest GPF in regards to contraception requirements for pediatric subjects.

#### RATIONALE:

This revision is made to align the study protocol with the current GPF and to provide pediatric-specific contraception requirements.

# 23. Clarify Abnormal Laboratory Findings

# DESCRIPTION OF CHANGE:

Updates are made to Appendix 12.4.1.1 to clarify abnormal laboratory findings and the process for reporting them.

# RATIONALE:

This revision is made in accordance to the Agency's comment on laboratory values,

# 24. Update List of Excluded Concomitant Medications

# **DESCRIPTION OF CHANGE:**

The List of Excluded Concomitant Medications in Appendix 12.6 is updated to include moderate and strong CYP3A4 inhibitors and inducers, and P-gp inhibitors and inducers

11 Feb 2021 Astellas 

Sponsor: APGD

EudraCT number 2016-001767-37


# RATIONALE:

This revision is made to incorporate the moderate and strong cytochrome CYP3A4/5 and P-gp inhibitors and inducers that are added to Exclusion Criterion #18.

ISN/Protocol: 178-CL-204

# 25. Add Appendix for Clinical Study Continuity

# **DESCRIPTION OF CHANGE:**

A Clinical Study Continuity appendix is added to the protocol. This appendix contains procedures for continuity of care during a crisis. An alternative schedule of assessments is provided. A reference to this appendix is added to Section 7.

# RATIONALE:

This appendix is added to provide acceptable alternate methods to assess safety and efficacy parameters in the event the clinical study is interrupted at the country, state, site or participant level during any crisis (e.g., natural disaster or pandemic).

# 26. Minor Administrative-type Changes

# **DESCRIPTION OF CHANGE:**

Include minor administrative-type changes (e.g., typos, format, numbering and consistency throughout the protocol); change 'woman of childbearing potential' to 'female of childbearing potential;=' revise wording of Inclusion Criterion #13 from 'must not donate' to 'must agree not to donate;' remove 'Draft' from 'Draft Results' in title of Table 4; add "or designee" as a reviewer for e-diary data in Section 7.1.1; and remove 'WOCBP' from the List of Abbreviations.

# RATIONALE:

To provide clarifications to the protocol and to ensure complete understanding of study procedures.

EudraCT number 2016-001767-37


# **II. Amendment Summary of Changes:**

# **IIA. Substantial Changes**

# 1 Protocol Summary

1.3 Schedule of Assessments

# WAS:

| | Screening Period/Urotherapy (4 weeks) | | - | Double-blind Placebo-controlled Period (12 weeks) | | | | Follow-up Period (2 weeks) |
|---|---|---|---|---|---|---|---|---|
| | Visit 1 | Visit 2/TC <sup>a</sup> | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 |
| Schedule of Assessments | Week -4 | Week -2 | Week 0 | Week 2 | Week 4 | Week 8 | Week 12 | Week 14 |
| | Screening | | Baseline | TCa | | $TC^a$ | (EoT) <sup>b</sup> | $(EoS)^{b,c}$ |
| | Day -28 | Day -14 | Day -1 | Day 14 | Day 28 | Day 56 | Day 84 | Day 98 |
| | (-3 days) | (± 5 days) | | (± 3 days) | (± 3 days) | $(\pm 3 \text{ days})$ | (± 3 days) | (+ 3 days) |
| Physical Examination | X | | | | | | X | |
| Height and Body Weight | X | | X | | | | | |
| Clinical Laboratory Tests (Hematology and Biochemistry) | X | | Xi | | Xi | | X | Xi |
| Clinical Laboratory Tests (Urinalysis) | X | | Xi | | X | | X | Xi |
| SBPM <sup>h</sup> | | | X | X | X | X | X | X |
| Pregnancy Test <sup>j</sup> | X | | | | | | | X |
| Bladder e-diary <sup>a,1</sup> | X | X | X | X | X | X | X | |

- h. SBPM will be measured once in the morning and evening during the 2 day weekend bladder e-diary collection period. SBPM will be measured on 2 consecutive days at 1 and 2 weeks after start of dosing with PED25 (day 1) and after up-titration to PED50, if not already covered by the scheduled SBPM. Measurements will be taken in the sitting position (when possible, otherwise supine, but always in the same position). Preferably, the right arm should be used. Subject should have been calm and without distress for at least 5 minutes. Morning measurement should be taken before IP intake and evening measurement should be taken prior to bedtime.
- i. Additional hematology, biochemistry and urinalysis (urinalysis dipstick) tests will be performed at visit 3/week 0 (baseline), visit 5/week 4 and visit 8/week 14 (EoS) only if an AE related to hematology, biochemistry or urinalysis parameters occurred since the previous visit or at the discretion of the investigator.
- j. Serum pregnancy test at screening and EoS (visit 8/week 14).
- 1. After a successful screening visit (visit 1/week -4 [screening]), all subjects will start with the completion of a 2-day bladder e-diary to get acquainted with the bladder e-diary and the assessments. Completion of this bladder e-diary should start in the weekend prior to week -2. Subjects will start with the 7-day bladder e diaries, approximately 7 days prior to the indicated visit (or TC). The bladder e-diary is used for a 7-day period to record micturition frequency and incontinence episodes; it also contains a 2-day weekend period to record additional volume measurements and vital signs.

EudraCT number 2016-001767-37


IS AMENDED TO:

**Physical Examination** 

Height and Body Weight

Clinical Laboratory Tests (Urinalysis)

Clinical Laboratory Tests (Hematology and Biochemistry)

before IP intake and evening measurement should be taken prior to bedtime.

#### Screening Period/Urotherapy Follow-up Period Double-blind Placebo-controlled Period (4 weeks) (2 weeks) (12 weeks) Visit 1 Visit 2/TCa Visit 3 Visit 4 Visit 5 Visit 7 Visit 8 Visit 6 Week -4 Week -2 Week 0 Week 2 Week 4 Week 8 Week 12 Week 14 Schedule of Assessments Baseline $TC^a$ $TC^a$ (EoT)b $(EoS)^{b,c}$ Screening

Day -14

 $(\pm 5 \text{ days})$ 

Day 14

 $(\pm 3 \text{ days})$ 

Day -1

X

 $\mathbf{X}^{i}$ 

 $X^{i}$ 

Day 28

 $(\pm 3 \text{ days})$ 

X

 $X^{i}$ 

X

Day 56

 $(\pm 3 \text{ days})$ 

Day 84

 $(\pm 3 \text{ days})$ 

X

X

X

X

Day 98

(+ 3 days)

 $X^i$ 

 $X^i$ 

| SBPM <sup>h</sup> | | X | X | X | X | X | X | X |
|---|---|---|---|---|---|---|---|---|
| Pregnancy Test <sup>j</sup> | X | | X | | X | | X | X |
| Bladder e-diary <sup>a,l</sup> | X | X | X | X | X | X | X | |
| h. SBPM will be measured once in the morning and evening during the 2 day weekend bladder e-diary collection period. SBPM measurements should start in the weekend prior to | | | | | | | | |
| week -2 and be taken in the weekend prior to the indicated visit (or TC). SBPM will be measured on 2 consecutive days at 1 and 2 weeks after start of dosing with PED25 (day | | | | | | | | |
| 1) and after up-titration to PED50, if not already covered by the scheduled SBPM. Measurements will be taken in the sitting position (when possible, otherwise supine, but always | | | | | | | | |
| in the same position). Preferably, the right arm should be u | in the same position). Preferably, the right arm should be used. Subject should have been calm and without distress for at least 5 minutes. Morning measurement should be taken | | | | | | | |

- i. Additional hematology, biochemistry and urinalysis (urinalysis dipstick) tests will be performed at visit 3/week 0 (baseline), visit 5/week 4-and visit 8/week 14 (EoS) only if an AE related to hematology, biochemistry or urinalysis parameters occurred since the previous visit or at the discretion of the investigator.
- j. UrineSerum pregnancy test will be performed for females of childbearing potential at screening and EoS (visit 8/week 14) all on-site visits.

Day -28

(-3 days)

X

X

X

X

1. At the end of After a successful screening visit (visit 1/week -4 [screening]), all subjects will be provided with a device to collect diary information. At start with the completion of a 2 day bladder e diary to get acquainted with the bladder e diary and the assessments. Completion of this bladder e diary should start in the weekend prior to the week -2 visit, the subject will complete the 2-day bladder e-diary to get acquainted with the data collection. The 2-day diary will be reviewed at the week -2 visit. If completion is successful, all. Ssubjects will start with the 7-day bladder e-diaryies-completion, approximately 7 days prior to the indicated visit (or TC). The bladder e-diary is used for a 7-day period to record micturition frequency and incontinence episodes; it also contains a 2-day weekend period to record additional volume measurements and vital signs.

EudraCT number 2016-001767-37


# 1 Protocol Summary and 5 Study Population

5.1 Inclusion Criterion #4

WAS:

Subject weighs at least 11 kg at screening.

IS AMENDED TO:

Subject weighs at least 1311 kg at screening.

# 1 Protocol Summary and 5 Study Population

5.1 Exclusion Criterion #11

WAS

Subject has a pulse > 99th percentile for age

IS AMENDED TO:

Subject has a pulse > 99th percentile for ageCriterion has been removed.

# 1 Protocol Summary and 5 Study Population

5.1 Exclusion Criterion #13

WAS:

Subject has QTcF > 440 msec on screening ECG or a risk of QT prolongation (e.g., hypokalemia, long QT syndrome [LQTS] or family history of LQTS or exercise-induced syncope).

# IS AMENDED TO:

Subject has QTcF > 440 msec on screening ECG, or a risk of QT prolongation (e.g., hypokalemia, long QT syndrome [LQTS] or family history of LQTS or exercise-induced syncope) or is currently taking medication known to prolong the QT interval.

# 1 Protocol Summary and 5 Study Population

5.1 Exclusion Criterion #18

WAS:

Subject uses any drugs that are sensitive cytochrome P450 2D6 (CYP2D6) substrates with a narrow therapeutic index or sensitive P-glycoprotein (P-gp) substrates after the start of washout.

# IS AMENDED TO:

Subject uses any drugs that are sensitive cytochrome P450 2D6 (CYP2D6) substrates with a narrow therapeutic index, or sensitive P-glycoprotein (P-gp) substrates, or moderate or strong cytochrome CYP3A4/5 or P-gp inhibitors or inducers after the start of washout.


# **IIB. Nonsubstantial Changes**



ISN/Protocol: 178-CL-204

# 2 Introduction

2.1 Background

#### ADDED:

Mirabegron activation of beta 3-AR in the human bladder results in a relaxation of the detrusor smooth muscle during the fill-void cycle without interfering with the voiding contraction.

#### 2 Introduction

2.1.2.2 Clinical Data (Table 4)

# WAS:

The data from Studies 178 CL 201 and 178 CL 202 were used to support the use of tablets in pediatric subjects with a body weight of  $\geq$  35 kg in this study. For those pediatric subjects that cannot be dosed with tablets because their body weight is < 35 kg or because they cannot be dosed with tablets, an oral suspension with a strength of 2 mg/mL was developed.

Study 178-CL-208 Draft Results: Relative Bioavailability of the Mirabegron 8 mg/mL Oral

11 Feb 2021 Astellas 


Suspension Formulation Versus 2 mg/mL Oral Suspension Formulation (Pharmacokinetics Analysis Set)

ISN/Protocol: 178-CL-204

The doses described in [Section 2.1.2.2 Clinical Data] suggest tablets for subjects with a body weight of  $\geq$  35 kg unless unable to swallow tablets and would be provided the oral suspension as an alternative, and the 8 mg/mL oral suspension for subjects with a body weight  $\leq$  35 kg or those who cannot be dosed with the tablets.

# IS AMENDED TO:

The data from Studies 178 CL 201 and 178 CL 202 were used to support the use of tablets in pediatric subjects with a body weight of  $\geq$  35 kg in this study. For those pediatric subjects that cannot be dosed with tablets because their body weight is < 35 kg or because they cannot be dosed withswallow the tablets, an oral suspension with a strength of 2 mg/mL was developed.

Study 178-CL-208 <del>Draft</del>-Results: Relative Bioavailability of the Mirabegron 8 mg/mL Oral Suspension Formulation Versus 2 mg/mL Oral Suspension Formulation (Pharmacokinetics Analysis Set)

The doses described in [Section 2.1.2.2 Clinical Data] suggest tablets for subjects with a body weight of  $\geq$  35 kg unless unable to swallow tablets and would be provided the oral suspension as an alternative, and the 8 mg/mL oral suspension for subjects with a body weight  $\leq$  35 kg or those who cannot be dosed with the tablets.

#### 2 Introduction

# 2.3 Risk-Benefit Assessment

# WAS:

• Potential UTI will be monitored by urinalysis at each visit in the clinic and will require discontinuation of study treatment

The blood draws for clinical laboratory tests have been minimized to lessen subject burden while ensuring subject safety. Additional hematology and biochemistry tests will be performed at visit 3/week 0 (baseline), visit 5/week 4 and visit 8/week 14 (end of study [EoS]) only if an AE related to hematology, biochemistry or urinalysis parameters occurred since the previous visit or at the discretion of the investigator.

#### IS AMENDED TO:

• Potential UTI will be monitored by urinalysis at each visit in the clinic and will require discontinuation of study treatment

The blood draws for clinical laboratory tests have been minimized to lessen subject burden while ensuring subject safety. Additional hematology and biochemistry tests will be performed at visit 3/week 0 (baseline), visit 5/week 4 and visit 8/week 14 (end of study [EoS]) only if an AE related to hematology, biochemistry or urinalysis parameters occurred since the previous visit or at the discretion of the investigator.


ponsor: APGD ISN/Protocol: 178-CL-204

# **1 Protocol Summary and 3 Study Objectives and Endpoints** *1.1 Synopsis*

# WAS:

| WAS: | |
|---|---|
| Secondary continued | |
| To evaluate the pharmacokinetics after multiple<br>dose administration of mirabegron in pediatric<br>subjects with OAB | Appropriate pharmacokinetic parameters will be calculated based on the population pharmacokinetic model used |
| Exploratory | |
| To evaluate the efficacy of mirabegron in pediatric subjects with OAB | <ul> <li>Percentage of subjects with a reduction in daytime incontinence episodes (&lt; 50% reduction [nonresponder], 50% [partial responder] and 100% [responder])</li> <li>Improvement from baseline in worst incontinence grading</li> <li>Change from baseline at the end of the 12-week treatment period adjusted for fluid intake: <ul> <li>Mean number of micturitions per 24 hours</li> </ul> </li> <li>Change from baseline at the end of the 12-week treatment period (adolescents only): <ul> <li>Mean number of daytime micturitions per 24 hours</li> <li>Mean volume voided per 24 hours</li> <li>Mean number of incontinence episodes per 24 hours</li> </ul> </li> <li>Number of dry (incontinence-free) days per 7 days at the end of the 12-week treatment period (adolescents only)</li> <li>Mean number of daytime grade 3 or 4 (PPIUS)</li> </ul> |

# IS AMENDED TO:

# Primary and secondary objectives and endpoints apply to children only; exploratory objectives and endpoints also apply to adolescents.

only)

Secondary continued

| • | To evaluate the pharmacokinetics after |
|---|-----------------------------------------------|
| | multiple dose administration of mirabegron in |
| | pediatric subjects with OAB |

Steady-state C<sub>max</sub>, AUC<sub>tau</sub>, C<sub>trough</sub>, T<sub>max</sub>, CL/F and Vz/F. Additional parameters may be calculated based on the population pharmacokinetic model used Appropriate pharmacokinetic parameters will be calculated based on the population pharmacokinetic model used

urgency episodes per 24 hours (adolescents

# Exploratory

• To evaluate the efficacy of mirabegron in pediatric subjects (5 to < 18 years) with OAB

- Percentage of subjects with a reduction in daytime incontinence episodes (< 50% reduction [nonresponder], 50% [partial responder] and 100% [responder])
- Improvement from baseline in worst incontinence grading
- Change from baseline at the end of the 12-week treatment period adjusted for fluid intake:

11 Feb 2021 Astellas 

Sponsor: APGD ISN/Protocol: 178-CL-204 EudraCT number 2016-001767-37


Mean number of micturitions per 24 hours Change from baseline at the end of the 12-week treatment period (adolescents only): Mean number of micturitions per 24 hours

- Mean number of daytime micturitions per
- 24 hours
- Mean volume voided per 24 hours
- Mean number of incontinence episodes per
- Number of dry (incontinence-free) days per 7 days at the end of the 12-week treatment period (adolescents only)
- Mean number of daytime grade 3 or 4 (PPIUS) urgency episodes per 24 hours (adolescents only)

# 1 Protocol Summary and 4 Study Design and Dose Rationale

4.1 Study Design

WAS:

Planned total number of study sites include approximately 50 study sites across Europe, Latin America, Africa, Middle East, and Asia-Pacific and North America.

# IS AMENDED TO:

Planned total number of study sites includes approximately 6550 study sites across Europe, Latin America, Africa, Middle East, and Asia-Pacific and North America

# 4 Study Design and Dose Rationale

4.2 Dose Rationale

WAS:

For dosing with oral suspension, the weight range to be covered is from 11 kg (the approximate body weight of a 3 year old child, according to the National Health and Nutrition Examination Survey database [McDowell et al, 2008]) to 35 kg (above which pediatric subjects could be dosed with the tablet formulation). Subjects with a body weight < 11 kg will not be included in the study.

# IS AMENDED TO:

For dosing with oral suspension, the weight range to be covered is from 13<sup>11</sup> kg (the approximate body weight of a 53-year old child, according to the National Health and Nutrition Examination Survey database [McDowell et al, 2008]) to 35 kg (above which pediatric subjects could be dosed with the tablet formulation). Subjects with a body weight < 13+1 kg will not be included in the study.

# 1 Protocol Summary and 5 Study Population

5.1 Inclusion Criterion #9

WAS:

11 Feb 2021 Astellas 

EudraCT number 2016-001767-37


Female subject is not pregnant (see [Appendix 12.3 Contraception Requirements]) and at least 1 of the following conditions apply:

- c. Not a woman of childbearing potential (WOCBP) (see [Appendix 12.3 Contraception Requirements]).
- d. WOCBP who agrees to follow the contraceptive guidance (see [Appendix 12.3 Contraception Requirements]) from the time of informed consent/assent through at least 30 days after final IP administration.

# IS AMENDED TO:

Female subject is not pregnant (see [Appendix 12.3 Contraception Requirements]) and at least 1 of the following conditions apply:

- a. Not a womanfemale of childbearing potential (WOCBP) (see [Appendix 12.3 Contraception Requirements]).
- b. **Female of childbearing potential** WOCBP who agrees to follow the contraceptive guidance (see [Appendix 12.3 Contraception Requirements]) from the time of informed consent/assent through at least 30 days after final IP administration.

# 1 Protocol Summary and 5 Study Population

5.1 Inclusion Criterion #13

WAS:

Male subject must not donate sperm during the treatment period and for 30 days after final IP administration.

#### IS AMENDED TO:

Male subject must **agree** not **to** donate sperm during the treatment period and for 30 days after final IP administration.

# 1 Protocol Summary and 5 Study Population

5.1 Exclusion Criterion #19

WAS:

Subject is using or has used prohibited prior and/or concomitant medication(s) [Appendix 12.6 List of Excluded Concomitant Medications].

#### IS AMENDED TO:

Subject is using or has used prohibited prior and/or concomitant medication(s) [Appendix 12.6 List of Excluded Concomitant Medications] **that cannot be discontinued**.

# 1 Protocol Summary and 6 Investigational Product(s) and Other Study Treatment(s)

1.1 Synopsis, 6.1.1 Investigational Product(s)

WAS:

For detailed information on mirabegron prolonged release tablets and mirabegron granules for oral suspension, please refer to the current locally-available product information for mirabegron.

EudraCT number 2016-001767-37


| Table 7 Body Weight-based Doses for Tablets or Suspension | | | | |
|---|---|---|---|---|
| | | Body Weight Range†<br>(kg) | Oral Suspension Volume‡ (mL) | Tablet Dose (mg) |
| | | 11 to < 22 | 3 | - |
| PED25 | 22 to < 35 | 4 | - | |
| | ≥ 35‡ | 6 | 25 | |
| | | 11 to < 22 | 6 | - |
| PED50 | ED50 22 to < 35 | | 8 | - |
| | | ≥ 35‡ | 11 | 50 |

# IS AMENDED TO:

For detailed information on mirabegron prolonged release tablets and mirabegron granules for oral suspension, please refer to the current locally-available product information for mirabegron. For detailed information on mirabegron granules for oral suspension, please refer to the Investigator's Brochure and Investigational Medicinal Product Dossier.

Table 7 Body Weight-based Doses for Tablets or Suspension

| | Body Weight Range†<br>(kg) | Oral Suspension Volume‡ (mL) | Tablet Dose (mg) |
|---|---|---|---|
| | <b>13</b> <del>11</del> to < 22 | 3 | - |
| PED25 | 22 to < 35 | 4 | - |
| | ≥ 35‡ | 6 | 25 |
| | <b>13</b> <del>11</del> to < 22 | 6 | - |
| PED50 | PED50 22 to < 35 | | - |
| | ≥ 35‡ | 11 | 50 |

# 6 Investigational Product(s) and Other Study Treatment(s)

6.1.2 Other Study Treatment(s)

# WAS:

Urotherapy is to be discussed and confirmed with the subject or parent(s)/legal guardian(s) during each TC to ensure compliance.

# IS AMENDED TO:

Urotherapy is to be discussed and confirmed with the subject or parent(s)/legal guardian(s) during each **visit (or** TC) to ensure compliance.

# 6 Investigational Product(s) and Other Study Treatment(s)

6.4.1 Investigational Product(s)

#### WAS:

Subject compliance with IP and other study treatment(s) will be assessed at each visit. Compliance will be assessed by counting returned IP at each clinic visit.

11 Feb 2021 Astellas 

Sponsor: APGD ISN/Protocol: 178-CL-204 EudraCT number 2016-001767-37


#### IS AMENDED TO:

Subject compliance with IP and other study treatment(s) will be assessed at each visit. Compliance will be assessed by counting **or weighing** returned IP at each clinic visit.

# 6 Investigational Product(s) and Other Study Treatment(s)

6.4.2 Other Study Treatment(s)

#### ADDED:

Specific interventions include various forms of pelvic floor training (relaxation, contraction), behavioral modification, electrical stimulation, catherization and biofeedback (use of objective measures, e.g., uroflow or surface EMG to show children how far they relax their pelvic floor during voiding). Urotherapy can also include elements of cognitive behavioral therapy [Nevéus et al, 2006].

# 1 Protocol Summary and 6 Investigational Product(s) and Other Study Treatment(s)

1.1 Synopsis, Treatment Discontinuation Criteria, 6.5 Previous and Concomitant Treatment (Medication and Nonmedication Therapy)

WAS:

Subjects are not allowed to use ongoing treatment with any of the following prohibited medications after the start of the washout:

• Any medication, other than the IP, used for the treatment of OAB

#### IS AMENDED TO:

Subjects are not allowed to use ongoing treatment with any of the following prohibited medications after the start of the washout:

- Any medication, other than the IP, used for the treatment of OAB (including tricyclic antidepressants, 1st generation H1 antagonists and alpha blockers)
- Any medications known to prolong the QT interval
- Any medication that is a moderate or strong cytochrome CYP3A4/5 or P-gp inhibitor or inducers including natural and herbal remedies

These treatments are prohibited from being started after the start of the washout period. All other concomitant treatment use will be reported.

The use of previous and concomitant treatment within 30 days prior to signing the informed consent and throughout the study will be documented on the appropriate eCRF.

# 7 Study Procedures and Assessments

#### ADDED:

Refer to the Alternate Schedule of Assessments [Table 12] in [Appendix 12.13 Clinical Study Continuity] for acceptable alternate methods to assess safety and efficacy

11 Feb 2021 Astellas 


ISN/Protocol: 178-CL-204

parameters in the event the study is interrupted due to a crisis (e.g., natural disaster, pandemic).

# 7 Study Procedures and Assessments

7.1.1 Bladder Electronic-Diary

#### WAS:

The e-diary data is reviewed by the investigator prior to the start of visit 2 and discussed and confirmed with the subject or the subject's parent(s)/caregiver(s) during the (telephone) visit

# IS AMENDED TO:

The e-diary data is reviewed by the investigator **or designee** prior to the start of visit 2 and discussed and confirmed with the subject or the subject's parent(s)/caregiver(s) during the (telephone) visit 2.

# 7 Study Procedures and Assessments

7.2.2 Laboratory Assessments

# WAS:

Pregnancy test in female subjects will be performed in serum at screening and visit 8/week 14 (EoS).

Additional hematology, biochemistry and urinalysis (urinalysis dipstick) tests will be performed at visit 3/week 0 (baseline), visit 5/week 4 and visit 8/week 14 (EoS) only if an AE related to hematology, biochemistry or urinalysis parameters occurred since the previous visit or at the discretion of the investigator.

# IS AMENDED TO:

A urine Ppregnancy test in female subjects of childbearing potential will be performed in serum at screening and visit 8/week 14 (EoS) all on-site visits.

Scheduled blood sampling will only be performed at screening (visit 1), week 4 (visit 5) and EoT (visit 7) to keep the burden to subjects at a minimum. Additional hematology, biochemistry and urinalysis (urinalysis dipstick) tests will be performed at visit 3/week 0 (baseline), visit 5/week 4 and visit 8/week 14 (EoS) only if an AE related to hematology, biochemistry or urinalysis parameters occurred since the previous visit or at the discretion of the investigator.

Refer to the Alternate Schedule of Assessments [Table 12] for acceptable alternate methods to assess safety and efficacy parameters in the event the study is interrupted due to a crisis (e.g., natural disaster, pandemic).

# 7 Study Procedures and Assessments

7.2.3.1 Clinic-measurement of Vital Signs and Electrocardiograms

WAS:

11 Feb 2021 Astellas 


Body temperature will be measured with an ear thermometer. Clinic measurements will be used to assess eligibility.

ISN/Protocol: 178-CL-204

#### IS AMENDED TO:

Body temperature will be measured with an ear thermometer **as per standard of care**. Clinic measurements will be used to assess eligibility.

# 7 Study Procedures and Assessments

7.2.4 Physical Examination

# ADDED:

In this study, the physical examination will be done to evaluate general physical condition and encompasses standard, full physical examinations to assess general appearance, skin, eyes, ears, nose, throat, neck, cardiovascular, chest and lungs, abdomen, musculoskeletal, neurologic status, mental status and lymphatic systems.

# 7 Study Procedures and Assessments

7.4 Pharmacokinetics

# WAS:

Blood samples for the analysis of ED178/mirabegron and ethanol in plasma will be collected as indicated in the Schedule of Assessments [Table 1] for the evaluation of pharmacokinetics.

# IS AMENDED TO:

Blood samples for the analysis of ED178/mirabegron and ethanol in plasma will be collected as indicated in the Schedule of Assessments [Table 1] for the evaluation of pharmacokinetics.

The pharmacokinetic parameters that will be calculated as part of the secondary pharmacokinetic endpoint are steady-state  $C_{max}$ ,  $AUC_{tau}$ ,  $C_{trough}$ ,  $T_{max}$ , CL/F and Vz/F. Additional parameters may be calculated based on the population pharmacokinetic model used.

# 7 Study Procedures and Assessments

7.6 Electronic Clinical Outcome Assessment

# WAS:

For this study, it has been decided that there are justifiable scientific reasons (i.e., recall bias) to limit subject reported changes to changes reported by the subject to the site within 1 business day of its entry, as changes outside of this window could potentially impact the data integrity of the study. The data that will be under this rule are: all subject/guardian/parent entered, primary and secondary endpoints data. However, the site/investigator can remove/inactivate any data that they determine to be in error at any time.

Subject bladder diaries, questionnaires and other data completed by the subject or the


subject's parent(s)/legal guardian(s) will be entered on an electronic device (e-diary). The information on the electronic device will be automatically uploaded to a central website. The investigator or site designee should review the diaries and questionnaire data on the website for correct completion before each planned visit of the subject (on site visit or TC) and discuss the results or retrain the subject and/or subject's parent(s)/legal guardian(s) if applicable. In case clinically relevant adverse changes are noticed during review of the e diary, these will be recorded as an AE [Appendix 12.4.1 Definition of Adverse Events]. The bladder e-diary, questionnaire results and other data collected in the e-diary will be transferred electronically to sponsor or designee at predefined intervals during the study. The vendor will provide sponsor or designee with a complete and clean copy of the data.

ISN/Protocol: 178-CL-204

# IS AMENDED TO:

For this study, it has been decided that there are justifiable scientific reasons (i.e., recall bias) to limit subject reported changes to changes reported by the subject to the site within 1 business day of its entry, as changes outside of this window could potentially impact the data integrity of the study. The data that will be under this rule are: all subject/guardian/parent-entered, primary and secondary endpoints data. However, the site/investigator can remove/inactivate any data that they determine to be in error at any time with source documentation to support the change including subject confirmation. Data will never be deleted from the electronic database by the electronic clinical outcome assessment (eCOA) service provider, but will be removed logically as per investigator's request and approval. All data changes are audit trailed showing the original entries alongside all changes including who requested the change, why it was requested, who made the change and when it was made. Audit trails are reviewed by the sponsor/clinical research organization (CRO) to ensure adherence to the protocol and appropriate source exists at site to substantiate the change.

Subject bladder diaries, questionnaires and other data **will be** completed by the subject or the subject's parent(s)/legal guardian(s)/**caregiver(s)** will be entered on an electronic device (ediary). The information on the electronic device will be automatically uploaded to a central website. The investigator or site designee should review the diaries and questionnaire data on the website for correctto ensure completion and protocol compliance before each planned visit of the subject (on site visit or TC) and discuss the results or retrain the subject and/or subject's parent(s)/legal guardian(s)/**caregiver(s)**, if applicable. In case clinically relevant adverse changes are noticed during review of the e diary, these will be recorded as an AE [Appendix 12.4.1 Definition of Adverse Events].

The bladder e-diary, questionnaire results and other data collected in the e-diary will be transferred electronically to the sponsor or designee at predefined intervals during the study. The vendor will provide the sponsor or designee with a complete and clean copy of the study data. The ownership of this data is with the investigator and subsequently any changes requested to these subject-reported or nonsubject reported data will be made using the vendor's established process (e.g., a data clarification form to the vendor). The requested change must be supported by documented evidence at study site.

Sponsor: APGD

EudraCT number 2016-001767-37


# 7 Study Procedures and Assessments

7.8 Total Amount of Blood (Table 8)

#### WAS:

| Sample Type | Number of Samples | Sample Volume (mL) | Total Volume (mL) |
|---|---|---|---|
| Pharmacokinetics | 2 | 5.0 | 10.0 |
| Clinical Laboratory Tests† | 2 | 4.5§‡ | 9.0 |
| Biochemistry/hematology | 2 | 4.38‡ | 9.0 |
| Total | | | 19.0 |

ISN/Protocol: 178-CL-204

- † Additional hematology and biochemistry tests of approximately 4.5 mL total will be performed at visit 3/week 0 (baseline), visit 5/week 4 and visit 8/week 14 (EoS) only if an adverse event related to hematology or biochemistry parameters occurred since the previous visit or at the discretion of the investigator.
- ‡ Includes pregnancy test in female subjects who experienced menarche (if blood is drawn); no additional blood is required. Volume does not take any unscheduled visits or repeat tests into account (e.g., follow up of adverse events).

#### IS AMENDED TO:

| Sample Type | Number of Samples | Sample Volume (mL) | Total Volume (mL) |
|---|---|---|---|
| Pharmacokinetics | 2 | 5.0 | 10.0 |
| Clinical Laboratory Tests† | <del>32</del> | 4.5 <del>§</del> ‡ | 13.59.0 |
| Biochemistry/hematology | <del>32</del> | 4.284 | |
| Total | | | <b>23.5</b> <del>19.0</del> |

- † Additional hematology and biochemistry tests of approximately 4.5 mL total will be performed at visit 3/week 0 (baseline), visit 5/wee 4 and visit 8/week 14 (EoS) only if an adverse event related to hematology or biochemistry parameters occurred since the previous visit or at the discretion of the investigator.
- ‡ Includes pregnancy test in female subjects who experienced menarche (if blood is drawn); no additional blood is required. Volume does not take any unscheduled visits or repeat tests into account (e.g., follow up of adverse events).

#### 8 Discontinuation

8.1 Discontinuation of Individual Subject(s) From Study Treatment(s)

#### ADDED:

A discontinuation from treatment is defined as a subject who is randomized and for whom study treatment is permanently discontinued for any reason.

The subject is free to withdraw from the study treatment and/or study for any reason and at any time without giving reason for doing so and without penalty or prejudice. The investigator is also free to discontinue the participant from study treatment or to terminate a subject's involvement in the study at any time if the subject's clinical condition warrants it.

• • •

The reason for discontinuation from study treatment must be documented in the subject's medical records.

Female subject becomes pregnant.

EudraCT number 2016-001767-37


- Prolongation of QT > QTcF > 440 msec and/or QT interval prolongation > 30 msec versus baseline.
- Subject with (systolic blood pressure ≥ 160 mm Hg or diastolic blood pressure ≥ 100 mmHg.

# 9 Statistical Methodology

9.1 Sample Size

ADDED:

These assumptions, together with levels for Type-1 error and power were agreed upon with Pediatric Committee in the current Pediatric Investigation Plan

# 9 Statistical Methodology

9.4.1.3 Subgroup Analysis

WAS:

For the primary efficacy endpoint, descriptive statistics (n, mean, 95% confidence interval around the mean, SD, minimum, median, maximum) will be calculated for mean change from baseline at each visit by sex, race, ethnicity, geographical region, formulation (tablets vs. oral suspension) and prior OAB treatment, with and without LOCF.

# IS AMENDED TO:

For the primary efficacy endpoint, descriptive statistics (n, mean, 95% confidence interval around the mean, SD, minimum, median, maximum) will be calculated for mean change from baseline at each visit by sex, race, ethnicity, geographical region, formulation (tablets vs. oral suspension), and prior OAB treatment, with and without LOCF and symptomatic UTI.

# 9 Statistical Methodology

9.4.3 Analysis of Exploratory Endpoints

ADDED:

Mean number of micturitions per 24 hours

# 9 Statistical Methodology

9.5.2 Laboratory Assessments

#### ADDED:

In cases where laboratory evaluations are conducted locally, the values obtained will be adjusted to values obtained by the central laboratory. Details will be described in the SAP.

Sponsor: APGD
EudraCT number 2016-001767-37

ISN/Protocol: 178-CL-204

# 9 Statistical Methodology

9.5.5 Electrocardiogram

ADDED:

ECGs will be recorded prior to blood draw.

# 9 Statistical Methodology

9.6.1 Estimation of Pharmacokinetic Parameters

WAS:

The plasma concentrations will be analyzed with nonlinear mixed effects modeling (population pharmacokinetics) using Non-Linear Mixed Effects Modeling software (version 7.3 or higher, ICON Development Solutions, Ellicott City, MD, US) to estimate the pharmacokinetic parameters. Results will be reported separately.

# IS AMENDED TO:

The plasma concentrations will be analyzed with nonlinear mixed effects modeling (population pharmacokinetics) using Non-Linear Mixed Effects Modeling (NONMEM) software (version 7.3 or higher, ICON Development Solutions, Ellicott City, MD, US) to estimate the pharmacokinetic parameters. Results will be reported separately.

# 10 Operational Considerations

10.1 Data Collection

#### DELETED.

The investigator or site designee is responsible to ensure that all data in the electronic case report forms and queries are accurate and complete and that all entries are verifiable with the source. These documents should be appropriately maintained by the study site.

The e diary and questionnaire data will be transferred electronically to the sponsor or designee at predefined intervals during the study. The vendor will provide the investigator with a complete and clean copy of the study site's data and will provide the sponsor or designee with a complete and clean copy of the study data. The ownership of this data is with the investigator and subsequently any changes requested to these subject reported data will be made using a data clarification form to the vendor. The requested change must be supported by documented evidence at study site.

| 10 Operational Considerations |
|-------------------------------|
| ADDED: |


# 10.4.2 Independent Data Analysis Center

An IDAC for this study will serve the 2 purposes: (1) to generate periodic safety overviews for the DSMB and (2) to calculate the futility analysis. The statistical member of the DSMB may also serve as the IDAC statistician, as described in the DSMB charter. A SAP describing the details of the periodic safety review or outputs will be developed with input from the DSMB members.

ISN/Protocol: 178-CL-204

#### 11 References

WAS:

Investigator's Brochure Mirabegron (ED178), Astellas.

IS AMENDED TO

Investigator's Brochure Mirabegron (YMED178), Astellas.

# 12 Appendices

12.1.6 Source Documents

#### ADDED:

- 3. The investigator must maintain accurate documentation (source data) that supports the information entered in the CRF.
- 5. Study monitors will perform ongoing source data review to confirm that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP and all applicable regulatory requirements.

# 12 Appendices

12.2.1 Study Monitoring

#### WAS:

The sponsor is responsible for monitoring the study to ensure that the rights, safety and well-being of subjects are protected, the study is properly conducted in adherence to the current protocol and GCP and the study data reported by the investigator/subinvestigator(s) are accurate, complete and verifiable with the source.

# IS AMENDED TO

The sponsor is responsible for monitoring the study to ensure that the rights, safety and well-being of subjects are protected, the study is properly conducted in adherence to the current protocol and GCP and the study data reported by the investigator/subinvestigator(s) are accurate, complete and verifiable with the source.

11 Feb 2021 Astellas 


# 12 Appendices

# 12.3 Contraception Requirements

# WAS:

WOCBP who are eligible for participation in the study, including those who choose complete abstinence, must have pregnancy tests as specified in the Schedule of Assessments. Pregnancy test results must confirm that the subject is not pregnant.

ISN/Protocol: 178-CL-204

# WOMEN OF CHILDBEARING POTENTIAL DEFINITIONS AND METHODS OF CONTRACEPTION DEFINITIONS

A female is considered fertile (i.e., WOCBP) following menarche and until becoming postmenopausal unless permanently sterile.

Females in the following categories are not considered WOCBP

- Premenarchal
- Premenopausal with 1 of the following (i.e., permanently sterile):
  - Documented hysterectomy
  - Documented bilateral salpingectomy
  - Documented bilateral oophorectomy

Documentation of any of these categories can come from the study site personnel's review of the female subject's medical records, medical examination or medical history interview.

# CONTRACEPTION GUIDANCE FOR FEMALE SUBJECTS OF CHILDBEARING POTENTIAL

Female subjects of childbearing potential are eligible for participation in the study if they agree to use 1 of the highly effective methods of contraception listed below from the time of signing the ICF/assent and until the end of relevant systemic exposure, defined as 30 days after the final IP administration.<sup>a</sup>

Highly effective methods of contraception (failure rate of < 1% per year when used consistently and correctly)<sup>b</sup>:

- Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation
  - o Oral
  - Intravaginal
  - Transdermal
- Progestogen-only hormonal contraception associated with inhibition of ovulation
  - o Oral
  - o Injectable
  - Implantable
- Other combined (estrogen- and progesterone-containing) methods
  - Vaginal ring
  - Injectable
  - Implantable

11 Feb 2021 Astellas 

Sponsor: APGD ISN/Protocol: 178-CL-204 EudraCT number 2016-001767-37


- Intrauterine hormone-releasing system or intrauterine device
- Bilateral tubal occlusion
- Vasectomized partner
- A vasectomized partner is a highly effective contraception method provided that the
  partner is the sole male sexual partner of the WOCBP and the absence of sperm has been
  confirmed. If not, an additional highly effective method of contraception should be
  used.
- Sexual abstinence
- Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the test product. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the subject. It is not necessary to use any other method of contraception when complete abstinence is elected.

<sup>a</sup>Local laws and regulations may require use of alternative and/or additional contraception methods.

# CONTRACEPTION GUIDANCE FOR MALE SUBJECTS WITH PARTNER(S) OF CHILDBEARING POTENTIAL

Male subjects with female partners of childbearing potential are eligible for participation in the study if they agree to the following during treatment and until the end of relevant systemic exposure defined as 30 days after final drug administration.<sup>a</sup>

- Inform any and all partner(s) of their participation in a clinical drug study and the need to comply with contraception instructions as directed by the investigator
- Use a condom
- Female partners of male subjects who have not undergone a vasectomy with the absence of sperm confirmed or a bilateral orchiectomy should consider use of effective methods of contraception

<sup>a</sup>Local laws and regulations may require use of alternative and/or additional contraception methods.

#### IS AMENDED TO:

# Contraception for Pediatric Male Subjects of Reproductive Potential

Male children/adolescents in the following categories are not considered of reproductive potential:

- 1. Tanner stage 1 development
- 2. Documented surgically sterile

Documentation from the site personnel's review of the male subject's medical records, medical exam and medical history interview is necessary.

Contraception guidance for male children/adolescents of reproductive potential:

• Male children/adolescents of reproductive potential (Tanner Stage 2 and above)

<sup>&</sup>lt;sup>b</sup>Typical use failure rates may differ from those when used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for subjects participating in clinical studies.

Sponsor: APGD ISN/Protocol: 178-CL-204 EudraCT number 2016-001767-37


receiving non-genotoxic agents should use a condom during treatment and for 3 weeks + 5  $\times$  half-life of drug after last dose.

- Male children/adolescents of reproductive potential receiving genotoxic agents should use a condom during treatment and for 90 days + 5 × half-life of drug after last dose.
- Male participants should inform their female partners that they are participating in a clinical trial and effective methods of contraception should be used.
- Female partners of male subjects who have not undergone bilateral orchiectomy should consider use of highly effective methods of contraception until the end of relevant systemic exposure, as defined above.

# **Contraception for Pediatric Female Subjects of Childbearing Potential**

Female children/adolescents in the following categories are not considered of childbearing potential:

- 1. Pre-menarchal
- 2. Documented surgically sterile (hysterectomy, bilateral salpingectomy, bilateral oophorectomy)

Documentation from the site personnel's review of the female subject's medical records, medical exam and medical history interview is necessary.

Contraception guidance for female children/adolescents of childbearing potential:

- Female children/adolescents of childbearing potential receiving non-genotoxic agents should use highly effective contraception during treatment and for 30 days after last dose.
- Female children/adolescents of childbearing potential receiving genotoxic agents should use contraception during treatment and for 180 days + 5  $\times$  half-life of drug after last dose.
- Pregnancy testing for female children/adolescents of childbearing potential
  - o At all on-site visits and 30 days after end of relevant systemic exposure

One of the highly effective methods of contraception listed below is required at the time of informed consent and until the end of relevant systemic exposure as defined above.

# **Highly Effective Birth Control Methods-failure rate < 1%/year**

- 1. Combined estrogen and progestogen containing hormonal contraception
  - a. Oral
  - b. Intravaginal
  - c. Transdermal-Patch
  - d. Injectable-Cyclofem, Mesigyna
  - e. Intrauterine device
  - f. Intrauterine hormone-releasing system
- 2. Progestogen-only hormonal contraception
  - d. Oral
Sponsor: APGD EudraCT number 2016-001767-37


- e. Injectable-DMPA-IM or -SC
- f. Implantable-Norplant
- 3. Bilateral tubal occlusion
- 4. Vasectomized male partner
- 5. True abstinence\*

\*True abstinence: When this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study drug. It is not necessary to use any other method of contraception when complete abstinence is elected.

ISN/Protocol: 178-CL-204

Birth control methods considered unacceptable:

- 1. Periodic abstinence (calendar, symptothermal, post-ovulation methods)
- 2. Withdrawal (coitus interruptus)
- 3. Spermicides only
- 4. Lactational amenorrhea

WOCBP who are eligible for participation in the study, including those who choose complete abstinence, must have pregnancy tests as specified in the Schedule of Assessments. Pregnancy test results must confirm that the subject is not pregnant.

WOMEN OF CHILDBEARING POTENTIAL DEFINITIONS AND METHODS OF CONTRACEPTION DEFINITIONS

A female is considered fertile (i.e., WOCBP) following menarche and until becoming postmenopausal unless permanently sterile.

Females in the following categories are not considered WOCBP

- Premenarchal
- Premenopausal with 1 of the following (i.e., permanently sterile):
  - Documented hysterectomy
  - Documented bilateral salpingectomy
  - Documented bilateral oophorectomy

Documentation of any of these categories can come from the study site personnel's review of the female subject's medical records, medical examination or medical history interview.

CONTRACEPTION GUIDANCE FOR FEMALE SUBJECTS OF CHILDBEARING POTENTIAL

Female subjects of childbearing potential are eligible for participation in the study if they agree to use 1 of the highly effective methods of contraception listed below from the time of signing the ICF/assent and until the end of relevant systemic exposure, defined as 30 days

Sponsor: APGD
EudraCT number 2016-001767-37

ISN/Protocol: 178-CL-204

#### after the final IP administration.<sup>a</sup>

Highly effective methods of contraception (failure rate of < 1% per year when used consistently and correctly)<sup>b</sup>:

- Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation
  - → Oral
  - Intravaginal
  - Transdermal
- Progestogen only hormonal contraception associated with inhibition of ovulation
  - Oral
  - Injectable
  - → Implantable
- Other combined (estrogen and progesterone containing) methods
  - Vaginal ring
  - Injectable
  - Implantable
  - Intrauterine hormone releasing system or intrauterine device
- Bilateral tubal occlusion
- Vasectomized partner
- A vasectomized partner is a highly effective contraception method provided that the
  partner is the sole male sexual partner of the WOCBP and the absence of sperm has been
  confirmed. If not, an additional highly effective method of contraception should be
  used.
- Sexual abstinence
- Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the test product. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the subject. It is not necessary to use any other method of contraception when complete abstinence is elected.

# CONTRACEPTION GUIDANCE FOR MALE SUBJECTS WITH PARTNER(S) OF CHILDBEARING POTENTIAL

Male subjects with female partners of childbearing potential are eligible for participation in the study if they agree to the following during treatment and until the end of relevant systemic exposure defined as 30 days after final drug administration.<sup>a</sup>

- Inform any and all partner(s) of their participation in a clinical drug study and the need to comply with contraception instructions as directed by the investigator
- Use a condom
- Female partners of male subjects who have not undergone a vasectomy with the absence

<sup>&</sup>lt;sup>a</sup>Local laws and regulations may require use of alternative and/or additional contraception methods.

<sup>&</sup>lt;sup>b</sup>Typical use failure rates may differ from those when used consistently and correctly. Use should be consistent with local regulations regarding the use of contraceptive methods for subjects participating in clinical studies.


D ISN/Protocol: 178-CL-204

of sperm confirmed or a bilateral orchicetomy should consider use of effective methods of contraception

\*Local laws and regulations may require use of alternative and/or additional contraception methods.

#### 12 Appendices

#### 12.4.1.1 Abnormal Laboratory Findings

#### WAS:

Any abnormal laboratory test result (e.g., hematology, biochemistry or urinalysis dipstick) or other safety assessment (e.g., vital signs, physical examination, ECGs or radiographic scans), including those that worsen from baseline, that is considered to be clinically significant in the medical and scientific judgment of the investigator and not related to underlying disease, is to be reported as an (S)AE.

Any clinically significant abnormal laboratory finding or other abnormal safety assessment, which is associated with the underlying disease, does not require reporting as an (S)AE, unless judged by the investigator to be more severe than expected for the subject's condition.

#### IS AMENDED TO:

Any abnormal laboratory test result (e.g., hematology, biochemistry or urinalysis dipstick) or other safety assessment (e.g., vital signs, physical examination, ECGs or radiographic scans), including those that worsen from baseline, that is considered to be elinically significant in the medical and scientific judgment of the investigator and not related to underlying disease, is should be considered to be reported as an (S)AE.

Any clinically significant abnormal laboratory finding or other abnormal safety assessment, which is associated with the underlying disease or with concomitant medication will not be considered an AE, does not require reporting as an (S)AE, unless judged by the investigator to be more severe than expected for the subject's condition or not associated with the known side effects of the concomitant medication. Additionally, minor laboratory deviations or fluctuations outside of normal ranges of preexisting disease(s) or condition(s) present or detected at the start of the study that do not worsen and/or that are not reproducible with re-testing will not to be considered an AE.

#### 12 Appendices

#### 12.6 List of Excluded Concomitant Medications

#### WAS:

| Anticholinergics/antimuscarinics | Tricyclic/heterocyclic antidepressants | 1st generation H1-antagonists† |
|---|---|---|
| Darifenacin | Alimemazine / Trimipramine | Tripelennamine |
| Dicyclomine/Dicycloverine | Amitriptyline | Dimenhydrinate |
| Fesoterodine | Amoxapine | Clemastine |
| Flavoxate | Clomipramine | Bromazine |
| Isopropamide | Desipramine | Orphenadrine |

Sponsor: APGD EudraCT number 2016-001767-37


| Oxybutynin | Dosulepin/ Dothiepin | Doxylamine |
|---|---|---|
| Oxyphencyclimine | Doxepine | Carbinoxamine |
| Propantheline | Imipramine | Diphenhydramine |
| Propiverine | Lofepramine | Cyclizine |
| Tolterodine | Maprotiline | Chlorcyclizine |
| Trospium | Mianserin | Hydroxyzine |
| Solifenacin | Mirtazapine | Meclizine |
| | Nortriptyline | |
| | Protriptyline | |
| pha-blockers | P2D6 with narrow therapeutic index | Sensitive P-gp substrates |
| Tamsulosin | Thioridazine | Digoxin |
| Alfuzosin | Flecainide | Dabigatran |
| Doxazosin | Propafenone | |
| Terazosin | Imipramine | |
| Silodosin | Desipramine | |
| Strong CYP3A4 inhibitors | Other | |
| Itraconazole | Mirabegron (except for study drug) | |
| Ketoconazole | Botulinum toxin | |
| Ritonavir | Opioids | |
| Clarthromycin | | |

### IS AMENDED TO

| Anticholinergics/antimuscarinics | Tricyclic/heterocyclic antidepressants | 1st generation H1-antagonists† |
|---|---|---|
| Darifenacin | Alimemazine /Trimipramine | Tripelennamine |
| Dicyclomine/Dicycloverine | Amitriptyline | Dimenhydrinate |
| Fesoterodine | Amoxapine | Clemastine |
| Flavoxate | Clomipramine | Bromazine |
| Isopropamide | Desipramine | Orphenadrine |
| Oxybutynin | Dosulepin/Dothiepin | Doxylamine |
| Oxyphencyclimine | Doxepine | Carbinoxamine |
| Propantheline | Imipramine | Diphenhydramine |
| Propiverine | Lofepramine | Cyclizine |
| Tolterodine | Maprotiline | Chlorcyclizine |
| Trospium | Mianserin | Hydroxyzine |
| Solifenacin | Mirtazapine | Meclizine |
| | Nortriptyline | |
| | Protriptyline | |
| Alpha-blockers | CYP2D6 with narrow therapeutic index | Sensitive P-gp substrates |
| Tamsulosin | Thioridazine | Digoxin |
| Alfuzosin | Flecainide | Dabigatran |
| Doxazosin | Propafenone | |

Sponsor: APGD EudraCT number 2016-001767-37


| Terazosin | Imipramine | |
|---|---|---|
| Silodosin | Desipramine | |
| Moderate CYP3A4 inhibitors | Strong CYP3A4 inhibitors Moderate CYP3A4 inducers | |
| Fluconazole | Itraconazole Cenobamate | |
| Ciprofloxacin | Ketoconazole Tipranavir | |
| Erythromycin | Ritonavir | Ritonavir |
| Clotrimazole | Clarthromycin | Thioridazine |
| Fluvoxamine | Voriconazole | Rifabutin |
| Verapamil | Posaconazole | Nafcillin |
| Dronedarone | Troleandomycin | Lopinavir |
| Cimetidine | Telithromycin | Modafinil |
| Grapefruit Juice | Tentinomythi | Phenobarbital |
| Strong CYP3A4 inducers | P-gp inhibitors‡ | P-gp Inducers‡ |
| Rifampin | | |
| Rifapentine | Amiodarone Rifampin | |
| Phenytoin | Carvedilol Carbamazepine | |
| | Clarithromycin Dexamethasone | |
| Carbamazepine | Dronedarone | Phenobarbital |
| Ct T 1 1 | | |
| St. John's wort | Itraconazole | Phenytoin |
| St. John's wort | Lopinavir, Ritonavir | Rifampicin |
| St. John's wort | Lopinavir, Ritonavir<br>Quinidine | Rifampicin<br>St. John's wort |
| | Lopinavir, Ritonavir Quinidine Verapamil | Rifampicin |
| QT prolongating medicationsStrong CYP3A4 inhibitors | Lopinavir, Ritonavir<br>Quinidine | Rifampicin<br>St. John's wort |
| QT prolongating medicationsStrong CYP3A4 | Lopinavir, Ritonavir Quinidine Verapamil | Rifampicin<br>St. John's wort<br>Trazodone |
| QT prolongating<br>medicationsStrong CYP3A4<br>inhibitors | Lopinavir, Ritonavir Quinidine Verapamil Other | Rifampicin<br>St. John's wort<br>Trazodone |
| QT prolongating medicationsStrong CYP3A4 inhibitors AmiodaroneIntraconazole | Lopinavir, Ritonavir Quinidine Verapamil Other Mirabegron (except for study dre | Rifampicin<br>St. John's wort<br>Trazodone |
| QT prolongating medicationsStrong CYP3A4 inhibitors AmiodaroneIntraconazole SotalolKetoconazole | Lopinavir, Ritonavir Quinidine Verapamil Other Mirabegron (except for study dru Botulinum toxin | Rifampicin<br>St. John's wort<br>Trazodone |
| QT prolongating medicationsStrong CYP3A4 inhibitors AmiodaroneIntraconazole SotalolKetoconazole QuinidineRitonavir Levofloxacin, | Lopinavir, Ritonavir Quinidine Verapamil Other Mirabegron (except for study dru Botulinum toxin | Rifampicin<br>St. John's wort<br>Trazodone |
| QT prolongating medicationsStrong CYP3A4 inhibitors AmiodaroneIntraconazole SotalolKetoconazole QuinidineRitonavir Levofloxacin, CiprofloxacinClarthromycin | Lopinavir, Ritonavir Quinidine Verapamil Other Mirabegron (except for study dru Botulinum toxin | Rifampicin<br>St. John's wort<br>Trazodone |
| QT prolongating medicationsStrong CYP3A4 inhibitors AmiodaroneIntraconazole SotalolKetoconazole QuinidineRitonavir Levofloxacin, CiprofloxacinClarthromycin Clarithromycin, Erythromycin | Lopinavir, Ritonavir Quinidine Verapamil Other Mirabegron (except for study dru Botulinum toxin | Rifampicin<br>St. John's wort<br>Trazodone |
| QT prolongating medicationsStrong CYP3A4 inhibitors AmiodaroneIntraconazole SotalolKetoconazole QuinidineRitonavir Levofloxacin, CiprofloxacinClarthromycin Clarithromycin, Erythromycin Ketoconazole, Itraconazole | Lopinavir, Ritonavir Quinidine Verapamil Other Mirabegron (except for study dru Botulinum toxin | Rifampicin<br>St. John's wort<br>Trazodone |
| QT prolongating medicationsStrong CYP3A4 inhibitors AmiodaroneIntraconazole SotalolKetoconazole QuinidineRitonavir Levofloxacin, CiprofloxacinClarthromycin Clarithromycin, Erythromycin Ketoconazole, Itraconazole Amitriptyline, Fluoxetine | Lopinavir, Ritonavir Quinidine Verapamil Other Mirabegron (except for study dru Botulinum toxin | Rifampicin<br>St. John's wort<br>Trazodone |
| QT prolongating medicationsStrong CYP3A4 inhibitors AmiodaroneIntraconazole SotalolKetoconazole QuinidineRitonavir Levofloxacin, CiprofloxacinClarthromycin Clarithromycin, Erythromycin Ketoconazole, Itraconazole Amitriptyline, Fluoxetine Haloperidol, Droperidol | Lopinavir, Ritonavir Quinidine Verapamil Other Mirabegron (except for study dru Botulinum toxin | Rifampicin<br>St. John's wort<br>Trazodone |

# 12 Appendices

ADDED:

# 12.13 Clinical Study Continuity

#### INTRODUCTION

Sponsor: APGD


EudraCT number 2016-001767-37

The purpose of this appendix is to provide acceptable alternate methods to assess safety and efficacy parameters, as appropriate, in the event the clinical study is interrupted at the country, state, site or participant level during any crisis (e.g., natural disaster, pandemic).

ISN/Protocol: 178-CL-204

#### **BENEFIT-RISK RATIONALE**

Maintaining the safety of clinical study participants and delivering continuity of care in the clinical study setting is paramount during any crisis. The site is expected to follow the protocol and associated Schedule of Assessments [Table 1] unless the site principal investigator discusses the need with the Astellas medical monitor to implement the alternate measures.

The approach outlined within this appendix defines which assessments are required to maintain a favorable benefit/risk to the participant, to maintain overall study integrity and to provide acceptable alternate methods to complete the study required assessments and procedures if study activities are unable to be performed as described in [Section 7 Study Procedures and Assessments] due to a crisis.

#### INFORMED CONSENT

Participants who need to follow any or all of the alternate measures outlined in this Appendix will be required to provide informed consent, which explicitly informs them of the nature of and rationale for these changes, and gain their agreement to continue participation in the study prior to the implementation of any of these changes. In the event the urgency of implementing the alternate measures does not allow for the participant to provide written consent prior to implementation, the principal investigator or designee will obtain oral agreement from the subject followed by written documentation as soon as is feasible. A separate addendum to the study informed consent will be provided to document the participant's consent of the changes.

#### PARTICIPANT PROCEDURES ASSESSMENT

Sites with participants who are currently enrolled into this clinical study may consider implementing the alternate methods outlined below if one or more of the following conditions are met due to the crisis:

- Regional or local travel has been restricted, inclusive of mandatory shelter in place measures, which makes participant travel to/from the study site nearly impossible
- Site facilities have been closed for clinical study conduct
- Site has been restricted to treating patients with conditions outside of the scope of the study
- Site personnel have temporarily relocated the conduct of the study to a location that place a burden on the participant with respect to time and travel
- Participant(s) have temporarily relocated from the current study site to an alternate study site to avoid placing a burden on the participant with respect to travel
- Participant(s) have temporarily relocated from their home location and the new distances from the site would cause undue burden with respect to time and travel

Sponsor: APGD ISN/Protocol: 178-CL-204

EudraCT number 2016-001767-37


• Participant has risk factors for which traveling to the site poses an additional risk to the participant's health and safety

Adherence to the original protocol as reflected in the Schedule of Assessments [Table 1] is expected, where plausible, in the case of a crisis. The alternate measures as noted in [Table 12] below are only permissible in the event of a crisis, and after discussing the need with the Astellas medical monitor to implement the alternate measures. This is to allow for continuity of receiving IP and maintaining critical safety and efficacy assessments for patients participating in the study at a time of crisis.

If one or more of the alternate measures noted below is implemented for a participant, the site should document in the participant's source document the justification for implementing the alternate measure and the actual alternate measures that were implemented, along with the corresponding time point(s).

Sponsor: APGD ISN/Protocol: 178-CL-204

EudraCT number 2016-001767-37


## 12 Appendices

### ADDED:

# Table 12 Alternate Schedule of Assessments in Response to a Crisis

| | | D | ouble-blind | Placebo-con<br>(12 weeks) | trolled Peri | od | Follow-up Period (2 weeks) |
|---|---|---|---|---|---|---|---|
| | | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 |
| Critical Assessments | Alternate Approach(es) | Week 0 | Week 2 | Week 4 | Week 8 | Week 12 | Week 14 |
| | | Baseline | TCa | | TCa | (EoT) <sup>b</sup> | (EoS) <sup>b,c</sup> |
| | | Day -1 | Day 14 | <b>Day 28</b> | Day 56 | Day 84 | <b>Day 98</b> |
| | | | (± 3 days) | (± 3 days) | (± 3 days) | (± 3 days) | (+ 3 days) |
| Previous and Concomitant Medication | Remote/Virtual/Telemedicine Visits allowed. Please refer to protocol schedule of assessments. | X | X | X | X | X | X |
| Physical Examination | The exam can be done at a local clinic and the results submitted to PI. | | | X | | X | |
| Height and Body Weight | Can be obtained at a local clinic or at home | X | | | | X | |
| Dose Titration <sup>d</sup> | Courier service directly to subject. Titration to occur based on PI's evaluation via phone. For tablets: subject to take spare 25 mg tablets until 50 mg wallet is delivered via courier. | | | X | | | |
| Dispense IP <sup>e</sup> | Courier service directly to subject | X | | X | | | |
| Drug Accountability | Used product can be shipped back to site via courier. | X | | | | X | |
| Vital Signs <sup>f</sup> | Can be performed at a local clinic and results submitted to PI for evaluation OR | X | | X | | X | X |
| | Blood pressure and pulse collected via | | 1 | | | <u> </u> | |

Sponsor: APGD ISN/Protocol: 178-CL-204

EudraCT number 2016-001767-37


| | SBPM and temperature collected at home and reported to site (respiration rate missing). | | | | | | |
|---|---|---|---|---|---|---|---|
| SBPM <sup>g</sup> | Will be sent to subject's home address | X | X | X | X | X | |
| Routine 12-lead ECG <sup>f</sup> | ECG testing can be completed at local clinic. | X | | X | | X | |
| Clinical Laboratory Tests (Hematology and Biochemistry) <sup>h</sup> | Visit collection of samples at local facility acceptable if results can be made available to investigative site. | Xi | | X | | X | Xi |
| Clinical Laboratory Tests (Urinalysis) <sup>h</sup> | Visit collection of samples at local facility acceptable if results can be made available to investigative site. | Xi | | X | | X | Xi |
| Pregnancy Test <sup>i</sup> | Visit collection of samples at local facility acceptable if results can be made available to investigative site. | X | | X | | X | X |
| AEs | Remote/Virtual/Telemedicine Visits allowed. Please refer to protocol schedule of assessments. | X | X | X | X | X | X |
| Bladder e-diary | Will be sent to subject's home address | X | X | X | X | X | |
| Acceptability and Palatability Questionnaire | To be performed remotely via e-diary. | | | | | X | |
| Pharmacokinetics <sup>k</sup> | Astellas Medical Monitor to assess. Not allowed at an alternate clinical due to special sample handling. | | | X | | X | |

AE: adverse event; ECG: electrocardiogram; e-diary: electronic diary; EoS: end of study; EoT: end of treatment; IP: investigational product; OAB: overactive bladder; PED25: pediatric equivalent dose 25 mg; PED50: pediatric equivalent dose 50 mg; PI: principal investigator; SBPM: self blood pressure monitoring; TC: telephone call

- a. For the visits where a TC is indicated, there is no need for the subject to visit the clinic provided that the bladder e-diary data are reviewed by the investigator prior to the TC and discussed and confirmed with the subject or parent(s)/legal guardian(s) during the TC. Urotherapy is also to be discussed and confirmed with the subject or parent(s)/legal guardian(s) during each TC as indicated in Table 1.
- b. Subjects who withdraw early from the study after having received IP should complete both the EoT and EoS visits.
- c. The EoS visit (visit 8/week 14 [EoS]) should take place at least 14 days after the EoT visit (visit 7/week 12 [EoT]).
- d. Dose up-titration to PED50 to occur at visit 5/week 4 unless investigator determines OAB is adequately controlled. Dose down-titration from PED50 to PED25 can be done at any time for safety reasons.

Sponsor: APGD

EudraCT number 2016-001767-37


e. Daily IP administration will start on day 1 (i.e., the day after visit 3/week 0 [baseline]).

- f. Blood pressure, pulse, body temperature and ECGs will all be measured in single measurements. Subject to be in the sitting position (when possible, otherwise supine, but always in the same position for each procedure). Subject should have been calm and without distress for at least 5 minutes. Preferably, the right arm should be used to measure vital signs. Body temperature will be measured with an ear thermometer. Clinic measurements will be used to assess eligibility.
- g. SBPM will be measured once in the morning and evening during the 2-day weekend bladder e-diary collection period. SBPM measurements should start in the weekend prior to week -2 and be taken in the weekend prior to the indicated visit (or TC). SBPM will be measured on 2 consecutive days at 1 and 2 weeks after start of dosing with PED25 (day 1) and after up-titration to PED50, if not already covered by the scheduled SBPM. Measurements will be taken in the sitting position (when possible, otherwise supine, but always in the same position). Preferably, the right arm should be used. Subject should have been calm and without distress for at least 5 minutes. Morning measurement should be taken before IP intake and evening measurement should be taken prior to bedtime.
- h. Additional hematology, biochemistry and urinalysis (urinalysis dipstick) tests will be performed at visit 3/week 0 (baseline) and visit 8/week 14 (EoS) only if an AE related to hematology, biochemistry or urinalysis parameters occurred since the previous visit or at the discretion of the investigator.
- i. Urine pregnancy test will be performed for females of childbearing potential at all on-site visits.
- j. The acceptability and palatability questionnaire will be completed on one weekend day preceding at visit 7/week 12 (EoT).
- k. There will be 2 pharmacokinetic sampling days at visit 5/week 4 and visit 7/week 12 (EoT). Both pharmacokinetic sampling days will consist of collecting 1 predose (trough) sample. On pharmacokinetic sampling days, dosing should occur in the clinic and breakfast should be eaten at the clinic within 1 hour before dosing.

#### INVESTIGATIONAL PRODUCT SUPPLY

If any of the conditions outlined above in the Participant Procedures Assessment are met, if the following mitigating strategy will be employed, as needed, to ensure continuity of IP supply to the participants:

- Increase stock of IP on site to reduce number of shipments required, if site space will allow.
- Direct-to-subject shipments of IP from the site to the subject's home.

#### DATA COLLECTION REQUIREMENTS

Additional data may be collected in order to indicate how participation in the study may have been affected by a crisis and to accommodate data collection resulting from alternate measures implemented to manage the conduct of the study and participant safety.

• Critical assessments for safety and efficacy based on study endpoints to be identified as missing or altered (performed virtually, at alternative locations, out of window, or other modifications) due to the crisis.

Sponsor: APGD ISN/Protocol: 178-CL-204

EudraCT number 2016-001767-37


| 12 Appendices 12.4 List of Abbreviations and Definition of Key Study Terms | |
|---|---|
| WAS: | |
| WOCBP | Woman of childbearing potential |
| IS AMENDED TO: | |
| NONMEM | non-linear mixed effects modeling |
| <del>WOCBP</del> | Woman of childbearing potential |

| 12 Appendices 12.4 List of Abbrev WAS: | viations and Definition of Key Study Terms |
|---|---|
| Intervention | The drug, device, therapy or process under investigation in a study that is believed to have an effect on outcomes of interest in a study (e.g., health-related quality of life, efficacy, safety and pharmacoeconomics). |
| IS AMENDED TO: | |
| Intervention | The drug, device, therapy or process under investigation in a study that is believed to have an effect on outcomes of interest in a study (e.g., health-related quality of life, efficacy, safety and pharmacokineticseconomies). |


# 14 COORDINATING INVESTIGATOR'S SIGNATURE

A Phase 3, Double-blind, Randomized, Multicenter, Parallel Group, Placebo-controlled Sequential Dose Titration Study to Evaluate Efficacy, Safety and Pharmacokinetics of Mirabegron in Pediatric Subjects from 5 to < 18 Years of Age with Overactive Bladder

ISN/Protocol: 178-CL-204

ISN/Protocol 178-CL-204

**Version 2.0 Incorporating Substantial Amendment 1** 

11 Feb 2021

| | pages of this protocol for which Astellas is the sponsor. I agree that it contains tion required to conduct this study. |
|---|---|
| Coordinating | Investigator: |
| Signature: | |
| | Date (DD Mmm YYYY) |
| Printed Name: | |
| Address: | |

Sponsor: APGD ISN/Protocol: 178-CL-204 EudraCT number 2016-001767-37


### 15 SPONSOR'S SIGNATURES

(Electronic signatures are attached at the end of the document.)

